| T <sub>0</sub> | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|----------------|----------------------|---------|-------------|
| PPD | ANALTTICAL UNIT | Version | 1.0 |

| STUDY TITLE | "Prospective, Single-dose, Randomized, Open-label, |
|---|---|
| STODI TITLE | . , |
| | Crossover, Comparative Study to Establish the |
| | Bioequivalence between Levothyroxine's New |
| | Formulation vs. Levothyroxine's Approved Formulation |
| | (Eutirox® from Merck S.A. de C.V.) Given Orally at |
| | Doses of 3 Tablets of 200 µg to healthy subjects" |
| Study code: | PPD /MS200125-0008 |
| Sponsor: | Merck S.A. de C.V. |
| Clinical Unit Responsible | PPD |
| Person: | |
| | Ph PPD |
| Analytical Unit Responsible | PPD |
| Person: | |
| | Ph PPD |

| Staff | Name | Signature | Date |
|---|---|---|---|
| Prepared by: Biostatistics Responsible Person | PPD | | |
| Reviewed by:<br>Quality Assurance<br>Responsible Person | PPD | | |

| Report Type: | Pharmaceutical • | Statistical • | Other: |
|--------------|------------------|---------------|--------|
|--------------|------------------|---------------|--------|



| Co | ontent | Page |
|---|---|---|
| 1. | Introduction | 3 |
| 1.1. | Summary | 3 |
| | Software used | |
| 1.3. | Design and Analysis Methods | 3 |
| 2. | Study Element and Dosage Schedule | 4 |
| 3. | Results | |
| 3.1. | Demographic Variables (Descriptive Statistics) | 4 |
| 3.2. | Concentration's Individual Data vs Time | 6 |
| | Concentration vs. Individual and Average Time (arithmetic and logarithmic scale) | |
| 3.4.<br>Forr | Descriptive Statistics of Biological Fluid Concentration Data as a Function of Time a | and<br>49 |
| 3.5. | mulation | 50 |
| 3.5. | 1.Individual Data and Descriptive Statistics of the Pharmacokinetic Parameters | 50 |
| 4. | Variance Analysis (ANOVA) | 53 |
| 5. | Study Variability | 54 |
| 6. | Pharmacokinetic Parameters Outliers Identification | 54 |
| 7. | Bioequivalence Statistics | 57 |
| 8. | Statistical Plan Deviation | 57 |
| 9. | Discussion and Conclusion | 57 |
| 10. | Annexes | 57 |
| 11. | References | 68 |
| 12. | History of Changes | |

| T <sub>0</sub> | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|----------------|----------------------|---------|-------------|
| PPD | ANALTTICAL UNIT | Version | 1.0 |

## 1. Introduction 1.1. Summary

To determine the bioavailability of two levothyroxine pharmaceutical forms, the *reference drug* (drug A: Eutirox® approved formulation) and the test drug (drug B: Eutirox® new formulation), in male and female healthy subjects, orally, in fasting state at a dose of 600 μg (3 tablets of 200 μg/mL) of each of the study products, and to establish bioequivalence.

The sample size proposed for this protocol was 44 male and female subjects (included allowance for drop-out to ensure 34 completers), who were randomized to each of the treatment sequences where the test and reference formulations were administered in two periods, separated by a 35-day wash-out period. One subject (subject 38) was positive for cannabinoids, prior to the second dosing; therefore, he was withdrawn from the study.

The statistical analysis to conclude the possible bioequivalence between both drugs is included in this report. This was carried out with 43 evaluable subjects (8 females and 35 males),

- 1.2. As per the sampling schedule, blood samples were collected from each subject and concentration of levothyroxine were determined from plasma. Software used
- Phoenix® WinNonlin® Version 8.2, Copyright ® 1998-2018, Certara L.P. All rights reserved.

### 1.3. Design and Analysis Methods

For conducting the bioequivalence study, a 2-period and 2-sequence crossover-design was used. The estimation of an AUC<sub>0-48</sub> could be determined with a 48-h sampling-time.

The pharmacokinetic analysis of plasma concentrations was made using the WinNonlin® software, for which a non-compartmental model and real-time were considered.

 $t_{max}$  and  $C_{max}$  values were obtained directly from the measurements made. The area under the curve of plasma concentrations from  $t_0$  (dosing) to  $t_n$  (AUC<sub>n-t</sub>) was estimated by means of the trapezoid method with linear interpolation. For the determination of the area under the curve from the last sampling time to the infinite time (AUC<sub>t-∞</sub>), the quotient of the last plasma concentration between the elimination constant was determined by linear regression using the sampling points from a terminal linear logarithm, which provided the best adjustment for a straight line. The AUC<sub>0-∞</sub> was determined by the sum of the AUC<sub>0-t</sub> and AUC<sub>t-∞</sub>. This value and, everything related to it, is shown for informative purposes only. Due to the sampling times used, it was not possible to determine at least the 80 % of the AUC. Therefore, it is a truncated design at 48 h. It is important to mention that all the pharmacokinetic and statistical results included in this report correspond to the corrected concentration values. Baseline uncorrected values are shown in the appropriate annex to this study report.

| La | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|
| PPD | ANALTTICAL UNIT | Version | 1.0 |

The statistical analysis was performed with WinNonlin® software using least squares with the generalized linear model (GLM) and 90 % confidence intervals were estimated. The intrasubject studentized residual analysis for the pharmacokinetic parameters was made with Excel®.

The following model was used for the analysis:

$$Y_{ijkl} = \mu + S_k + V(S)_{i(k)} + P_j + F_l + e_{ijkl}$$
 (Chow & Liu, 2009)

Where:

Yijki Is the response (pharmacokinetic parameters) in the ith subject, the jth period,

the kth sequence and the ith treatment.

 $\mu$  Is the general mean.

 $S_k$  Is the effect of the  $k^{th}$  sequence of administration.

 $V(S)_{i(k)}$  Is the subject's i<sup>th</sup> effect on the k<sup>th</sup> sequence is considered a random effect.

P<sub>j</sub> Is the period's j<sup>th</sup> effect (or administration's phase).

F<sub>1</sub> Is the treatment or formulation's i<sup>th</sup> effect.

eijkl Is the experimental error, intra-subject variability, and it is a random effect

assumed with normal distribution, mean zero, the constant and independent

variance of the subject nested in the sequence.

Based on the error mean square determination and the geometric means determination, the estimation of the classical confidence intervals at 90 % for the test to reference ratio was made, in logarithmically-transformed previous data.

## 2. Study Element and Dosage Schedule

Table 1 shows a description of the drugs administered to the clinical research subjects.

Table 1. Study Drugs' Description

| Information | Test drug (B) | Reference drug (A) |
|---|---|---|
| Drug substance name or<br>analyte determined | Levothyroxine | Levothyroxine |
| Dosage Form | Tablets | Tablets |
| Trademark | Eutirox® new formulation | Eutirox® approved formulation |

#### 3. Results

#### 3.1. Demographic Variables (Descriptive Statistics)

Tables 2 and 3 show the individual values and the descriptive statistics for the demographic variables of the subjects who were recruited in the study, respectively.



Table 2. Individual data for demographic variables.

| Subject | Sex | Age<br>(years) | Weight<br>(Kg) | Height (m) | BMI<br>(Kg/m²) | Sequence |
|---|---|---|---|---|---|---|
| 1 | Woman | 27 | 61 | 1.68 | 21.6 | BA |
| 2 | Man | 28 | 80 | 1.76 | 25.8 | BA |
| 3 | Woman | 40 | 57.5 | 1.62 | 21.9 | BA |
| 4 | Man | 21 | 73 | 1.80 | 22.5 | AB |
| 5 | Woman | 26 | 65 | 1.56 | 26.7 | AB |
| 6 | Man | 29 | 79 | 1.82 | 23.8 | BA |
| 7 | Man | 31 | 70 | 1.78 | 22.1 | AB |
| 8 | Man | 22 | 58 | 1.66 | 21.0 | AB |
| 9 | Man | 22 | 67 | 1.78 | 21.1 | AB |
| 10 | Woman | 30 | 64 | 1.59 | 25.3 | AB |
| 11 | Man | 35 | 70 | 1.66 | 25.4 | AB |
| 12 | Man | 24 | 74.2 | 1.72 | 25.1 | BA |
| 13 | Man | 22 | 75.5 | 1.70 | 26.1 | AB |
| 14 | Man | 29 | 72 | 1.71 | 24.6 | BA |
| 15 | Man | 21 | 74 | 1.74 | 24.4 | BA |
| 16 | Man | 23 | 81 | 1.76 | 26.1 | BA |
| 17 | Man | 22 | 73 | 1.72 | 24.7 | AB |
| 18 | Man | 28 | 76 | 1.75 | 24.8 | BA |
| 19 | Woman | 51 | 55 | 1.56 | 22.6 | AB |
| 20 | Man | 20 | 55 | 1.63 | 20.7 | BA |
| 21 | Man | 21 | 66 | 1.68 | 23.4 | BA |
| 22 | Man | 28 | 76.5 | 1.88 | 21.6 | AB |
| 23 | Man | 20 | 72 | 1.72 | 24.3 | BA |
| 24 | Man | 24 | 55.5 | 1.60 | 21.7 | AB |
| 25 | Man | 34 | 71 | 1.75 | 23.2 | AB |
| 26 | Man | 24 | 75.5 | 1.83 | 22.5 | AB |
| 27 | Man | 21 | 84 | 1.80 | 25.9 | BA |
| 28 | Woman | 25 | 59 | 1.55 | 24.6 | BA |
| 29 | Man | 30 | 76 | 1.78 | 24.0 | BA |
| 30 | Man | 23 | 61 | 1.76 | 19.7 | AB |
| 31 | Man | 24 | 72 | 1.73 | 24.1 | AB |
| 32 | Man | 26 | 81 | 1.74 | 26.8 | AB |
| 33 | Woman | 22 | 52 | 1.58 | 20.8 | AB |
| 34 | Man | 22 | 61 | 1.65 | 22.4 | AB |

| ANALYTICAL LINIT | Issue | 10-Mar-2020 |
|---|---|---|
| ANALYTICAL UNIT | Version | 1.0 |
| | | 6 of 68 |
| STATISTICAL DOCUMENT | Page | |
| | ANALYTICAL UNIT STATISTICAL DOCUMENT | ANALYTICAL UNIT Version |

Table 2. Individual data for demographic variables. (Continued)

| Subject | Sex | Age<br>(years) | Weight<br>(Kg) | Height (m) | BMI<br>(Kg/m²) | Sequence |
|---|---|---|---|---|---|---|
| 35 | Man | 30 | 69.5 | 1.80 | 21.5 | AB |
| 36 | Man | 22 | 52 | 1.60 | 20.3 | BA |
| 37 | Man | 27 | 65 | 1.68 | 23.0 | BA |
| 38 | Man | 27 | 67 | 1.74 | 22.1 | BA |
| 39 | Woman | 22 | 50 | 1.53 | 21.4 | BA |
| 40 | Man | 23 | 68 | 1.76 | 22.0 | BA |
| 41 | Man | 31 | 59 | 1.60 | 23.0 | BA |
| 42 | Man | 23 | 72 | 1.74 | 23.8 | AB |
| 43 | Man | 21 | 73 | 1.84 | 21.6 | BA |
| 44 | Man | 20 | 68 | -1.72 | 23.0 | AB |

Table 3. Descriptive statistics for demographic variables.

| | Age (years) | Weight (Kg) | Height (m) | BMI (Kg/m <sup>2</sup> ) |
|---|---|---|---|---|
| Arithmetic<br>Mean | 25.93 | 67.87 | 1.71 | 23.26 |
| Standard<br>Deviation | 5.93 | 8.75 | 0.09 | 1.86 |
| %CV | 22.86 | 12.89 | 5.09 | 7.98 |

#### 3.2. Concentration's Individual Data vs Time

Levothyroxine plasma concentration data versus time, for each subject, as well as its mean value are shown in tables 4 and 5 for the reference and test drugs, respectively. Since this is an endogenous molecule, baseline levels are expected. Therefore, concentrations shown in this report correspond to the adjusted levels; i. e., the average value obtained from 3 pre-dose concentrations. The mean of the pre-doses values (corresponding to the times -0.5, -0.25 and 0.0) was subtracted from each of the individual values after administration. Any negative value obtained from the initial correction were designated as zero (0), for reference product (A), twenty seven (27) data were designated as zero, sixteen (16) cases, after the pre dose adjustment had concentration greater than zero. For the test product (B), twenty-five (25) data were designated as zero, eighteen (18) cases, after the pre dose adjustment had concentration greater than zero.

The unadjusted values, including pre-dose values used for baseline adjustment, are presented in Annex section



Table 4. Table of individual base line corrected concentrations corresponding to levothyroxine (reference drug [A]). Adjusted data, N = 43 subjects

| l | | (reference drug [A]). Adjusted data. N = 43 subjects | | | | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Form | Volunteer | | | | | | | | | | | | Time | | | | | | | | | | | | |
| | Totalisto | 0.00 | 0.50 | 1.00 | 150 | 2.00 | 2.50 | 3.00 | 3.25 | 3.50 | 3.75 | 4.00 | 4.25 | 4.50 | 4.75 | 5.00 | 5.50 | 6.00 | 6.50 | 8.00 | 10.00 | 12.00 | 24.00 | 36.00 | 48.00 |
| A | 1 | 0.00 | 0.00 | 18.08 | 25.76 | 33.62 | 59.36 | 73.07 | 77.18 | 83.03 | 73.97 | 96.39 | 98.33 | 89.28 | 90.42 | 86.81 | 79.36 | 70.08 | 72.76 | 66.78 | 58.76 | 64.49 | 57.99 | 50.27 | 45.44 |
| A | 2 | 0.95 | 3.10 | 19.25 | 33.71 | 42.76 | 45.60 | 46.32 | 54.44 | 52.37 | 51.29 | 49.24 | 55.16 | 53.62 | 4956 | 59.08 | 45.50 | 44.61 | 44.62 | 45.91 | 44.13 | 38.01 | 34.60 | 38.14 | 39.62 |
| A | 3 | 0.04 | 5.41 | 45.45 | 55.09 | 61.00 | 45.19 | 40.08 | 52.74 | 36.22 | 32.34 | 40.98 | 43.74 | 4237 | 35.11 | 31.35 | 32.92 | 32.87 | 40.23 | 29.26 | 23.10 | 27.04 | 22.63 | 22.89 | 19.76 |
| A | 4 | 0.24 | 2.22 | 15.74 | 39.37 | 55.52 | 56.51 | 59.29 | 52.39 | 51.70 | 67.12 | 49.86 | 62.41 | 59.12 | 47.28 | 48.65 | 51.19 | 41.04 | 45.56 | 47.40 | 37.83 | 38.98 | 30.15 | 29.06 | 23.10 |
| A | 5 | 0.00 | 1.31 | 22.68 | 32.52 | 36.69 | 37.64 | 53.06 | 45.51 | 52.17 | 47.12 | 51.78 | 51.68 | 52.20 | 48.46 | 46.44 | 48.39 | 41.28 | 34.87 | 33.99 | 32.68 | 26.28 | 25.10 | 19.42 | 28.01 |
| A | 6 | 0.00 | 2.13 | 4.16 | 21.55 | 49.91 | 64.49 | 63.06 | 57.44 | 57.84 | 58.86 | 49.98 | 57.66 | 51.39 | 55.90 | 53.28 | 53.25 | 52.89 | 55.45 | 53.91 | 44.06 | 42.77 | 36.80 | 32.71 | 28.96 |
| A | 7 | 0.00 | 3.04 | 16.50 | 28.04 | 29.99 | 34.44 | 57.68 | 48.23 | 54.39 | 64.47 | 56.21 | 63.47 | 49.44 | 53.45 | 41.29 | 40.28 | 43.31 | 41.76 | 53.16 | 33.20 | 27.71 | 38.43 | 28.84 | 30.49 |
| A | 8 | 0.00 | 3.03 | 31.05 | 44.07 | 58.34 | 64.72 | 57.08 | 63.33 | 49.74 | 58.34 | 60.40 | 60.22 | 57.79 | 55.20 | 61.69 | 54.74 | 61.39 | 47.24 | 51.10 | 45.10 | 39.51 | 32.40 | 24.89 | 23.33 |
| A | 9 | 0.00 | 7.14 | 11.53 | 15.62 | 12.87 | 19.26 | 26.65 | 47.89 | 54.01 | 64.75 | 59.99 | 77.35 | 76.86 | 84.71 | 80.43 | 71.34 | 71.58 | 62.30 | 60.40 | 49.55 | 39.32 | 45.23 | 37.58 | 38.79 |
| A | 10 | 0.00 | 0.00 | 1.86 | 36.34 | 52.20 | 58.30 | 62.78 | 71.37 | 70.04 | 56.75 | 74.84 | 79.08 | 75.58 | 81.77 | 61.19 | 74.82 | 63.72 | 58.42 | 62.81 | 55.65 | 48.99 | 41.36 | 31.64 | 30.82 |
| A | 11 | 0.00 | 0.00 | 14.75 | 27.54 | 68.86 | 40.49 | 52.38 | 55.51 | 51.51 | 55.85 | 61.42 | 60.76 | 64.98 | 59.66 | 58.66 | 58.59 | 51.79 | 41.77 | 39.55 | 36.52 | 30.60 | 40.18 | 43.35 | 25.62 |
| A | 12 | 0.00 | 6.19 | 26.38 | 50.30 | 54.73 | 63.00 | 69.82 | 61.41 | 63.27 | 65.19 | 60.02 | 65.76 | 56.83 | 51.26 | 52.95 | 55.53 | 54.36 | 47.84 | 57.10 | 45.06 | 42.70 | 40.25 | 32.52 | 29.49 |
| A | 13 | 0.00 | 7.13 | 29.24 | 59.72 | 46.49 | 62.06 | 60.77 | 60.84 | 58.21 | 50.85 | 40.75 | 60.79 | 53.75 | 5437 | 50.33 | 55.28 | 52.64 | 41.59 | 48.04 | 47.04 | 35.90 | 42.43 | 43.72 | 34.56 |
| A | 14 | 1.25 | 3.33 | 24.00 | 43.40 | 49.00 | 61.37 | 54.90 | 63.59 | 57.32 | 59.44 | 62.16 | 63.16 | 56.87 | 69.84 | 61.81 | 55.00 | 58.65 | 55.78 | 58.93 | 29.87 | 48.92 | 40.85 | 32.00 | 31.63 |
| A | 15 | 0.22 | 0.00 | 5.43 | 0.00 | 13.29 | 25.09 | 22.85 | 30.79 | 43.23 | 41.27 | 36.76 | 40.83 | 44.14 | 4051 | 51.95 | 42.80 | 39.20 | 34.20 | 31.48 | 41.79 | 36.83 | 23.05 | 15.76 | 25.49 |
| A | 16 | 0.00 | 8.00 | 26.69 | 33.12 | 35.23 | 55.66 | 56.88 | 66.06 | 67.07 | 61.11 | 56.07 | 49.65 | 49.91 | 58.86 | 48.93 | 60.42 | 55.01 | 53.01 | 37.59 | 40.86 | 36.36 | 30.10 | 20.19 | 29.89 |
| A | 17 | 0.00 | 4.78 | 11.47 | 14.59 | 24.96 | 42.11 | 66.14 | 60.41 | 54.70 | 50.91 | 59.30 | 62.16 | 46.06 | 5230 | 58.93 | 50.21 | 49.20 | 54.71 | 54.37 | 43.89 | 41.10 | 36.45 | 23.89 | 14.73 |
| A | 18 | 0.00 | 2.12 | 33.99 | 4.4 | 52.12 | 58.14 | 63.81 | 61.51 | 60.94 | 67.71 | 63.07 | 61.82 | 58.70 | 56.20 | 55.17 | 58.14 | 56.91 | 47.85 | 48.84 | 42.38 | 45.57 | 39.15 | 29.68 | 29.96 |
| A | 19 | 0.09 | 4.33 | 43.58 | 51.94 | 49.37 | 59.52 | 60.20 | 58.16 | 64.98 | 60.57 | 49.71 | 73.11 | 55.00 | 52.70 | 51.18 | 55.10 | 42.80 | 45.87 | 49.52 | 39.35 | 39.24 | 50.09 | 35.00 | 34.00 |
| A | 20 | 0.00 | 6.32 | 34.84 | 68.56 | 71.10 | 66.47 | 74.56 | 67.80 | 74.61 | 68.09 | 68.12 | 67.97 | 64.24 | 63.56 | 67.60 | 67.08 | 59.46 | 56.90 | 60.97 | 49.31 | 44.45 | 48.93 | 49.42 | 37.82 |
| A | 21 | 0.00 | 2.99 | 27.13 | 56.35 | 53.46 | 61.00 | 68.61 | 64.96 | 62.32 | 62.87 | 68.94 | 65.30 | 65.99 | 60.89 | 58.27 | 57.45 | 43.04 | 48.99 | 54.87 | 38.81 | 35.62 | 40.28 | 34.92 | 32.53 |
| A | 22 | 0.00 | 0.00 | 5.47 | 10.20 | 13.43 | 18.87 | 24.83 | 24.02 | 34.94 | 35.63 | 30.05 | 32.89 | 50.81 | 27.92 | 26.94 | 30.33 | 31.08 | 30.71 | 24.96 | 31.68 | 24.79 | 24.17 | 23.12 | 14.56 |
| A | 23 | 0.00 | 2.03 | 36.97 | 47.98 | 46.30 | 49.23 | 47.93 | 48.24 | 44.80 | 50.16 | 45.70 | 48.89 | 45.05 | 37.36 | 44.33 | 40.72 | 37.82 | 34.38 | 36.27 | 28.80 | 21.73 | 25.25 | 26.87 | 19.00 |
| A | 24 | 0.00 | 0.00 | 23.24 | 45.18 | 53.90 | 75.62 | 66.74 | 63.45 | 71.36 | 69.87 | 65.15 | 66.94 | 55.11 | 53.43 | 49.25 | 55.26 | 46.69 | 41.32 | 41.62 | 34.62 | 35.28 | 39.99 | 22.34 | 19.02 |
| A | 25 | 0.00 | 0.00 | 32.21 | 53.96 | 47.94 | 53.88 | 29.00 | 43.37 | 37.39 | 37.45 | 41.45 | 59.68 | 41.38 | 45.81 | 35.74 | 42.69 | 43.87 | 40.04 | 38.76 | 29.82 | 26.81 | 24.73 | 26.95 | 26.58 |
| A | 26 | 3.32 | 4.41 | 10.30 | 27.04 | 37.86 | 49.47 | 40.82 | 46.52 | 36.61 | 42.67 | 34.47 | 39.69 | 35.68 | 30.91 | 36.29 | 43.15 | 35.12 | 42.01 | 51.65 | 37.41 | 33.72 | 36.45 | 34.34 | 25.45 |
| A | 27 | 0.65 | 0.00 | 17.31 | 34.50 | 41.84 | 42.94 | 48.06 | 46.90 | 44.91 | 46.60 | 42.51 | 47.33 | 40.83 | 33.39 | 36.48 | 42.11 | 42.24 | 39.78 | 37.72 | 36.08 | 30.58 | 29.83 | 23.78 | 23.70 |
| A | 28 | 0.00 | 5.77 | 15.58 | 47.72 | 61.94 | 68.74 | 121.16 | 65.30 | 80.02 | 71.97 | 68.57 | 57.51 | 63.91 | 52.81 | 77.31 | 46.12 | 54.33 | 56.03 | 52.65 | 51.64 | 51.99 | 41.44 | 56.27 | 41.17 |
| A | 29 | 0.74 | 12.68 | 11.63 | 31.89 | 56.96 | 65.35 | 39.34 | 55.86 | 54.04 | 41.67 | 55.05 | 53.18 | 50.24 | 46.79 | 41.93 | 42.84 | 36.96 | 36.07 | 49.20 | 36.21 | 31.70 | 41.18 | 28.21 | 20.81 |
| A | 30 | 1.66 | 4.82 | 24.29 | 33.91 | 29.16 | 52.40 | 32.50 | 68.88 | 55.06 | 63.72 | 53.08 | 58.09 | 57.83 | 52,74 | 51.52 | 49.09 | 43.36 | 40.22 | 48.23 | 42.74 | 42.01 | 40.28 | 48.76 | 37.67 |
| A | 31 | 0.00 | 4.57 | 9.30 | 34.95 | 34.96 | 45.12 | 39.65 | 40.99 | 39.33 | 39.99 | 38.43 | 45.02 | 49.54 | 48.10 | 36.09 | 23.02 | 30.45 | 31.71 | 32.90 | 17.75 | 18.83 | 27.31 | 10.97 | 15.01 |
| A | 32 | 3.18 | 6.59 | 50.40 | 53.47 | 61.04 | 43.57 | 39.55 | 38.07 | 39.94 | 44.61 | 36.54 | 42.04 | 36.95 | 3454 | 35.68 | 39.39 | 33.26 | 34.52 | 34.90 | 38.95 | 25.06 | 30.26 | 30.86 | 30.84 |
| A | 33 | 3.27 | 8.57 | 37.56 | 45.26 | 57.55 | 76.35 | 71.51 | 77.89 | 82.25 | 76.90 | 79.66 | 86.93 | 85.56 | 73.60 | 81.06 | 85.56 | 65.23 | 73.26 | 64.06 | 59.41 | 64.31 | 50.72 | 58.18 | 55.61 |
| A | 34 | 0.00 | 0.00 | 9.17 | 12.53 | 22.41 | 25.61 | 40.22 | 48.91 | 60.92 | 47.62 | 48.59 | 57.50 | 43.24 | 4453 | 38.47 | 42.39 | 36.95 | 27.96 | 40.18 | 31.81 | 30.39 | 36.36 | 22.47 | 26.44 |
| A | 35 | 0.00 | 3.18 | 38.87 | 59.17 | 59.46 | 54.39 | 53.87 | 48.81 | 45.85 | 45.87 | 46.05 | 54.19 | 44.10 | 31.48 | 43.13 | 45.66 | 41.79 | 43.02 | 47.03 | 48.06 | 34.11 | 39.58 | 36.52 | 31.71 |
| A | 36 | 3.49 | 4.87 | 51.03 | 62.19 | 56.79 | 52.03 | 65.33 | 74.82 | 61.33 | 64.84 | 57.09 | 59.12 | 52.43 | 54.17 | 51.54 | 51.65 | 46.36 | 45.53 | 41.02 | 42.03 | 35.39 | 15.52 | 29.58 | 30.34 |
| A | 37 | 0.00 | 0.00 | 36.37 | 47.22 | 60.30 | 55.05 | 54.15 | 57.78 | 59.60 | 55.54 | 52.78 | 54.60 | 52.35 | 47.95 | 49.44 | 53.06 | 53.52 | 47.45 | 48.10 | 38.77 | 42.02 | 36.21 | 33.56 | 29.36 |
| A | 39 | 2.71 | 7.98 | 81.95 | 90.27 | 85.98 | 100.38 | 86.78 | 82.14 | 79.05 | 82.19 | 83.16 | 89.05 | 86.73 | 78.73 | 73.45 | 85.70 | 79.63 | 77.27 | 68.79 | 68.89 | 64.91 | 51.98 | 47.47 | 49.11 |
| A | 40 | 9.72 | 5.85 | 19.24 | 30.92 | 38.85 | 73.16 | 76.71 | 80.95 | 81.27 | 85.18 | 84.23 | 90.55 | 87.54 | 83.46 | 86.80 | 64.95 | 86.35 | 79.86 | 79.95 | 70.52 | 66.20 | 48.16 | 49.29 | 34.43 |
| A | 41 | 0.00 | 3.33 | 36.99 | 51.23 | 57.14 | 52.66 | 64.01 | 64.35 | 65.86 | 59.42 | 61.18 | 62.57 | 72.78 | 52.99 | 46.20 | 40.05 | 52.40 | 46.42 | 48.37 | 39.45 | 32.90 | 45.04 | 27.53 | 30.69 |
| A | 42 | 0.00 | 2.16 | 6.44 | 17.24 | 24.25 | 20.91 | 22.88 | 30.64 | 39.15 | 40.03 | 40.06 | 44.51 | 42.99 | 38.71 | 35.24 | 35.24 | 32.46 | 34.83 | 33.72 | 23.89 | 22.85 | 25.08 | 27.12 | 27.15 |
| A | 43 | 0.00 | 9.75 | 0.00 | 51.13 | 47.33 | 44.91 | 48.87 | 41.58 | 43.98 | 45.80 | 45.19 | 49.97 | 43.30 | 45.06 | 44.44 | 39.67 | 40.08 | 35.99 | 44.86 | 30.43 | 31.86 | 29.09 | 34.59 | 23.61 |
| A | 44 | 1.00 | 4.89 | 22.37 | 35.41 | 45.79 | 51.87 | 48.87 | 48.92 | 46.34 | 44.27 | 43.36 | 50.47 | 44.87 | 40.22 | 41.19 | 38.69 | 39.78 | 35.92 | 30.08 | 30.31 | 30.37 | 27.85 | 26.68 | 26.28 |
| | netic Mean | 0.76 | 3.81 | 24.20 | 39.66 | 46.34 | 52.39 | 54.72 | 56.28 | 56.36 | 56.07 | 55.10 | 59.79 | 55.98 | 52.95 | 52.29 | 51.27 | 48.73 | 46.65 | 47.46 | 40.66 | 37.87 | 36.39 | 32.59 | 29.62 |
| - | rd Deviation | 1.75 | 3.08 | 16.08 | 17.36 | 16.00 | 16.33 | 18.63 | 13.46 | 13.52 | 12.82 | 14.49 | 14.14 | 13.92 | 15.08 | 14.89 | 13.83 | 12.98 | 12.44 | 11.90 | 11.07 | 11.57 | 9.34 | 10.70 | 8.70 |
| | %CV | 231.17 | 80.71 | 66.46 | 43.78 | 34.52 | 31.17 | 34.04 | 23.91 | 23.99 | 22.87 | 26.30 | 23.65 | 24.86 | 28.48 | 28.47 | 26.98 | 26.64 | 26.66 | 25.06 | 27.24 | 30.56 | 25.68 | 32.83 | 29.39 |



Table 5. Table of individual base line corrected concentrations corresponding to levothyroxine (test drug [B]). Adjusted data. N = 43 subjects

| | | | | | | | | | | | | | Time | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Form | Volunteer | 0.00 | 0.50 | 1.00 | 150 | 2.00 | 2.50 | 3.00 | 3.25 | 3.50 | 3.75 | 4.00 | 4.25 | 4.50 | 4.75 | 5.00 | 5.50 | 6.00 | 6.50 | 8.00 | 10.00 | 12.00 | 24.00 | 36.00 | 48.00 |
| Ь | 1 | 0.36 | 2.79 | 17.91 | 31.20 | 40.46 | 46.99 | 54.85 | 69.43 | 65.89 | 84.97 | 82.64 | 75.96 | 75.05 | 74.65 | 73.40 | 58.34 | 55.21 | 49.74 | 58.80 | 50.79 | 43.11 | 40.03 | 41.77 | 21.93 |
| B | 2 | 0.00 | 3.77 | 34.31 | 49.71 | 55.52 | 52.76 | 57.53 | 48.95 | 52.17 | 46.50 | 47.92 | 52.87 | 49.14 | 47.08 | 40.16 | 42.16 | 59.26 | 36.21 | 33.32 | 27.19 | 30.20 | 28.83 | 23.76 | 18.41 |
| l B | 3 | 0.00 | 4.56 | 42.17 | 56.41 | 39.98 | 44.50 | 35.97 | 34.31 | 41.07 | 39.67 | 24.39 | 34.59 | 48.09 | 36.40 | 36.96 | 24.59 | 25.43 | 20.77 | 6.44 | 12.78 | 13.72 | 20.74 | 27.56 | 24.82 |
| В | 4 | 0.00 | 5.29 | 16.63 | 39.25 | 54.71 | 55.69 | 63.95 | 60.72 | 55.17 | 54.09 | 53.89 | 52.11 | 47.96 | 42.13 | 41.46 | 42.58 | 43.26 | 40.44 | 41.92 | 37.87 | 37.55 | 30.28 | 31.89 | 19.31 |
| B | 5 | 0.00 | 3.60 | 5.15 | 9.40 | 9.21 | 13.56 | 15.13 | 20.55 | 12.57 | 26.79 | 23.36 | 37.49 | 41.91 | 59.02 | 53.80 | 47.48 | 40.41 | 42.82 | 37.95 | 30.38 | 23.75 | 29.37 | 27.62 | 24.90 |
| B | 6 | 0.24 | 0.00 | 4.78 | 15.29 | 14.54 | 16.90 | 16.01 | 25.48 | 28.34 | 33.35 | 39.92 | 48.64 | 45.53 | 40.81 | 33.57 | 38.87 | 34.07 | 33.18 | 29.28 | 28.03 | 30.25 | 25.72 | 17.88 | 23.41 |
| l B | 7 | 0.53 | 8.73 | 36.06 | 41.76 | 49.65 | 54.84 | 69.43 | 55.04 | 55.85 | 42.18 | 45.25 | 46.82 | 50.46 | 45.27 | 55.71 | 51.90 | 50.42 | 49.95 | 43.06 | 45.35 | 38.26 | 40.62 | 36.32 | 39.65 |
| B | 8 | 0.00 | 22.49 | 48.49 | 61.64 | 66.18 | 57.51 | 58.67 | 60.60 | 59.30 | 53.33 | 53.95 | 60.19 | 52.90 | 54.45 | 47.68 | 53.99 | 49.81 | 44.60 | 40.06 | 38.55 | 37.62 | 31.20 | 44.63 | 31.79 |
| B | 9 | 2.13 | 0.00 | 25.40 | 43.56 | 69.04 | 86.57 | 93.54 | 87.80 | 97.45 | 98.59 | 101.74 | 104.57 | 94.06 | 96.22 | 97.71 | 95.00 | 96.72 | 80.81 | 73.49 | 63.24 | 63.56 | 42.01 | 56.25 | 35.96 |
| В | 10 | 0.00 | 1.43 | 20.93 | 48.51 | 67.80 | 73.54 | 79.88 | 97.25 | 96.00 | 79.94 | 74.34 | 82.17 | 85.29 | 8434 | 89.85 | 70.20 | 82.59 | 77.27 | 76.82 | 57.96 | 74.36 | 52.40 | 44.80 | 41.12 |
| В | 11 | 0.39 | 4.73 | 23.43 | 59.64 | 67.87 | 71.66 | 67.73 | 72.27 | 69.20 | 62.75 | 61.72 | 63.41 | 57.79 | 63.43 | 62.11 | 56.08 | 64.38 | 62.71 | 53.65 | 51.28 | 41.67 | 49.91 | 50.30 | 32.51 |
| В | 12 | 0.00 | 1.73 | 24.09 | 40.62 | 54.56 | 63.04 | 54.30 | 58.19 | 57.49 | 57.61 | 60.91 | 69.15 | 55.95 | 56.19 | 53.60 | 48.72 | 52.36 | 44.18 | 53.11 | 38.15 | 35.54 | 48.57 | 40.50 | 27.35 |
| B | 13 | 0.00 | 4.26 | 32.89 | 49.68 | 47.43 | 51.61 | 49.51 | 42.51 | 46.20 | 36.71 | 46.03 | 51.70 | 46.62 | 43.99 | 42.89 | 43.98 | 42.75 | 30.11 | 40.77 | 31.17 | 32.40 | 19.77 | 37.89 | 34.95 |
| B | 14 | 0.20 | 6.14 | 33.16 | 53.17 | 55.00 | 63.97 | 53.37 | 56.39 | 60.64 | 61.77 | 62.86 | 63.12 | 63.19 | 61.68 | 61.09 | 68.12 | 65.83 | 60.17 | 62.76 | 55.44 | 52.45 | 40.06 | 50.94 | 35.83 |
| В | 15 | 0.00 | 1.87 | 19.48 | 33.62 | 24.27 | 41.18 | 46.90 | 50.19 | 44.68 | 45.12 | 44.01 | 53.99 | 44.32 | 54.48 | 39.59 | 38.31 | 47.15 | 39.17 | 53.60 | 39.42 | 38.73 | 31.88 | 33.06 | 36.67 |
| B | 16 | 6.49 | 2.41 | 17.61 | 33.54 | 55.03 | 45.07 | 44.78 | 43.47 | 41.31 | 39.68 | 43.17 | 48.86 | 45.04 | 41.85 | 39.92 | 45.29 | 36.25 | 41.96 | 38.01 | 34.67 | 29.87 | 43.55 | 27.70 | 20.88 |
| В | 17 | 0.00 | 2.89 | 17.25 | 28.91 | 44.51 | 50.85 | 52.11 | 42.23 | 68.33 | 66.23 | 58.97 | 67.80 | 63.88 | 51.40 | 51.40 | 51.97 | 45.41 | 38.59 | 55.86 | 42.85 | 36.91 | 34.72 | 34.95 | 11.84 |
| B | 18 | 0.00 | 7.27 | 35.61 | 47.18 | 54.82 | 65.71 | 68.11 | 62.74 | 63.33 | 61.82 | 60.32 | 65.35 | 57.65 | 5451 | 55.82 | 53.49 | 51.41 | 51.62 | 53.01 | 51.62 | 47.24 | 37.26 | 34.72 | 30.84 |
| В | 19 | 0.30 | 2.50 | 29.64 | 42.62 | 56.02 | 41.53 | 52.48 | 46.66 | 42.04 | 38.77 | 36.36 | 50.90 | 47.34 | 47.19 | 43.10 | 45.24 | 55.43 | 49.00 | 41.15 | 38.82 | 37.83 | 29.34 | 23.85 | 25.A7 |
| В | 20 | 0.01 | 7.07 | 39.40 | 53.19 | 56.06 | 54.98 | 59.97 | 56.63 | 49.46 | 49.00 | 48.20 | 60.44 | 48.90 | 4234 | 37.45 | 36.18 | 39.47 | 39.90 | 43.58 | 32.28 | 24.00 | 29.55 | 33.42 | 23.14 |
| B | 21 | 3.56 | 15.88 | 35.26 | 58.93 | 59.18 | 66.13 | 66.40 | 59.28 | 65.38 | 62.22 | 62.60 | 67.03 | 61.85 | 49.99 | 53.00 | 53.79 | 54.12 | 59.51 | 64.38 | 46.40 | 43.97 | 39.84 | 41.86 | 24.83 |
| В | 22 | 1.39 | 0.00 | 18.07 | 34.38 | 30.99 | 38.85 | 43.21 | 42.46 | 37.15 | 39.86 | 40.72 | 37.81 | 36.49 | 32.74 | 43.65 | 35.78 | 37.49 | 37.29 | 30.36 | 32.87 | 28.72 | 28.66 | 24.22 | 26.61 |
| В | 23 | 1.89 | 11.64 | 49.76 | 70.84 | 68.59 | 73.24 | 60.25 | 66.61 | 61.33 | 60.29 | 61.24 | 67.83 | 61.56 | 54.26 | 53.77 | 49.82 | 48.79 | 4434 | 40.53 | 40.50 | 38.97 | 39.37 | 32.88 | 30.72 |
| В | 24 | 0.76 | 0.00 | 0.00 | 0.00 | 9.34 | 11.89 | 16.72 | 10.93 | 12.35 | 1855 | 39.45 | 55.64 | 54.80 | 60.54 | 51.26 | 45.55 | 29.73 | 33.85 | 36.69 | 21.42 | 26.65 | 34.25 | 24.89 | 26.37 |
| В | 25 | 0.00 | 20.25 | 50.91 | 60.79 | 55.35 | 47.89 | 56.13 | 42.26 | 55.71 | 62.69 | 42.97 | 51.28 | 40.88 | 54.72 | 45.57 | 57.57 | 41.01 | 53.43 | 44.70 | 50.85 | 34.92 | 47.30 | 31.89 | 26.78 |
| В | 26 | 0.00 | 0.00 | 11.65 | 25.16 | 35.14 | 51.11 | 54.58 | 50.08 | 49.19 | 53.50 | 48.08 | 46.87 | 46.09 | 46.22 | 47.47 | 45.86 | 40.73 | 45.93 | 49.16 | 42.23 | 41.84 | 36.91 | 35.69 | 25.87 |
| В | 27 | 0.00 | 1.22 | 26.36 | 39.15 | 42.23 | 49.84 | 44.22 | 42.60 | 46.63 | 45.42 | 51.14 | 52.34 | 42.09 | 38.86 | 45.57 | 39.84 | 46.78 | 32.39 | 40.71 | 30.76 | 30.65 | 29.61 | 24.19 | 14.63 |
| В | 28 | 0.00 | 10.78 | 40.05 | 31.95 | 44.49 | 35.97 | 105.75 | 93.10 | 57.87 | 91.63 | 58.16 | 45.44 | 69.72 | 71.26 | 80.92 | 49.71 | 12.65 | 45.55 | 25.46 | 34.32 | 40.80 | 41.93 | 32.50 | 24.17 |
| В | 29 | 0.00 | 0.46 | 0.00 | 0.00 | 36.95 | 40.43 | 41.45 | 40.61 | 47.14 | 44.64 | 44.35 | 60.17 | 57.37 | 5235 | 49.79 | 49.87 | 45.56 | 39.91 | 44.89 | 26.18 | 37.92 | 34.80 | 0.00 | 6.82 |
| В | 30 | 3.11 | 3.63 | 25.34 | 46.10 | 42.17 | 53.40 | 36.85 | 65.54 | 54.82 | 71.68 | 55.55 | 49.89 | 49.80 | 47.11 | 46.88 | 43.70 | 41.96 | 40.53 | 37.15 | 36.33 | 35.24 | 38.98 | 41.39 | 34.86 |
| В | 31 | 0.00 | 3.80 | 33.71 | 46.73 | 52.87 | 51.74 | 62.01 | 49.53 | 53.25 | 50.33 | 46.42 | 46.59 | 48.00 | 42.24 | 56.14 | 46.41 | 55.85 | 38.69 | 40.30 | 32.69 | 30.85 | 35.30 | 38.03 | 24.01 |
| В | 32 | 0.00 | 9.47 | 44.44 | 56.18 | 47.62 | 56.23 | 57.42 | 50.04 | 44.53 | 62.17 | 38.50 | 48.71 | 47.84 | 42.93 | 35.65 | 38.00 | 42.37 | 35.78 | 39.37 | 30.91 | 32.49 | 36.47 | 24.68 | 22.33 |
| В | 33 | 0.00 | 20.22 | 62.72 | 82.18 | 79.02 | 69.15 | 69.81 | 61.80 | 61.79 | 6231 | 64.57 | 66.39 | 66.69 | 60.32 | 61.34 | 53.11 | 54.58 | 54.40 | 52.44 | 42.43 | 45.74 | 43.60 | 28.55 | 30.88 |
| В | 34 | 1.28 | 10.99 | 30.74 | 50.42 | 63.83 | 70.24 | 58.56 | 55.87 | 57.01 | 58.08 | 59.78 | 68.78 | 57.30 | 51.35 | 47.19 | 41.26 | 47.67 | 40.39 | 36.00 | 28.07 | 38.33 | 29.43 | 24.24 | 17.34 |
| В | 35 | 0.17 | 0.00 | 0.00 | 16.04 | 20.92 | 49.01 | 52.07 | 36.70 | 41.30 | 49.07 | 28.33 | 38.25 | 44.89 | 44.85 | 39.72 | 35.70 | 51.67 | 45.29 | 37.17 | 26.76 | 35.85 | 36.73 | 24.02 | 41.01 |
| В | 36 | 1.83 | 17.66 | 60.21 | 64.87 | 70.08 | 66.77 | 45.41 | 52.85 | 63.36 | 47.07 | 57.71 | 63.12 | 54.05 | 56.11 | 50.51 | 50.47 | 40.10 | 42.39 | 46.20 | 42.17 | 32.18 | 29.81 | 35.13 | 36.58 |
| В | 37 | 0.00 | 6.08 | 3.52 | 25.64 | 40.87 | 52.82 | 60.91 | 61.67 | 62.32 | 64.41 | 57.07 | 61.67 | 51.50 | 54.86 | 57.06 | 68.30 | 54.04 | 50.03 | 46.56 | 45.74 | 43.97 | 43.70 | 37.54 | 39.90 |
| В | 39 | 0.00 | 21.11 | 58.94 | 82.41 | 86.16 | 91.74 | 86.69 | 73.80 | 73.91 | 84.89 | 84.48 | 70.66 | 94.09 | 85.59 | 77.05 | 60.60 | 52.98 | 58.79 | 62.34 | 55.82 | 45.68 | 48.10 | 33.44 | 35.15 |
| В | 40 | 0.00 | 0.00 | 16.31 | 31.43 | 43.30 | 58.76 | 65.02 | 68.52 | 74.09 | 71.22 | 70.39 | 78.08 | 75.35 | 70.39 | 72.83 | 71.95 | 65.40 | 65.58 | 65.92 | 59.63 | 58.56 | 42.80 | 37.96 | 38.58 |
| В | 41 | 0.00 | 14.77 | 39.58 | 62.91 | 57.36 | 79.08 | 49.75 | 52.69 | 57.46 | 38.34 | 54.72 | 63.73 | 47.79 | 41.76 | 36.95 | 59.50 | 40.42 | 34.98 | 63.09 | 26.06 | 40.04 | 32.28 | 25.61 | 17.70 |
| В | 42 | 0.00 | 5.13 | 20.63 | 29.26 | 20.68 | 31.73 | 33.98 | 30.70 | 33.13 | 32.32 | 31.38 | 33.26 | 26.93 | 29.62 | 29.99 | 27.70 | 27.90 | 27.14 | 31.69 | 23.39 | 20.83 | 27.09 | 24.76 | 27.53 |
| В | 43 | 0.98 | 5.77 | 41.87 | 50.89 | 50.10 | 56.81 | 46.08 | 50.09 | 47.89 | 54.80 | 50.80 | 48.40 | 41.95 | 4031 | 46.32 | 40.53 | 37.32 | 32.31 | 36.35 | 33.93 | 29.34 | 22.89 | 21.13 | 30.42 |
| В | 44 | 0.00 | 5.77 | 37.85 | 47.59 | 41.39 | 37.75 | 41.29 | 37.34 | 38.76 | 39.51 | 36.07 | 41.87 | 43.03 | 39.25 | 36.83 | 30.10 | 39.51 | 33.49 | 34.83 | 27.96 | 28.45 | 28.68 | 16.07 | 27.54 |
| Arithm | netic Mean | 0.60 | 6.47 | 28.66 | 43.09 | 48.40 | 53.33 | 54.62 | 53.17 | 53.55 | 5451 | 52.43 | 57.09 | 54.47 | 52.68 | 51.69 | 49.01 | 47.59 | 44.77 | 45.18 | 38.26 | 37.47 | 35.68 | 32.10 | 27.71 |
| Standar | d Deviation | 1.26 | 6.44 | 16.39 | 18.77 | 17.54 | 17.09 | 18.05 | 17.42 | 16.73 | 17.20 | 15.71 | 13.97 | 14.10 | 14.12 | 14.93 | 12.97 | 14.27 | 12.34 | 13.45 | 11.31 | 10.93 | 7.92 | 10.24 | 8.06 |
| | KCV | 211.29 | 99.62 | 57.18 | 43.57 | 36.23 | 32.05 | 33.05 | 32.76 | 31.24 | 31.56 | 29.97 | 24.48 | 25.89 | 26.81 | 28.88 | 26.47 | 29.99 | 27.57 | 29.77 | 29.56 | 29.18 | 22.18 | 31.89 | 29.09 |

As can be seen in tables 4 and 5 for the reference (A) and test drugs (B), at time 0.00 h, the levothyroxine plasma concentrations values were other than 0.00 ng/mL for some of the subjects. However, subjects with pre-dose concentrations other than 0.00 ng/mL were reported. Table 6 shows subjects with concentrations other than 0.00 ng/mL.

| T <sub>a</sub> | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|----------------|----------------------|---------|-------------|
| PPD | ANALI IICAL ONII | Version | 1.0 |
| PPD | | | 9 of 68 |
| | STATISTICAL DOCUMENT | Page | |

Table 6. Subjects with concentrations other than 0.00 ng/mL at time zero.

| Subject | Form | Pre-dose<br>concentration<br>(ng/mL) | C <sub>max</sub> (ng/mL) | % pre-dose<br>concentration<br>with respect to<br>C <sub>max</sub> |
|---|---|---|---|---|
| 2 | Α | 0.95 | 59.08 | 1.60 |
| 3 | Α | 0.04 | 61.00 | 0.07 |
| 4 | Α | 0.24 | 67.12 | 0.36 |
| 14 | Α | 1.25 | 69.84 | 1.79 |
| 15 | Α | 0.22 | 51.95 | 0.42 |
| 19 | Α | 0.09 | 73.11 | -0.13 |
| 26 | Α | 3.32 | 51.65 | 6.42 |
| 27 | Α | 0.65 | 48.06 | 1.36 |
| 29 | Α | 0.74 | 65.35 | 1.14 |
| 30 | Α | 1.66 | 68.88 | 2.41 |
| 32 | Α | 3.18 | 61.04 | 5.21 |
| 33 | Α | 3.27 | 86.93 | 3.76 |
| 36 | Α | 3.49 | 74.82 | 4.66 |
| 39 | Α | 2.71 | 100.38 | 2.70 |
| 40 | Α | 9.72 | 90.55 | 10.74 |
| 44 | Α | 1.00 | 51.87 | 1.93 |
| 1 | В | 0.36 | 84.97 | 0.42 |
| 6 | В | 0.24 | 48.64 | 0.50 |
| 7 | В | 0.53 | 69.43 | 0.76 |
| 9 | В | 2.18 | 104.57 | 2.03 |
| 11 | В | 0.39 | 72.27 | 0.54 |
| 14 | В | 0.20 | 68.12 | 0.29 |
| 16 | В | 6.49 | 55.03 | 11.80 |
| 19 | В | 0.30 | 56.02 | 0.53 |
| 20 | В | 0.01 | 60.44 | 0.02 |
| 21 | В | 3.56 | 67.03 | 5.31 |
| 22 | В | 1.39 | 43.65 | 3.19 |
| 23 | В | 1.89 | 73.24 | 2.58 |
| 24 | В | 0.76 | 60.54 | 1.26 |
| 30 | В | 3.11 | 71.68 | 4.34 |
| 34 | В | 1.28 | 70.24 | 1.82 |
| 35 | В | 0.17 | 52.07 | 0.33 |
| 36 | В | 1.83 | 70.08 | 2.61 |
| 43 | В | 0.98 | 56.81 | 1.73 |

As per data shown in table 6, subjects 26, 32, and 40 with the reference formulation (A), and subjects 16 and 21 with the test formulation(B) had pre-dose concentrations higher than 5 % of the  $C_{\text{max}}$  corresponding value. Thus, as per annex C.5, part a) of the Mexican Official Standard, NOM-177-SSA1-2013, the data of these subjects must be removed from the statistical analysis. Therefore, from now on, all results shown do not include subjects 16, 21, 26, 32, and 40.

| L | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|
| PPD | ANALI HOAL ONII | Version | 1.0 |

# 3.3. Concentration vs. Individual and Average Time (arithmetic and logarithmic scale)

The non-adjusted plasma concentration time profiles of levothyroxine for test (B) and reference (A) products are shown from figures 1 to 38 in the arithmetic scale, from 39 to 76 in the logarithmic scale and in figures 77 and 78 those corresponding to the average plots in the arithmetic and logarithmic scale, respectively.

Volunteer=1



Figure 1. Levothyroxine concentration vs. subject 1's time plot, on an arithmetic scale, postdose of the test-drug, and reference-drug.

Volunteer=2



Figure 2. Levothyroxine concentration vs. subject 2's time plot, on an arithmetic scale, postdose of the test-drug and reference-drug.

| | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|
| PPU | | | 11 of 68 |
| | STATISTICAL DOCUMENT | Page | |



Figure 3. Levothyroxine concentration vs. subject 3's time plot, on an arithmetic scale, post-dose of the test-drug, and reference-drug.



Figure 4. Levothyroxine concentration vs. subject 4's time plot, on an arithmetic scale, postdose of the test-drug and reference-drug.

| La | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|



Figure 5. Levothyroxine concentration vs. subject 5's time plot, on an arithmetic scale, postdose of the test-drug and reference-drug.



Figure 6. Levothyroxine concentration vs. subject 6's time plot, on an arithmetic scale, postdose of the test-drug, and reference-drug.

| ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|----------------------|---------|-------------|



Figure 7. Levothyroxine concentration vs. subject 7's time plot, on an arithmetic scale, postdose of the test-drug and reference-drug.



Figure 8. Levothyroxine concentration vs. subject 8's time plot, on an arithmetic scale, postdose of the test-drug and reference-drug.

| L | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|



Figure 9. Levothyroxine concentration vs. subject 9's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.



Figure 10. Levothyroxine concentration vs. subject 10's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.

| ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|----------------------|---------|-------------|



Figure 11. Levothyroxine concentration vs. subject 11's time plot, on an arithmetic scale, post-dose of the test-drug, and reference-drug.



Figure 12. Levothyroxine concentration vs. subject 12's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.

| · · | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|



Figure 13. Levothyroxine concentration vs. subject 13's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.



Figure 14. Levothyroxine concentration vs. subject 14's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.

| | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|
| PPD | | | 17 of 68 |
| | STATISTICAL DOCUMENT | Page | |



Figure 15. Levothyroxine concentration vs. subject 15's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.



Figure 16. Levothyroxine concentration vs. subject 17's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.

| · · | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|



Figure 17. Levothyroxine concentration vs. subject 18's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.



Figure 18. Levothyroxine concentration vs. subject 19's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.

| · · | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|



Figure 19. Levothyroxine concentration vs. subject 20's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.



Figure 20. Levothyroxine concentration vs. subject 22's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.

| La | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|



Figure 21. Levothyroxine concentration vs. subject 23's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.



Figure 22. Levothyroxine concentration vs. subject 24's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.

| L | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|



Figure 23. Levothyroxine concentration vs. subject 25's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.



post-dose of the test-drug and reference-drug.

| | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|
| PPD | | | 22 of 68 |
| | STATISTICAL DOCUMENT | Page | |



Figure 25. Levothyroxine concentration vs. subject 28's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.



| | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|
| PPD | ANALITICAL ONIT | Version | 1.0 |
| PPU | | _ | 23 of 68 |
| | STATISTICAL DOCUMENT | Page | |



Figure 27. Levothyroxine concentration vs. subject 30's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.



| L | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|



Figure 29. Levothyroxine concentration vs. subject 33's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.



Figure 30. Levothyroxine concentration vs. subject 34's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.

| | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|
| PPU | | | 25 of 68 |
| | STATISTICAL DOCUMENT | Page | |



Figure 31. Levothyroxine concentration vs. subject 35's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.



post-dose of the test-drug and reference-drug.

| ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|----------------------|---------|-------------|



Figure 33. Levothyroxine concentration vs. subject 37's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.



Figure 34. Levothyroxine concentration vs. subject 39's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.

| La | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|



Figure 35. Levothyroxine concentration vs. subject 41's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.



Figure 36. Levothyroxine concentration vs. subject 42's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.

| La | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|
| PPD | ANALI HOAL ONH | Version | 1.0 |



Figure 37. Levothyroxine concentration vs. subject 43's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.



Figure 38. Levothyroxine concentration vs. subject 44's time plot, on an arithmetic scale, post-dose of the test-drug and reference-drug.

| L | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|



Figure 39. Levothyroxine concentration vs. subject 1's time plot, on a logarithmic scale, postdose of the test-drug and reference-drug.



Figure 40. Levothyroxine concentration vs. subject 2's time plot, on a logarithmic scale, postdose of the test-drug and reference-drug.

| ANALYTICAL UNIT | Issue | 10-Mar-2020 | |
|-----------------|----------------------|-------------|----------|
| PPD | ANALT TICAL ONT | Version | 1.0 |



Figure 41. Levothyroxine concentration vs. subject 3's time plot, on a logarithmic scale, postdose of the test-drug and reference-drug.



Figure 42. Levothyroxine concentration vs. subject 4's time plot, on a logarithmic scale, post-dose of the test-drug and reference-drug.

| ANALYTICAL UNIT | Issue | 10-Mar-2020 | |
|-----------------|----------------------|-------------|----------|
| PPD | ANALTHCAL ONT | Version | 1.0 |



Figure 43. Levothyroxine concentration vs. subject 5's time plot, on a logarithmic scale, post-dose of the test-drug and reference-drug.



Figure 44. Levothyroxine concentration vs. subject 6's time plot, on a logarithmic scale, postdose of the test-drug and reference-drug.

| ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----------------|----------------------|-------------|



Figure 45. Levothyroxine concentration vs. subject 7's time plot, on a logarithmic scale, post-dose of the test-drug and reference-drug.



Figure 46. Levothyroxine concentration vs. subject 8's time plot, on a logarithmic scale, postdose of the test-drug and reference-drug.

| ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----------------|----------------------|-------------|



Figure 47. Levothyroxine concentration vs. subject 9's time plot, on a logarithmic scale, postdose of the test-drug and reference-drug.



Figure 48. Levothyroxine concentration vs. subject 10's time plot, on a logarithmic scale, post-dose of the test-drug and reference-drug.

| ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----------------|----------------------|-------------|



Figure 49. Levothyroxine concentration vs. subject 11's time plot, on a logarithmic scale, post-dose of the test-drug and reference-drug.



| L | ANALYTICAL UNIT | Issue 10-Mar-2020 | 10-Mar-2020 |
|-----|----------------------|-------------------|-------------|
| FFD | | | 35 of 68 |
| | STATISTICAL DOCUMENT | Page | |



Figure 51. Levothyroxine concentration vs. subject 13's time plot, on a logarithmic scale, post-dose of the test-drug and reference-drug.



post-dose of the test-drug and reference-drug.

| T <sub>0</sub> | ANALYTICAL UNIT | Issue 10-Mar-2020 | 10-Mar-2020 |
|----------------|----------------------|-------------------|-------------|
| PPD | ANALTHCAL ONT | Version | 1.0 |



Figure 53. Levothyroxine concentration vs. subject 15's time plot, on a logarithmic scale, post-dose of the test-drug and reference-drug.



Figure 54. Levothyroxine concentration vs. subject 17's time plot, on a logarithmic scale, post-dose of the test-drug and reference-drug.
| T <sub>a</sub> | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|----------------|----------------------|---------|-------------|
| PPD | | | 37 of 68 |
| | STATISTICAL DOCUMENT | Page | |



Figure 55. Levothyroxine concentration vs. subject 18's time plot, on a logarithmic scale, post-dose of the test-drug and reference-drug.



| La | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|



Figure 57. Levothyroxine concentration vs. subject 20's time plot, on a logarithmic scale, post-dose of the test-drug and reference-drug.



Figure 58. Levothyroxine concentration vs. subject 22's time plot, on a logarithmic scale, post-dose of the test-drug and reference-drug.

| La | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|



Figure 59. Levothyroxine concentration vs. subject 23's time plot, on a logarithmic scale, post-dose of the test-drug and reference-drug.



| T <sub>0</sub> | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|----------------|----------------------|---------|-------------|
| PPU | OTATIOTICAL DOCUMENT | _ | 40 of 68 |
| | STATISTICAL DOCUMENT | Page | |



Figure 61. Levothyroxine concentration vs. subject 25's time plot, on a logarithmic scale, post-dose of the test-drug and reference-drug.



Figure 62. Levothyroxine concentration vs. subject 27's time plot, on a logarithmic scale, post-dose of the test-drug and reference-drug.

| T <sub>a</sub> | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|----------------|----------------------|---------|-------------|



Figure 63. Levothyroxine concentration vs. subject 28's time plot, on a logarithmic scale, post-dose of the test-drug and reference-drug.



| L | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|



Figure 65. Levothyroxine concentration vs. subject 30's time plot, on a logarithmic scale, post-dose of the test-drug and reference-drug.



post-dose of the test-drug and reference-drug.

| L | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|



Figure 67. Levothyroxine concentration vs. subject 33's time plot, on a logarithmic scale, post-dose of the test-drug and reference-drug.



post-dose of the test-drug and reference-drug.

| | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|
| PPD | | | 44 of 68 |
| | STATISTICAL DOCUMENT | Page | |



Figure 69. Levothyroxine concentration vs. subject 35's time plot, on a logarithmic scale, post-dose of the test-drug and reference-drug.



Figure 70. Levothyroxine concentration vs. subject 36's time plot, on a logarithmic scale, post-dose of the test-drug and reference-drug.

| · · | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|
| PPD | STATISTICAL DOCUMENT | Page | 45 of 68 |



Figure 71. Levothyroxine concentration vs. subject 37's time plot, on a logarithmic scale, post-dose of the test-drug and reference-drug.



| L | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|



Figure 73. Levothyroxine concentration vs. subject 41's time plot, on a logarithmic scale, post-dose of the test-drug and reference-drug.



Figure 74. Levothyroxine concentration vs. subject 42's time plot, on a logarithmic scale, post-dose of the test-drug and reference-drug.

| L | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|



Figure 75. Levothyroxine concentration vs. subject 43's time plot, on a logarithmic scale, post-dose of the test-drug and reference-drug.



Figure 76. Levothyroxine concentration vs. subject 44's time plot, on a logarithmic scale, post-dose of the test-drug and reference-drug.

| T <sub>a</sub> | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|----------------|----------------------|---------|-------------|



Figure 77. Levothyroxine average concentration vs. time plot, on a logarithmic scale, postdose of the test-drug and reference-drug (standard deviation bars).



| L | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|

# 3.4. Descriptive Statistics of Biological Fluid Concentration Data as a Function of Time and Formulation

Table 7 shows the average values of the levothyroxine concentrations, as well as their descriptive statistics obtained from the assessed products.

Table 7. Descriptive statistics of the levothyroxine concentration in biological fluid, adjusted data. (N = 38).

| | | Eu | rtirox® approv | ved formulati | on | | | | Eutirox® test | formulation | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time | Arithmetic | | Minimum | Maximum | Standard | W.CV | Arithmetic | Modion | Minimum | Maximum | Standard | WCV. |
| | mean | Median | value | value | Deviation | %CV | mean | Median | value | value | Deviation | %CV |
| 0.00 | 0.43 | 0.00 | 0.00 | 3.49 | 0.91 | 211.46 | 0.41 | 0.00 | 0.00 | 3.11 | 0.75 | 182.21 |
| 0.50 | 3.58 | 3.14 | 0.00 | 12.68 | 3.14 | 87.72 | 6.59 | 4.65 | 0.00 | 22.49 | 6.46 | 98.09 |
| 1.00 | 23.86 | 22.53 | 0.00 | 81.95 | 16.39 | 68.69 | 29.13 | 30.19 | 0.00 | 62.72 | 16.78 | 57.58 |
| 1.50 | 39.59 | 41.38 | 0.00 | 90.27 | 17.95 | 45.33 | 43.35 | 46.42 | 0.00 | 82.41 | 19.33 | 44.59 |
| 2.00 | 46.48 | 49.19 | 12.87 | 85.98 | 16.63 | 35.78 | 48.45 | 51.49 | 9.21 | 86.16 | 18.42 | 38.02 |
| 2.50 | 51.84 | 53.27 | 18.87 | 100.38 | 16.92 | 32.63 | 53.05 | 52.79 | 11.89 | 91.74 | 18.00 | 33.94 |
| 3.00 | 54.48 | 54.53 | 22.85 | 121.16 | 19.08 | 35.02 | 54.23 | 53.83 | 15.13 | 105.75 | 18.98 | 35.00 |
| 3.25 | 55.88 | 56.65 | 24.02 | 82.14 | 13.14 | 23.52 | 53.03 | 52.77 | 10.93 | 97.25 | 18.28 | 34.47 |
| 3.50 | 56.22 | 54.54 | 34.94 | 83.03 | 13.00 | 23.12 | 53.37 | 55.44 | 12.35 | 97.45 | 17.20 | 32.22 |
| 3.75 | 55.64 | 56.30 | 32.34 | 82.19 | 12.38 | 22.24 | 54.08 | 51.83 | 18.55 | 98.59 | 17.86 | 33.03 |
| 4.00 | 54.98 | 52.93 | 30.05 | 96.39 | 13.77 | 25.04 | 52.41 | 52.51 | 23.36 | 101.74 | 16.14 | 30.80 |
| 4.25 | 60.10 | 59.40 | 32.89 | 98.33 | 13.35 | 22.21 | 56.98 | 54.82 | 33.26 | 104.57 | 14.16 | 24.85 |
| 4.50 | 56.09 | 53.03 | 40.83 | 89.28 | 12.97 | 23.13 | 54.34 | 50.13 | 26.93 | 94.09 | 14.40 | 26.51 |
| 4.75 | 52.84 | 52.50 | 27.92 | 90.42 | 14.42 | 27.29 | 52.99 | 51.87 | 29.62 | 96.22 | 14.52 | 27.40 |
| 5.00 | 52.17 | 50.76 | 26.94 | 86.81 | 14.27 | 27.35 | 51.94 | 48.73 | 29.99 | 97.71 | 15.15 | 29.17 |
| 5.50 | 51.04 | 49.65 | 23.02 | 85.70 | 14.26 | 27.93 | 48.76 | 48.10 | 24.59 | 95.00 | 13.12 | 26.91 |
| 6.00 | 48.49 | 45.49 | 30.45 | 79.63 | 11.81 | 24.36 | 47.56 | 46.96 | 12.65 | 96.72 | 14.70 | 30.90 |
| 6.50 | 45.99 | 43.82 | 27.96 | 77.27 | 11.81 | 25.69 | 44.12 | 41.46 | 20.77 | 80.81 | 12.35 | 27.99 |
| 8.00 | 46.90 | 48.07 | 24.96 | 68.79 | 11.09 | 23.64 | 44.37 | 41.54 | 6.44 | 76.82 | 13.43 | 30.27 |
| 10.00 | 40.04 | 39.40 | 17.75 | 68.89 | 10.69 | 26.70 | 37.67 | 37.10 | 12.78 | 63.24 | 11.33 | 30.09 |
| 12.00 | 37.67 | 36.37 | 18.83 | 64.91 | 11.19 | 29.70 | 36.95 | 37.23 | 13.72 | 74.36 | 10.93 | 29.58 |
| 24.00 | 36.31 | 37.62 | 15.52 | 57.99 | 9.64 | 26.54 | 35.13 | 34.49 | 19.77 | 52.40 | 8.20 | 23.34 |
| 36.00 | 32.42 | 29.63 | 10.97 | 58.18 | 10.86 | 33.50 | 31.91 | 32.69 | 0.00 | 56.25 | 10.63 | 33.32 |
| 48.00 | 29.49 | 29.16 | 14.56 | 55.61 | 9.20 | 31.20 | 27.87 | 27.44 | 6.82 | 41.12 | 8.26 | 29.63 |

| T <sub>a</sub> | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|----------------|----------------------|---------|-------------|

# 3.5. Pharmacokinetic Parameters 3.5.1. Individual Data and Descriptive Statistics of the Pharmacokinetic Parameters

The pharmacokinetic analysis was carried out by means of the non-compartmental analysis, using Phoenix® WinNonlin® Version 8.2 and real times, following the administration of levothyroxine 600  $\mu$ g (3 tablets of 200  $\mu$ g). Table 8 shows levothyroxine individual values and descriptive statistics used for determining bioequivalence statistics. The uncorrected pharmacokinetic parameters are presented in table A2.4

Table 8. Individual data and descriptive statistics for the levothyroxine pharmacokinetic parameters for adjusted data (C<sub>max</sub> in ng/mL, AUC<sub>0-t</sub> in ng\*h/mL and AUC<sub>0-∞</sub> in ng\*h/mL).

| | Peri | iod | | | C, | nax | | | AU | Coe | | | AUG | C <sub>0-m</sub> | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Volunteer | For | rm | Sequence | Fo | rm | | | Fo | rm | | | Fo | rm | | |
| | Α | В | | Α | В | B/A | Ln(B/A) | Α | В | B/A | Ln(B/A) | Α | В | B/A | Ln(B/A) |
| 1 | 2 | 1 | BA | 98.33 | 84.97 | 0.86 | -0.15 | 2689.21 | 1962.33 | 0.73 | -0.32 | 7629.83 | 3185.87 | 0.42 | -0.87 |
| 2 | 2 | 1 | BA | 59.08 | 59.26 | 1.00 | 0.00 | 1837.68 | 1370.21 | 0.75 | -0.29 | 11399.25 | 2354.71 | 0.21 | -1.58 |
| 3 | 2 | 1 | BA | 61.00 | 56.41 | 0.92 | -0.08 | 1226.05 | 1089.98 | 0.89 | -0.12 | 3779.67 | 3779.06 | 1.00 | 0.00 |
| 4 | 1 | 2 | AB | 67.12 | 63.95 | 0.95 | -0.05 | 1590.66 | 1566.01 | 0.98 | -0.02 | 3376.25 | 2805.99 | 0.83 | -0.19 |
| 5 | 1 | 2 | AB | 53.06 | 59.02 | 1.11 | 0.11 | 1278.88 | 1313.99 | 1.03 | 0.03 | 2779.56 | 4931.11 | 1.77 | 0.57 |
| 6 | 2 | 1 | BA | 64.49 | 48.64 | 0.75 | -0.28 | 1808.01 | 1158.58 | 0.64 | -0.45 | 4711.82 | 3048.40 | 0.65 | -0.44 |
| 7 | 1 | 2 | AB | 64.47 | 69.43 | 1.08 | 0.07 | 1613.07 | 1922.93 | 1.19 | 0.18 | 4049.63 | 7788.41 | 1.92 | 0.65 |
| 8 | 1 | 2 | AB | 64.72 | 66.18 | 1.02 | 0.02 | 1631.27 | 1868.76 | 1.15 | 0.14 | 2856.95 | 4471.12 | 1.56 | 0.45 |
| 9 | 1 | 2 | AB | 84.71 | 104.57 | 1.23 | 0.21 | 2039.40 | 2607.86 | 1.28 | 0.25 | 4687.59 | 4314.79 | 0.92 | -0.08 |
| 10 | 1 | 2 | AB | 81.77 | 97.25 | 1.19 | 0.17 | 1996.53 | 2646.91 | 1.33 | 0.28 | 3703.43 | 6718.92 | 1.81 | 0.60 |
| 11 | 1 | 2 | AB | 68.86 | 72.27 | 1.05 | 0.05 | 1819.05 | 2275.38 | 1.25 | 0.22 | 3550.37 | 4959.64 | 1.40 | 0.33 |
| 12 | 2 | 1 | BA | 69.82 | 69.15 | 0.99 | -0.01 | 1891.54 | 1974.42 | 1.04 | 0.04 | 4532.18 | 3117.89 | 0.69 | -0.37 |
| 13 | 1 | 2 | AB | 62.06 | 51.70 | 0.83 | -0.18 | 2001.99 | 1534.42 | 0.77 | -0.27 | 6086.19 | 7351.71 | 1.21 | 0.19 |
| 14 | 2 | 1 | BA | 69.84 | 68.12 | 0.98 | -0.03 | 1917.57 | 2269.15 | 1.18 | 0.17 | 4363.45 | 5362.42 | 1.23 | 0.21 |
| 15 | 2 | 1 | BA | 51.95 | 54.48 | 1.05 | 0.05 | 1200.24 | 1699.42 | 1.42 | 0.35 | 2732.81 | 7146.60 | 2.62 | 0.96 |
| 17 | 2 | 1 | BA | 66.14 | 68.33 | 1.03 | 0.03 | 1568.88 | 1626.36 | 1.04 | 0.04 | 1958.82 | 2041.21 | 1.04 | 0.04 |
| 18 | 1 | 2 | AB | 67.71 | 68.11 | 1.01 | 0.01 | 1843.99 | 1934.69 | 1.05 | 0.05 | 4232.42 | 5847.55 | 1.38 | 0.32 |
| 19 | 2 | 1 | BA | 73.11 | 56.02 | 0.77 | -0.27 | 2003.56 | 1500.57 | 0.75 | -0.29 | 4108.73 | 3382.13 | 0.82 | -0.19 |
| 20 | 1 | 2 | AB | 74.61 | 60.44 | 0.81 | -0.21 | 2335.69 | 1506.84 | 0.65 | -0.44 | 5650.88 | 3602.09 | 0.64 | -0.45 |
| 22 | 2 | 1 | BA | 50.81 | 43.65 | 0.86 | -0.15 | 1094.52 | 1347.80 | 1.23 | 0.21 | 2115.19 | 4591.17 | 2.17 | 0.77 |
| 23 | 2 | 1 | BA | 50.16 | 73.24 | 1.46 | 0.38 | 1288.89 | 1856.73 | 1.44 | 0.37 | 2389.96 | 6212.32 | 2.60 | 0.96 |
| 24 | 1 | 2 | AB | 75.62 | 60.54 | 0.80 | -0.22 | 1586.03 | 1327.55 | 0.84 | -0.18 | 2452.72 | 3747.07 | 1.53 | 0.42 |
| 25 | 2 | 1 | BA | 59.68 | 62.69 | 1.05 | 0.05 | 1371.46 | 1872.58 | 1.37 | 0.31 | 3601.75 | 3002.55 | 0.83 | -0.18 |
| 27 | 1 | 2 | AB | 48.06 | 52.34 | 1.09 | 0.09 | 1393.96 | 1342.50 | 0.96 | -0.04 | 3106.51 | 1840.81 | 0.59 | -0.52 |
| 28 | 1 | 2 | AB | 121.16 | 105.75 | 0.87 | -0.14 | 2365.84 | 1777.47 | 0.75 | -0.29 | 6969.94 | 2831.05 | 0.41 | -0.90 |
| 29 | 1 | 2 | AB | 65.35 | 60.17 | 0.92 | -0.08 | 1614.49 | 1100.34 | 0.68 | -0.38 | 2346.45 | 1261.22 | 0.54 | -0.62 |
| 30 | 2 | 1 | BA | 68.88 | 71.68 | 1.04 | 0.04 | 2047.90 | 1855.80 | 0.91 | -0.10 | 7698.37 | 7971.33 | 1.04 | 0.03 |
| 31 | 2 | 1 | BA | 49.54 | 62.01 | 1.25 | 0.22 | 984.41 | 1681.30 | 1.71 | 0.54 | 1682.68 | 3464.68 | 2.06 | 0.72 |
| 33 | 2 | 1 | BA | 86.93 | 82.18 | 0.95 | -0.06 | 2777.76 | 1965.99 | 0.71 | -0.35 | 9404.14 | 4083.85 | 0.43 | -0.83 |
| 34 | 1 | 2 | AB | 60.92 | 70.24 | 1.15 | 0.14 | 1423.86 | 1469.25 | 1.03 | 0.03 | 3357.06 | 2278.33 | 0.68 | -0.39 |
| 35 | 1 | 2 | AB | 59.46 | 52.07 | 0.88 | -0.13 | 1828.60 | 1575.38 | 0.86 | -0.15 | 5260.60 | 8928.32 | 1.70 | 0.53 |
| 36 | 1 | 2 | AB | 74.82 | 70.08 | 0.94 | -0.07 | 1468.93 | 1750.43 | 1.19 | 0.18 | 2996.07 | 4872.32 | 1.63 | 0.49 |
| 37 | 1 | 2 | AB | 60.30 | 68.30 | 1.13 | 0.12 | 1801.46 | 2017.01 | 1.12 | 0.11 | 4862.37 | 9642.45 | 1.98 | 0.68 |
| 39 | 1 | 2 | AB | 100.38 | 94.09 | 0.94 | -0.06 | 2746.26 | 2212.77 | 0.81 | -0.22 | 6141.94 | 4801.43 | 0.78 | -0.25 |
| 41 | 1 | 2 | AB | 72.78 | 79.08 | 1.09 | 0.08 | 1795.04 | 1564.48 | 0.87 | -0.14 | 4528.22 | 2357.15 | 0.52 | -0.65 |
| 42 | 2 | 1 | BA | 44.51 | 33.98 | 0.76 | -0.27 | 1250.47 | 1221.60 | 0.98 | -0.02 | 4821.73 | 8527.56 | 1.77 | 0.57 |
| 43 | 2 | 1 | BA | 51.13 | 56.81 | 1.11 | 0.11 | 1529.05 | 1337.85 | 0.87 | -0.13 | 3297.62 | 3246.45 | 0.98 | -0.02 |
| 44 | 2 | 1 | BA | 51.87 | 47.59 | 0.92 | -0.09 | 1406.46 | 1262.19 | 0.90 | -0.11 | 8009.03 | 3183.88 | 0.40 | -0.92 |
| | N | | | 38.00 | 38.00 | 38.00 | 38.00 | 38.00 | 38.00 | 38.00 | 38.00 | 38.00 | 38.00 | 38.00 | 38.00 |
| Ge | ometri | ic Mea | in | 65.66 | 64.69 | 0.99 | NA | 1687.14 | 1651.82 | 0.98 | NA | 4083.25 | 4088.43 | 1.00 | NA |
| Ari | thmeti | ic Mea | in | 67.24 | 66.44 | 1.00 | -0.01 | 1738.65 | 1693.89 | 1.01 | -0.02 | 4506.11 | 4554.04 | 1.18 | 0.00 |
| Stan | dard D | eviati | ion | 15.77 | 15.77 | 0.15 | 0.15 | 438.93 | 389.50 | 0.25 | 0.25 | 2151.01 | 2145.52 | 0.64 | 0.61 |
| | %C | ٧ | | 23.45 | 23.73 | 15.13 | -1006.61 | 25.25 | 22.99 | 25.03 | -1161.73 | 47.74 | 47.11 | 54.46 | 47802.1 |
| M | inimun | n Valu | e | 44.51 | 33.98 | 0.75 | -0.28 | 984.41 | 1089.98 | 0.64 | -0.45 | 1682.68 | 1261.22 | 0.21 | -1.58 |
| | Medi | ian | | 65.04 | 65.07 | 1.00 | 0.00 | 1713.16 | 1653.83 | 0.98 | -0.02 | 4079.18 | 3931.45 | 1.02 | 0.02 |
| 14 | aximun | n Valu | in a | 121.16 | 105.75 | 1.46 | 0.38 | 2777.76 | 2646.91 | 1.71 | 0.54 | 11399.25 | 9642.45 | 2.62 | 0.96 |

| L | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|
| PPD | ANALI HOAL ONI | Version | 1.0 |

Table 9 shows the average results for the levothyroxine pharmacokinetic parameters. There, it can be seen  $t_{\text{max}}$  values of 3.41 h and 3.51 h, and  $C_{\text{max}}$  values of 67.24 ng/mL, and 66.44 ng/mL for the reference and test drugs, respectively. Based on these results, it can be inferred that there are no differences in the extent and rate which levothyroxine needs for reaching the circulation.

On the other hand, average AUC<sub>0-t</sub> was 1738.65  $\mu$ g\*h/mL and 1693.89 ng\*h/mL for the reference and test drugs, respectively. AUC<sub>0-∞</sub> is only shown for informative purposes, since their values result in a greater extrapolation than 20%. Values were 4506.11 ng\*h/mL and 4554.04 ng\*h/mL for the reference and test drugs, respectively. Based on these values, it can be seen that the drug's bioavailability for both formulations does not show differences.

Table 9. Levothyroxine Pharmacokinetic Parameters Results, adjusted data.

| | | | | Fo | rm | | | |
|---|---|---|---|---|---|---|---|---|
| Mariahla | E | utirox® appro | ved formulation | | | Eutirox® test formulation (B) | | |
| Variable | N | Arithmetic<br>Mean | Standard<br>Deviation | %CV | N | Arithmetic<br>Mean | Standard<br>Deviation | %CV |
| Extrapolated AUC (%) | 38.00 | 56.70 | 12.83 | 22.62 | 38.00 | 55.87 | 18.07 | 32.35 |
| AUC <sub>0-∞</sub> (ng*h/mL) | 38.00 | 4506.11 | 2151.01 | 47.74 | 38.00 | 4554.04 | 2145.52 | 47.11 |
| AUC <sub>0-t</sub> (ng*h/mL) | 38.00 | 1738.65 | 438.93 | 25.25 | 38.00 | 1693.89 | 389.50 | 22.99 |
| CI/F (mL/h) | 38.00 | 161.15 | 69.74 | 43.28 | 38.00 | 164.22 | 83.82 | 51.04 |
| C <sub>max</sub> (ng/mL) | 38.00 | 67.24 | 15.77 | 23.45 | 38.00 | 66.44 | 15.77 | 23.73 |
| t 1/2 (h) | 38.00 | 61.60 | 32.44 | 52.67 | 38.00 | 65.16 | 37.04 | 56.85 |
| Kel (1/h) | 38.00 | 0.01 | 0.01 | 46.76 | 38.00 | 0.01 | 0.01 | 57.13 |
| TMR (h) | 38.00 | 92.27 | 45.99 | 49.85 | 38.00 | 97.32 | 54.70 | 56.21 |
| T <sub>lag</sub> (h) | 38.00 | 0.11 | 0.21 | 196.25 | 38.00 | 0.00 | 0.00 | NA |
| T <sub>max</sub> (h) | 38.00 | 3.41 | 0.99 | 29.07 | 38.00 | 3.51 | 1.17 | 33.46 |
| Vd/F (L) | 38.00 | 12118.29 | 3202.28 | 26.43 | 38.00 | 12182.01 | 2720.22 | 22.33 |

NA: Not applicable

Table 10 shows the box and whiskers plots for the parameters used for assessing the levothyroxine absorption rate and bioavailability.

| | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-----------------|
| PPU | | | 52 <b>of</b> 68 |
| | STATISTICAL DOCUMENT | Page | |

Table 10. Box and Whiskers Plot for the Levothyroxine Pharmacokinetic Parameters



a) t<sub>max</sub> parameter plot, b) C<sub>max</sub> parameter plot C) AUC<sub>0-t</sub> parameter plot; and d) AUC<sub>0-∞</sub> parameter plot Form A and form B correspond to the reference and test formulations, respectively.

Graphically, it is confirmed that there are no differences in the absorption rate or in the bioavailability between both formulations since those representations are very similar to each other.

| <b>L</b> a | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|------------|----------------------|---------|-------------|

### 4. Variance Analysis (ANOVA)

The analysis of variance was made considering all data obtained in the levothyroxine pharmacokinetic analysis, under the same statistical considerations and the same general linear model previously described for estimating the F statistical value, based on the variance results of the fixed and random factors or effects in each of the pharmacokinetic parameters requested for establishing the bioequivalence. Results of the analysis of variance for the assessed parameters C<sub>max</sub>, AUC<sub>0-t</sub>, and AUC<sub>0-∞</sub> for levothyroxine are shown in Table 11.

Table 11. ANOVA table for the analysis of the levothyroxine logarithmically-transformed pharmacokinetic parameters, for adjusted data (Ln).

| Assessed<br>Variable | Source of Variation | Degrees of<br>Freedom | Square Sum | Squared Means | F Value | P Value | Criterion (P > 0.05) |
|---|---|---|---|---|---|---|---|
| Ln(C <sub>max</sub> ) | Sequence | 1 | 0.08 | 0.08 | 0.84 | 0.36 | Pass |
| Ln(C <sub>max</sub> ) | Sequence*Volunteer | 36 | 3.28 | 0.09 | | | Not applicable |
| Ln(C <sub>max</sub> ) | Form | 1 | 0.00 | 0.00 | 0.36 | 0.55 | Pass |
| $Ln(C_{max})$ | Period | 1 | 1.92x10 <sup>-7</sup> | 1.92x10 <sup>-7</sup> | 1.69x 10 <sup>-5</sup> | 1.00 | Pass |
| $Ln(C_{max})$ | Error | 36 | 0.41 | 0.01 | | | Not applicable |
| Ln(AUC₀+) | Sequence | 1 | 0.01 | 0.01 | 0.15 | 0.70 | Pass |
| Ln(AUC₀+) | Sequence*Volunteer | 36 | 3.05 | 0.08 | | | Not applicable |
| Ln(AUC₀+) | Form | 1 | 0.01 | 0.01 | 0.29 | 0.59 | Pass |
| Ln(AUC₀+) | Period | 1 | 0.07 | 0.07 | 2.45 | 0.13 | Pass |
| Ln(AUC₀+) | Error | 36 | 1.05 | 0.03 | | | Not applicable |
| Ln(AUC₀∞) | Sequence | 1 | 0.03 | 0.03 | 0.11 | 0.74 | Pass |
| Ln(AUC₀∞) | Sequence*Volunteer | 36 | 8.90 | 0.25 | | | Not applicable |
| Ln(AUC <sub>0∞</sub> ) | Form | 1 | 3.06x 10 <sup>-5</sup> | 3.06x 10 <sup>-5</sup> | 0.00 | 0.99 | Pass |
| Ln(AUC <sub>∪∞</sub> ) | Period | 1 | 0.50 | 0.50 | 2.85 | 0.10 | Pass |
| Ln(AUC <sub>0∞</sub> ) | Error | 36 | 6.30 | 0.18 | | | Not applicable |

Regarding the analysis of variance for the logarithmically-transformed pharmacokinetic data, no statistical significance was seen in all sources of variations used for the parameters which determine the bioequivalence (C<sub>max</sub> and AUC<sub>0-t</sub>). Therefore, the 90 % confidence interval was calculated.

| <b>L</b> a | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|------------|----------------------|---------|-------------|

## 5. Study Variability

Coefficients of variation obtained in this study for levothyroxine by means of the crossover 2 x 2 design are shown in Table 12.

Table 12. Inter- and Intra-subject Coefficients of Variation Obtained for Levothyroxine adjusted data

| Pharmacokinetic Parameter | Inter-subject<br>CV | Intra-subject<br>CV |
|---------------------------|---------------------|---------------------|
| C <sub>max</sub> | 20.18 | 10.66 |
| AUC <sub>0-t</sub> | 16.79 | 17.17 |
| AUC <sub>0-∞</sub> | 19.16 | 43.74 |

#### 6. Pharmacokinetic Parameters Outliers Identification

Outliers analysis was made using the intra-subject studentized residuals determination as per the Mexican Official Standard, NOM-177-SSA1-2013, which specifies that the possible outliers are those exceeding the ± 2 studentized-residuals criterion. Table 13 shows the values exceeding this limit, meanwhile figures 79, 80, and 81 show the studentized residual plots vs. the logarithm for the levothyroxine assessed pharmacokinetic parameter.

Table 13. Subjects exceeding the ± 2 levothyroxine studentized residuals criterion.

| Pharmacokinetic<br>Parameter | Subject | Studentized Residual<br>Value |
|------------------------------|---------|-------------------------------|
| LnCmax | 23 | ± 2.65 |
| LnAUC <sub>0-t</sub> | 31 | ± 2.09 |
| LnAUC₀∞ | 2 | ± 2.43 |

| ANALYTICAL LINIT | Issue | 10-Mar-2020 |
|---|---|---|
| ANALITICAL ONIT | Version | 1.0 |
| | | 55 of 68 |
| STATISTICAL DOCUMENT | Page | |
| | ANALYTICAL UNIT STATISTICAL DOCUMENT | ANALYTICAL UNIT Version |



Figure 79. Studentized Residuals Plot for the Levothyroxine Intra-subject Pharmacokinetic Parameter Ln C<sub>max</sub>.



Figure 80. Studentized Residuals Plot for the Levothyroxine Intra-subject Pharmacokinetic Parameter AUC<sub>0-t</sub>.

| T <sub>0</sub> | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|----------------|----------------------|---------|-------------|



Figure 81. Studentized Residuals Plot for the Levothyroxine Intra-subject Pharmacokinetic Parameter AUC<sub>0-∞</sub>.

As seen in Table 13 and the figures shown above, subjects 2, 23, and 31 were found as outliers in this study since they exceeded the ± 2 studentized residuals.

As stated in the current national standards, a statistical analysis was made removing subjects 2, 23, and 31. As the results of the confidence intervals do not change, they are not considered influencing-outliers.

As per the current national standards, the Clinical and the Analytical Units jointly with Quality Assurance conducted the appropriate research. The results of this research showed that there were no events that render questionable the results obtained. Therefore, there is no scientific reason to justify the removal of subjects 2, 23, and 31 from the analysis. Therefore, results shown in this report include all subjects who were assessed.

| L | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|
| PPD | ANALI TICAL ONT | Version | 1.0 |

#### 7. Bioequivalence Statistics

Table 14 shows the results of the bioequivalence statistics for the levothyroxine logarithmically-transformed pharmacokinetic data.

Table 14. Statistics of the Levothyroxine Bioequivalence Determination for adjusted value.

| Parameter | 90 % Co | onfidence | | mann's<br>d-side t | Power | Acceptance | Meets<br>the |
|---|---|---|---|---|---|---|---|
| rarameter | Inte | erval | P < 80 % | P<br>> 125 % | rowei | Criterion | Criterion |
| LnC <sub>max</sub> | 94.55 102.68 | | 0.00 | 0.00 | 100.00 | (80-125) | YES |
| LnAUC <sub>0-t</sub> | 91.34 | 104.26 | 0.00 | 0.00 | 99.98 | (80-125) | YES |

As established in the Mexican Official Standard, NOM-177-SSA1-2013, the parameters to establish the conclusion about the possible bioequivalence of the products are  $C_{\text{max}}$  as a rate of absorption indicator and the AUC as the amount absorbed indicator.

The confidence interval for parameters  $C_{\text{max}}$  and  $AUC_{0-t}$  for establishing bioequivalence are within the established acceptance criteria (80 % to 125 %). Therefore, it is shown that there are no statistically significant differences in the absorption rate or in the drug's bioavailability. Even though the  $AUC_{0-\infty}$  is also within the bioequivalence limits, bioequivalence is established only with the results of  $C_{\text{max}}$  and  $AUC_{0-t}$ .

#### 8. Statistical Plan Deviation

None

#### 9. Discussion and Conclusion

The 90 % confidence intervals for C<sub>max</sub> and AUC<sub>0-t</sub> are contained in the acceptance region for bioequivalence, thus showing that the test formulation has an absorption rate and bioavailability that is equivalent to the one of the reference formulation.

As per the results obtained, it is concluded that the test drug "Eutirox®, new formulation" is bioequivalent to the reference drug "Eutirox®, the approved formulation".

#### 10. Annexes

Annex 1. Quality Assurance Report

Annex 2. Statistical information on unadjusted data per baseline levels.



**Annex 3**. Statistical information with all subjects, including a greater than 5% predose concentration.

Table A2.1 Table of individual concentrations corresponding to unadjusted levothyroxine (reference drug [A]). N = 43 subjects.

| | | | | | | | | | | | | | | Ti | ne | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Form | Volunteer | -0.50 | -0.25 | 0.00 | 0.50 | 1.00 | 1.50 | 2.00 | 2.50 | 3.00 | 3.25 | 3.50 | 3.75 | 4.00 | 4.25 | 4.50 | 4.75 | 5.00 | 5.50 | 6.00 | 6.50 | 8.00 | 10.00 | 12.00 | 24.00 | 36.00 | 48.00 |
| A | 1 | 51.32 | 64.16 | 53.26 | 4734 | 74.32 | 82.00 | 89.87 | 115.60 | 129.31 | 133.43 | 139.27 | 130.22 | 152.63 | 154.58 | 145.53 | 145.66 | 143.06 | 135.60 | 126.33 | 129.01 | 123.03 | 115.01 | 120.74 | 114.24 | 106.52 | 102.69 |
| Â | 2 | 81.52 | 81.75 | 83.05 | 85.21 | 101.35 | 115.81 | 124.86 | 127.71 | 128.42 | 136.55 | 134.A7 | 133.39 | 131.35 | 137.26 | 135.73 | 131.66 | 141.18 | 127.61 | 126.72 | 126.73 | 128.01 | 126.24 | 120.12 | 116.70 | 120.24 | 121.73 |
| A | 3 | 67.24 | 59.78 | 63.57 | 68.93 | 108.98 | 118.62 | 124.53 | 108.72 | 103.61 | 116.27 | 99.75 | 95.87 | 104.50 | 107.27 | 105.89 | 98.64 | 94.88 | 96.45 | 96.40 | 103.76 | 92.79 | 86.63 | 90.57 | 86.16 | 86.42 | 83.29 |
| A | 4 | 77.82 | 77.88 | 78.21 | 80.19 | 93.71 | 117.34 | 133.48 | 134.48 | 137.25 | 130.36 | 129.67 | 145.08 | 127.82 | 14038 | 137.09 | 125.25 | 126.62 | 129.16 | 119.01 | 123.52 | 125.37 | 115.80 | 116.95 | 108.11 | 107.03 | 101.07 |
| _ ^ | 5 | 81.33 | 75.34 | 76.83 | 79.14 | 100.51 | 110.35 | 114.52 | 115.47 | 130.89 | 123.34 | 130.00 | 124.95 | 129.61 | 129.51 | 130.03 | 126.29 | 124.27 | 126.22 | 119.11 | 112.70 | 111.82 | 110.51 | 104.11 | 102.93 | 97.25 | 105.84 |
| A | 6 | 54.46 | 57.33 | 54.72 | 57.63 | 59.66 | 77.05 | 105.41 | 119.99 | 118.56 | 112.95 | 113.34 | 114.36 | 105.48 | 113.16 | 106.90 | 111.40 | 108.78 | 108.75 | 108.39 | 110.95 | 109.41 | 99.56 | 98.27 | 92.30 | 88.21 | 84.47 |
| A | 7 | ថាជា | 57.02 | 53.83 | 62.55 | 76.01 | 87.55 | 89.50 | 93.95 | 117.19 | 107.74 | 113.89 | 123.98 | 115.72 | 122.98 | 108.95 | 112.95 | 100.80 | 99.79 | 102.82 | 101.27 | 112.66 | 92.70 | 87.22 | 97.94 | 88.35 | 89.99 |
| A | 8 | 76.72 | 68.81 | 67.61 | 74.08 | 102.10 | 115.11 | 129.39 | 135.77 | 128.13 | 134.38 | 120.79 | 129.39 | 131.45 | 131.27 | 128.83 | 126.25 | 132.74 | 125.79 | 132.44 | 118.29 | 122.15 | 116.15 | 110.56 | 103.45 | 95.93 | 94.37 |
| A | 9 | 90.07 | 85.62 | 71.38 | 89.50 | 93.89 | 97.98 | 95.22 | 101.62 | 109.01 | 130.24 | 136.36 | 147.11 | 142.34 | 159.70 | 159.21 | 167.06 | 162.79 | 153.70 | 153.94 | 144.65 | 142.75 | 131.91 | 121.68 | 128.59 | 119.94 | 121.15 |
| A | 10 | 81.37 | 78.12 | 75.32 | 72.70 | 80.13 | 114.61 | 130.46 | 136.57 | 141.05 | 149.64 | 148.31 | 135.02 | 153.11 | 157.35 | 153.84 | 160.04 | 139.45 | 153.09 | 141.98 | 136.69 | 141.07 | 133.92 | 127.26 | 119.63 | 109.91 | 109.09 |
| _ | - | | | | | | | | - | | | - | | | | - | | | | 131.25 | - | | | | | | |
| A | 11 | 87.13 | 74.20 | 77.05 | 75.73 | 94.21 | 107.00 | 148.32 | 119.95 | 131.84 | 134.97<br>133.18 | 130.97 | 135.31 | 140.88 | 140.22 | 144.44 | 139.12 | 138.12 | 138.05 | | 121.22 | 119.01 | 115.98<br>116.84 | 110.06 | 119.64 | 122.81<br>104.30 | 105.08 |
| A | 12<br>13 | 72.69<br>69.17 | 71.52<br>64.00 | 71.11<br>53.70 | 77.96<br>69.42 | 98.16<br>91.53 | 122.07<br>122.01 | 126.51<br>108.78 | 134.78<br>124.35 | 141.60<br>123.06 | 123.13 | 135.04<br>120.50 | 136.97<br>113.14 | 131.79<br>103.04 | 137.53<br>123.08 | 128.60<br>116.04 | 123.03<br>116.66 | 124.72<br>112.62 | 127.30<br>117.57 | 126.13<br>114.93 | 119.61<br>103.88 | 128.87<br>110.33 | 109.33 | 114.47<br>98.19 | 112.03<br>104.72 | 106.01 | 101.26<br>96.85 |
| _ | 14 | 66.40 | 64.46 | 67.30 | 69.39 | | 109.45 | 115.05 | | 120.95 | 129.65 | 123.37 | 125.50 | 128.21 | 12921 | 122.93 | 135.90 | 127.86 | 121.05 | 124.71 | 121.83 | 124.99 | 95.93 | 114.97 | 106.90 | 98.05 | 97.69 |
| A | | | | | ***** | 90.05 | | | 127.43 | | | | - | - | | | | | | | | - | | | | | _ |
| A | 15 | 90.13 | 88.14 | 89.45 | 83.99 | 94.68 | 85.71 | 102.53 | 114.34 | 112.09 | 120.03 | 132.47 | 130.51 | 126.00 | 130.07 | 133.38 | 129.75 | 141.19 | 132.04 | 128.44 | 123.44 | 120.72 | 131.03 | 126.07 | 112.29 | 105.00 | 114.73 |
| A | 16 | 83.94 | 84.37 | 75.45 | 89.25 | 107.94 | 11437 | 116.48<br>108.80 | 136.92 | 138.13 | 147.32<br>144.25 | 148.33<br>138.54 | 142.36<br>134.74 | 143.14 | 130.90<br>146.00 | 131.16<br>129.90 | 140.11 | 130.18 | 141.67 | 136.26 | 134.26<br>138.55 | 118.85 | 127.73 | 117.61<br>124.94 | 111.35 | 101.44 | 111.14 |
| A | 17 | 90.72 | 78.61 | 82.18 | 88.62 | 95.31 | 98.43 | | 125.95 | 149.98 | | | | | - | - | 136.14 | | 134.05 | 133.04 | | 138.21 | | | | 107.72 | 98.56 |
| A | 18 | 55.88 | 56.60 | 55.98 | 58.28 | 90.14 | 100.60 | 108.28 | 114.30 | 119.96 | 117.66 | 117.09 | 123.86 | 119.22 | 117.97 | 114.85 | 112.36 | 111.33 | 114.29 | 113.06 | 104.01 | 104.99 | 98.53 | 101.72 | 95.30 | 85.84 | 86.11 |
| A | 19<br>20 | 61.49 | 57.91 | 59.83 | 64.08 | 103.32<br>110.28 | 111.68 | 109.11<br>146.54 | 119.26 | 119.94 | 117.90 | 124.72 | 120.32 | 109.45 | 132.85 | 114.74 | 112.44 | 110.92<br>143.04 | 114.84 | 102.54 | 105.61<br>132.34 | 109.26 | 99.10<br>124.74 | 98.98<br>119.89 | 109.84<br>124.37 | 94.74<br>124.86 | 93.74<br>113.26 |
| A | | 75.47 | 76.86 | 73.99 | 81.76 | | | | 141.91 | 150.00 | - | 150.05 | 143.53 | 143.56 | 143.41 | 139.68 | 139.00 | | 142.52 | | | 136.40 | - | | | | $\overline{}$ |
| A | 21 | 65.09 | 61.09 | 62.88 | 66.01 | 90.15 | 119.37 | 116.48 | 124.02 | 131.63 | 127.98 | 125.34 | 125.89 | 131.96 | 128.32 | 129.01 | 123.91 | 121.29 | 120.48 | 106.06 | 112.01 | 117.89 | 101.83 | 98.64 | 103.30 | 97.94 | 95.55 |
| A | 22 | 73.63 | 68.17 | 67.24 | 65.19 | 75.16 | 79.88 | 83.11 | 88.55 | 9451 | 93.70 | 104.63 | 105.31 | 99.73 | 102.57 | 120.49 | 97.61 | 96.62 | 100.01 | 100.76 | 100.39 | 94.64 | 101.36 | 94.47 | 93.85 | 92.80 | 84.24 |
| A | 23 | 86.59 | 82.82 | 81.95 | 85.82 | 120.76 | 131.76 | 130.09 | 133.02 | 131.71 | 132.03 | 128.58 | 133.94 | 129.48 | 132.67 | 128.83 | 121.14 | 128.11 | 124.50 | 121.61 | 118.17 | 120.06 | 112.58 | 105.52 | 109.04 | 110.66 | 102.79 |
| A | 24 | 81.23 | 79.76 | 73.25 | 77.61 | 101.32 | 123.26 | 131.98 | 153.70 | 144.82 | 141.53 | 149.44 | 147.95 | 143.23 | 145.02 | 133.19 | 131.51 | 127.33 | 133.34 | 124.77 | 119.40 | 119.70 | 112.70 | 113.36 | 118.07 | 100.42 | 97.10 |
| A | 25 | 70.50 | 69.32 | 66.64 | 60.18 | 101.03 | 122.78 | 116.76 | 122.70 | 97.82 | 112.19 | 106.21 | 106.27 | 110.27 | 128.50 | 110.20 | 114.63 | 104.56 | 111.51 | 112.69 | 108.85 | 107.58 | 98.64 | 95.63 | 93.55 | 95.77 | 95.40 |
| A | 26 | 86.68 | 84.43 | 90.53 | 91.62 | 97.52 | 114.25 | 125.07 | 136.68 | 128.03 | 133.73 | 123.83 | 129.89 | 121.68 | 126.90 | 122.89 | 118.13 | 123.50 | 130.36 | 122.33 | 129.23 | 138.86 | 124.62 | 120.93 | 123.66 | 121.56 | 112.67 |
| A | 27 | 80.58 | 78.26 | 80.40 | 79.25 | 97.06 | 114.25 | 121.59 | 122.69 | 127.81 | 126.64 | 124.66 | 126.35 | 122.26 | 127.08 | 120.57 | 113.14 | 116.23 | 121.86 | 121.99 | 119.53 | 117.47 | 115.83 | 110.33 | 109.58 | 103.53 | 103.45 |
| A | 28 | 55.23 | 53.72 | 38.94 | 55.06 | 64.88 | 97.02 | 111.24 | 118.04 | 170.46 | 114.59 | 129.32 | 121.27 | 117.86 | 106.81 | 113.21 | 102.11 | 126.61 | 95.42 | 103.62 | 105.32 | 101.94 | 100.94 | 101.29 | 90.74 | 105.57 | 90.47 |
| A | 29 | 78.49 | 77.86 | 79.29 | 91.23 | 90.18 | 110,44 | 135.51 | 143.90 | 117.89 | 134.41 | 132.59 | 120.22 | 133.59 | 131.73 | 128.79 | 125.34 | 120.48 | 121.39 | 115.51 | 114.62 | 127.75 | 114.76 | 110.25 | 119.73 | 106.76 | 99.36 |
| A | 30 | 58.94 | 51.97 | 57.95 | 61.10 | 80.58 | 90.20 | 85.45 | 108.69 | 88.78 | 125.17 | 111.35 | 120.01 | 109.37 | 11438 | 114.11 | 109.03 | 107.81 | 105.38 | 99.64 | 96.50 | 104.52 | 99.03 | 98.30 | 96.57 | 105.05 | 93.96 |
| A | 31 | 77.90 | 70.91 | 73.73 | 78.75 | 83.48 | 109.13 | 109.14 | 119.30 | 113.83 | 115.17 | 113.51 | 114.17 | 112.61 | 119.20 | 123.72 | 122.28 | 110.27 | 97.20 | 104.63 | 105.89 | 107.08 | 91.93 | 93.01 | 101.49 | 85.15 | 89.19 |
| A | 32 | 71.01 | 70.48 | 75.52 | 78.92 | 122.73 | 125.80 | 133.37 | 115.90 | 111.88 | 110.41 | 112.27 | 116.95 | 108.88 | 11437 | 109.29 | 106.88 | 108.02 | 111.72 | 105.59 | 106.85 | 107.24 | 111.29 | 97.39 | 102.59 | 103.19 | 103.18 |
| A | 33 | 70.27 | 66.60 | 73.34 | 78.64 | 107.64 | 11533 | 127.62 | 145.42 | 141.58 | 147.96 | 152.33 | 346.97 | 149.73 | 157.00 | 155.63 | 143.67 | 151.13 | 155.63 | 135.30 | 143.33 | 134.14 | 129.48 | 134.38 | 120.80 | 128.25 | 125.68 |
| A | 34 | 9631 | 85.91 | 87.45 | 88.16 | 99.06 | 102.42 | 112.30 | 115.50 | 130.11 | 138.80 | 150.81 | 137.51 | 138.48 | 147.39 | 133.14 | 134.42 | 128.36 | 132.29 | 126.84 | 117.85 | 130.07 | 121.71 | 120.29 | 126.26 | 112.37 | 116.33 |
| A | 35 | 80.06 | 74.32 | 75.30 | 79.74 | 115.43 | 135.73 | 136.03 | 130.95 | 130.43 | 125.37 | 122.A1 | 122.43 | 122.61 | 130.75 | 120.66 | 108.04 | 119.69 | 122.23 | 118.35 | 119.58 | 123.59 | 124.62 | 110.68 | 116.14 | 113.08 | 108.27 |
| A | 36 | 89.46 | 84.72 | 92.32 | 93.70 | 139.86 | 151.02 | 145.62 | 140.86 | 154.16 | 163.65 | 150.16 | 153.67 | 145.92 | 147.95 | 141.26 | 143.00 | 140.37 | 140.48 | 135.19 | 134.36 | 129.85 | 130.86 | 124.22 | 104.35 | 118.41 | 119.17 |
| A | 37 | 79.45 | 75.66 | 76.18 | 75.75 | 113.46 | 124.32 | 137.40 | 132.15 | 131.25 | 134.88 | 136.69 | 132.63 | 129.88 | 131.70 | 129.45 | 125.04 | 126.53 | 130.15 | 130.61 | 124.54 | 125.19 | 115.87 | 119.11 | 11331 | 110.65 | 106.45 |
| A | 39 | 76.83 | 71.87 | 78.42 | 83.69 | 157.65 | 165.98 | 161.69 | 176.09 | 162.49 | 157.84 | 154.76 | 157.89 | 158.87 | 164.76 | 162.43 | 154.43 | 149.15 | 161.A1 | 155.34 | 152.98 | 144.49 | 144.60 | 140.61 | 127.69 | 123.18 | 124.82 |
| A | 40 | 75.00 | 71.11 | 87.64 | 83.77 | 97.16 | 108.84 | 116.77 | 151.08 | 154.63 | 158.86 | 159.19 | 163.10 | 162.15 | 168.47 | 165.46 | 161.38 | 164.72 | 142.87 | 164.27 | 157.78 | 157.87 | 148.44 | 144.12 | 126.08 | 127.21 | 112.35 |
| A | 41 | 75.54 | 71.44 | 71.19 | 76.06 | 109.71 | 123.96 | 129.86 | 125.39 | 136.74 | 137.07 | 138.59 | 132.15 | 133.91 | 135.29 | 145.51 | 125.71 | 118.93 | 112.78 | 125.12 | 119.15 | 121.10 | 112.17 | 105.63 | 118.76 | 100.26 | 103.41 |
| A | 42 | 61.34 | 56.47 | 57.98 | 60.75 | 65.04 | 75.88 | 82.84 | 79.51 | 81.48 | 89.24 | 97.75 | 98.63 | 98.65 | 103.11 | 101.59 | 97.30 | 93.84 | 93.84 | 91.05 | 93.42 | 92.31 | 82.48 | 81.44 | 83.68 | 85.72 | 85.75 |
| A | 43 | 75.58 | 74.46 | 73.34 | 84.20 | 71.63 | 125.59 | 121.79 | 119.37 | 123.33 | 116.04 | 118.44 | 120.26 | 120.65 | 124.43 | 117.76 | 119.52 | 118.90 | 114.12 | 114.54 | 110.45 | 119.31 | 104.89 | 106.32 | 103.54 | 109.05 | 98.07 |
| A | - 44 | 63.89 | 64.05 | 65.47 | 69.36 | 86.83 | 99.88 | 110.26 | 116.34 | 113.34 | 113.39 | 110.81 | 108.74 | 107.83 | 114.93 | 109.34 | 104.69 | 105.65 | 103.16 | 104.25 | 100.39 | 94.54 | 94.78 | 94.84 | 92.32 | 91.15 | 90.75 |
| | etic mean | 74.70 | 71.35 | 71.41 | 75.36 | 96.62 | 112.06 | 118.83 | 124.88 | 127.20 | 128.76 | 128.85 | 128.55 | 127.59 | 132.28 | 128.47 | 125.43 | 124.78 | 123.76 | 121.22 | 119.14 | 119.95 | 113.14 | 110.35 | 108.88 | 105.08 | 102.11 |
| | rd deviation | 10.92 | 9.82 | 11.63 | 11.27 | 18.78 | 18.88 | 17.98 | 17.35 | 18.67 | 15.90 | 15.64 | 14.98 | 16.47 | 16.21 | 15.95 | 17.24 | 17.17 | 17.16 | 16.09 | 15.03 | 14.79 | 15.10 | 14.08 | 11.95 | 12.05 | 11.45 |
| | CV% | 14.62 | 13.76 | 16.29 | 14.96 | 19.44 | 16.84 | 15.13 | 13.90 | 14.68 | 12.35 | 12.14 | 11.65 | 12.91 | 12.25 | 12.41 | 13.74 | 13.76 | 13.86 | 1327 | 12.62 | 12.33 | 13.34 | 12.76 | 10.98 | 11.47 | 11.22 |



Table A2.2 Table of individual concentrations corresponding to unadjusted levothyroxine (test drug [B]). N = 43 subjects.

| Note | | | | | | | | | | <u> </u> | | _ | | | _ | | | _ | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | Form | Volunteer | *** | | | | | | | | | | | | | | | | | | | | *** | | | | *** | |
| | | | | | | | | | | | | | | | | | | | | | | | | | | | | - |
| 3 | | _ | | | | | | | | | | | | | | | | | | | | | | | | | | |
| No. | | _ | | | | | | | | | | | | | | | | | | | | | | | | | | |
| S | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| S | | | | | | | | | | | | | | | | | | | | | | | | | | | | - |
| No. | | | | | | | | | 81.96 | | | | | | | | | | | | | - 4000 | h | | 96.50 | | | - |
| S | | | | | | | | | | | | | | | | | | | | | | | 700000 | | | | | |
| S | | _ | | - | | | | | | | | | | | | | | | | | | | | 10000 | | | | - |
| S | | _ | | | | | | | | | | | | | | | | | | | | | | - | | 10000 | - | - |
| S | | _ | | | | | | | | | | | | | | | | | - | | | | | | - | | | |
| S | | | | | | | | | | | | | | | | | | 4000000 | | ******* | | | | | | | | |
| S | | | | | 74.52 | | | 133.77 | | | | | 143.33 | | | | - 40 | | | | 1000 | | | | | | | |
| S | | | | | | | | | | | | | | | | | | | | | 9000 | | | | | | | - |
| S | | | | | | | | | | | | | | | | | 1000000 | | | | | | | | | | | - |
| B | | | | | | | | | | | | | | | 400 | | - | | | | | | | | | | | - |
| S | | | | | | | | | | | | | | | | 0. 2000 | 10000- | | | | | | | | | | | |
| S | _ | | 84.99 | 77.05 | 90.76 | 86.67 | 101.88 | 117.81 | | 129.34 | 129.04 | | | 4000000 | | ******* | 130.31 | 000000000000000000000000000000000000000 | 100000 | 129.56 | | 126.23 | | 11894 | 114.14 | | | |
| S | _ | | | | | | | | | | | 122.13 | - 10 | 100 | | | 10000A | | | | | 118.48 | | | 116.81 | | | - |
| B 20 S.4 S.5 S | _ | | | | | | | | | | | | | 100000 | | 0000 | 70 | | | | | | | | | | | |
| B 21 9.56 7.52 6.52 7.53 6.52 7.54 7.55 6.52 7.55 6.52 7.55 | _ | | | | | | | | | | | | | | | | | 4000 | | | | | | | | | | - |
| B | _ | 20 | | | | | | | | | 145.02 | 100 | 134.51 | 100000 | | 100. | 4000 | | | - | | | | 117.33 | | | | |
| B 23 79.66 73.54 79.53 82.86 127.40 184.40 184.22 193.80 137.90 144.55 138.77 137.90 138.80 138.90 138.9 | | 21 | 59.65 | 57.52 | 63.92 | 76.24 | 95.62 | 119.30 | 119.55 | 126.49 | 126.77 | 119.65 | 125.74 | 122.58 | 122.96 | 127.39 | 111.11 | 110.35 | 113.36 | 114.16 | 114.48 | 119.87 | 124.75 | 106.76 | 10A.33 | 100.20 | 102.22 | - |
| 8 24 7.18 6.62 70.30 6.65 75.4 93.9 78.87 81.2 86.5 80.7 81.89 80.9 19.89 12.18 12.31 12.01 12.71 15.00 99.7 19.30 10.62 99.5 95.8 19.81 19.81 19.80 19.87 19.85 19.80 1 | | 22 | 68.84 | 62.73 | 67.87 | 65.27 | 84.55 | | 97.47 | 105.33 | 109.69 | 108.94 | 103.64 | 106.34 | 107.20 | 104.29 | 102.97 | 99.22 | 110.13 | 102.27 | 103.97 | 103.77 | 96.84 | 99.35 | 95.21 | 95.14 | | - |
| 8 25 57.5 70.8 68.7 88.5 19.8 | В | 23 | 79.86 | 73.54 | 79.53 | 89.28 | 127.40 | 148.48 | 146.23 | 150.89 | 137.90 | 144.25 | 138.97 | 137.93 | 138.88 | 145.47 | 139.20 | 131.91 | 131.42 | 127.46 | 126.44 | 121.98 | 118.18 | 11815 | 116.62 | 117.02 | 110.53 | 108.36 |
| 8 | | 24 | | 66.42 | 70.30 | | | | 1000000 | 81.42 | | 700000 | | | | | 124.33 | | | | | 103.39 | | | ***** | | | |
| 8 27 819 7951 818 1067 11951 1229 1303 1245 1255 1259 1270 1265 1259 1270 1265 1270 | | 25 | 67.95 | 70.48 | 68.27 | 89.15 | 119.81 | 129.69 | 124.25 | 116.80 | 125.03 | 111.16 | 124.61 | 131.59 | 111.88 | 120.18 | 109.78 | 123.62 | 114.47 | 126.A7 | 109.91 | 122.33 | 113.60 | 119.75 | 103.82 | 116.20 | | |
| 8 28 66.97 61.66 59.88 73.5 302.82 94.70 107.85 98.74 188.52 155.87 120.64 157.84 120.93 199.71 132.48 134.09 134.09 136.99 132.48 78.49 136.71 137.00 138.75 125.67 135.49 136.75 135.49 136.75 135.49 136.75 136.74 137.09 138.49 138.4 | В | 26 | 85.21 | 83.51 | 83.28 | 82.65 | 95.65 | 109.16 | 119.14 | 135.11 | 138.58 | 134.03 | 133.20 | 137.50 | 132.08 | 130.88 | 130.09 | 130.22 | 131.48 | 129.86 | 124.73 | 129.93 | 133.16 | 126.23 | 125.84 | 120.91 | 119.69 | 109.87 |
| 8 29 97.34 87.84 87.28 91.29 82.77 78.70 127.77 131.25 132.77 131.25 132.77 131.41 137.95 135.45 135.77 130.99 143.13 146.13 146.15 146.15 146.15 136.39 130.14 135.71 117.00 128.75 125.53 85.25 97.64 8 30 48.27 6.25 92.42 105.44 111.58 110.44 120.72 108.24 111.95 109.04 105.12 105.30 106.71 100.99 114.85 105.11 114.56 97.60 99.01 91.38 89.55 94.01 95.74 87.71 8 32.77 17.77 73.00 82.92 17.88 128.05 121.07 129.68 130.87 123.46 117.99 156.24 111.95 109.04 115.15 112.05 106.05 | В | 27 | 81.93 | 79.61 | 79.52 | 81.58 | 106.71 | 119.51 | 122.59 | 130.19 | 124.58 | 122.95 | 126.99 | 125.77 | 131.49 | 132.69 | 122.45 | 119.21 | 125.92 | 120.20 | 127.14 | 112.75 | 121.06 | 111.11 | 111.01 | 109.97 | 104.54 | 94.99 |
| 8 30 48.77 52.86 50.07 60.99 82.30 103.06 99.13 11036 93.81 122.50 111.76 128.65 112.50 106.25 106.75 104.07 108.84 100.66 98.92 97.89 97.80 94.11 93.29 92.20 95.94 98.34 91.81 8 31 59.76 58.68 57.68 62.51 92.42 105.44 111.58 110.44 120.72 108.24 117.98 125.62 111.94 122.16 121.28 116.37 109.04 114.85 105.11 114.55 17.40 99.01 91.39 89.55 94.01 95.74 82.71 8 32.88 128.63 121.07 122.68 130.87 122.49 117.98 125.62 111.94 122.16 121.28 116.37 109.01 111.44 115.81 109.23 112.82 104.36 105.94 109.92 98.12 95.78 8 34 85.80 85.71 87.57 97.29 117.04 136.71 150.13 156.54 144.85 142.16 148.31 144.83 146.08 155.08 144.31 145.04 127.51 122.51 | В | 28 | 66.97 | 61.66 | 59.68 | 73.55 | 102.82 | 94.72 | 107.26 | 98.74 | 168.52 | 155.87 | 120.64 | 154.40 | 120.93 | 109.21 | 132.49 | 134.03 | 143.69 | 112.48 | 75.42 | 108.32 | 88.23 | 97.09 | 103.57 | 104.70 | 95.27 | 86.94 |
| 8 31 59.76 58.68 57.88 62.51 52.42 107.88 119.65 121.07 128.68 130.87 123.49 117.99 125.62 111.49 122.16 121.87 108.30 111.44 115.81 109.20 111.48 115.81 109.20 112.82 108.35 109.20 112.82 109.35 109.73 10 | В | 29 | 97.34 | 87.84 | 87.29 | 91.29 | 82.72 | 76.70 | 127.77 | 131.26 | 132.27 | 131.44 | 137.96 | 135.46 | 135.17 | 150.99 | 148.19 | 143.18 | 140.61 | 140.69 | 136.39 | 130.74 | 135.71 | 117.00 | 128.75 | 125.63 | 86.25 | 97.64 |
| 8 32 74.57 77.77 73.00 82.92 117.88 129.63 121.07 129.68 130.77 129.68 129.78 130.78 1 | В | 30 | 48.27 | 62.54 | 60.07 | 60.59 | 82.30 | 103.06 | 99.13 | 110.36 | 93.81 | 122.50 | 111.78 | 128.63 | 112.50 | 106.85 | 106.76 | 104.07 | 103.84 | 100.66 | 98.92 | 97.49 | 94.11 | 93.29 | 92.20 | 95.94 | 98.34 | 91.81 |
| 8 33 85,82 74,62 75.11 99.07 141.56 161.02 157.87 147.99 148.66 140.65 140.68 155.08 143.99 137.64 133.49 127.56 133.97 126.69 122.29 114.37 124.52 115.72 110.54 103.64 8 35. 79.92 75.24 77.83 75.58 75.75 93.70 98.58 126.68 129.74 114.37 118.96 126.74 166.00 115.91 122.55 122.51 117.39 113.66 121.30 123.99 127.50 123.95 123.86 123.29 114.37 124.62 115.72 110.54 103.64 8 36.80 79.92 75.84 77.17 70.06 78.77 76.21 98.33 113.56 125.51 133.60 134.37 135.01 137.10 125.76 124.50 124.59 127.55 128.75 124.59 126.74 126.30 122.95 118.48 116.66 116.39 110.23 112.59 8 39 79.24 73.20 75.19 96.99 134.82 158.28 152.04 167.61 162.56 149.67 149.79 160.77 160.35 146.53 169.96 161.46 152.92 136.48 128.85 134.67 138.21 131.69 121.55 123.97 109.32 111.02 8 44.00 88.75 78.71 78.88 80.61 98.42 113.55 125.42 140.87 147.13 150.63 156.04 133.70 136.64 141.41 122.30 138.67 147.88 131.75 125.72 120.91 143.46 124.37 118.94 147.04 110.01 123.99 116.24 109.57 109.57 109.58 8 42 58.13 53.78 53.58 60.29 75.79 84.43 75.84 66.89 89.15 85.86 88.30 87.89 86.54 88.43 82.10 84.78 85.15 82.87 83.06 82.30 86.86 78.56 75.99 82.26 79.92 82.69 8 44 60.88 58.94 59.19 65.44 97.52 107.56 101.06 97.42 100.97 97.01 98.43 99.18 95.74 101.50 102.70 98.22 96.50 88.77 99.18 93.16 94.50 148.27 117.86 118.27 110.55 106.77 105.08 100.77 1 | | | 59.76 | 58.68 | 57.68 | | 92.42 | 105.44 | 111.58 | 110.44 | 120.72 | 108.24 | 111.95 | 109.04 | 105.12 | | 106.71 | | 114.85 | 105.11 | | 97.40 | | 91.39 | 89.55 | | | |
| 8 34 85.60 85.71 87.57 97.29 117.04 136.71 150.13 156.54 144.85 142.16 143.31 144.38 146.08 155.08 143.59 137.64 133.49 127.56 133.97 126.69 122.29 114.37 124.62 115.72 110.54 103.64 8 35 79.92 75.24 77.83 75.89 75.75 93.70 98.58 126.68 129.74 114.37 118.96 126.74 106.00 115.91 122.55 122.51 117.39 113.36 129.33 122.55 114.84 104.42 113.51 114.40 101.69 118.67 8 36 80.90 79.65 83.02 98.85 141.40 145.06 151.27 147.96 126.60 134.04 144.55 128.26 138.90 144.31 135.24 137.31 131.70 131.66 121.30 123.59 127.39 123.36 113.38 111.00 116.32 117.77 8 8 37 75.94 77.17 70.06 78.77 76.21 98.33 113.56 125.51 133.60 124.37 135.01 137.10 129.76 134.36 124.19 127.55 129.75 140.99 126.73 122.72 119.25 118.43 116.66 116.39 110.23 112.99 8 8 39 79.24 73.20 75.19 96.99 134.82 158.28 152.04 167.61 162.56 149.67 149.79 160.77 160.35 145.53 169.96 161.45 152.92 136.48 128.85 134.67 138.21 131.69 121.55 123.97 109.32 111.02 8 8 40 88.75 78.71 78.88 80.61 98.42 113.55 125.42 140.87 147.13 150.63 156.20 153.34 152.50 150.19 157.47 152.50 154.94 154.06 147.52 147.69 148.03 141.74 140.67 124.92 120.07 120.69 8 41 88.90 80.53 82.44 98.73 123.53 146.66 141.31 163.04 133.70 136.64 141.41 122.30 138.67 147.68 131.75 125.77 120.91 143.46 124.37 118.94 147.04 110.01 123.99 116.24 109.57 101.65 8 42.55 134.55 134.55 135.85 80.85 80.8 | | | 400000000 | 200000 | | | | | | | | | | | | | | | | | | | | | | | | - |
| B 35 79.92 75.24 77.83 75.86 75.75 93.70 98.58 126.68 129.74 114.37 118.95 126.74 106.00 115.91 122.55 122.51 117.39 113.36 129.33 122.55 114.84 104.42 113.51 114.40 101.69 118.67 B 36 80.90 79.65 83.02 98.65 141.40 146.06 151.27 147.96 126.60 134.04 144.55 128.26 138.90 144.31 135.24 137.31 131.70 131.66 121.30 123.59 127.39 123.36 113.38 111.00 116.32 117.77 B 37 75.84 72.17 70.06 78.77 76.21 98.33 113.56 125.51 133.60 134.37 135.01 137.10 129.76 134.36 124.19 127.55 129.75 149.99 126.73 122.72 119.25 118.43 116.66 116.39 110.23 112.59 129.98 134.82 138.28 152.04 167.61 162.56 149.67 149.79 160.77 160.35 145.53 169.96 161.46 152.92 136.48 128.85 134.67 138.21 131.69 121.55 123.97 109.32 111.02 132.99 126.73 127.07 120.99 126.73 127.71 78.88 80.61 98.42 113.55 125.42 140.87 147.13 150.63 156.20 153.34 152.50 150.19 157.47 152.50 154.94 154.06 147.52 147.69 148.03 141.74 140.67 124.92 120.07 120.69 18 41 88.99 80.53 82.44 98.73 123.53 146.66 141.31 163.04 133.70 136.64 141.41 122.30 138.67 147.68 131.75 125.77 120.91 143.46 124.37 118.94 147.04 110.01 123.99 116.24 109.57 101.65 18 42 98.13 137.85 133.85 | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| B 36 80.90 79.65 83.02 98.85 141.40 145.06 151.27 147.96 126.60 134.04 144.55 128.26 138.90 144.31 135.24 137.31 131.70 131.66 121.30 123.99 127.39 123.36 113.86 110.03 110.23 112.79 B 37 75.84 77.17 70.06 78.77 76.21 98.33 113.56 125.51 133.60 134.37 135.01 137.10 129.76 134.36 124.19 127.55 129.75 140.99 126.73 122.72 119.25 118.43 116.66 116.39 110.23 112.59 B 39 79.24 73.20 75.19 96.99 134.82 158.28 162.04 167.61 162.56 148.79 160.77 160.35 146.53 169.96 161.46 152.92 136.48 128.05 134.67 138.21 131.69 121.55 123.97 109.32 111.02 B 40 88.75 78.71 78.88 80.61 98.42 113.55 125.42 140.87 147.13 150.63 156.20 153.34 152.50 150.19 157.47 152.50 154.94 154.06 147.52 147.69 148.03 141.74 140.67 124.92 120.07 120.69 B 41 88.90 80.53 82.44 98.73 123.53 146.86 141.31 163.04 133.70 136.64 141.41 122.30 138.67 147.68 131.75 125.72 120.91 143.46 124.37 118.94 147.04 110.01 123.99 116.24 109.57 101.65 B 42 58.13 53.78 53.58 60.29 75.79 84.43 75.84 86.89 89.15 85.86 88.30 87.49 86.54 88.43 82.10 84.78 82.15 125.51 116.16 112.95 107.94 111.98 109.56 104.97 98.52 96.75 106.05 B 44 60.89 58.94 59.19 65.44 97.52 107.26 101.06 97.42 100.97 97.01 98.43 99.18 99.18 102.40 102.70 98.92 96.50 88.77 99.18 99.16 94.50 87.69 88.12 88.35 75.74 87.11 Arithmetic mean 74.79 71.97 72.49 79.29 101.47 115.84 121.69 126.61 127.71 125.26 126.64 127.59 125.51 130.18 127.55 125.76 124.78 122.10 120.67 117.86 118.27 111.05 100.57 105.08 100.79 13.40 100.79 10.79 | В | | 70000 | | | | | | | | | | | | | ****** | | | | | | | | | | | | - |
| B 37 75.84 72.17 70.06 78.77 76.21 98.33 13.56 125.51 133.60 134.37 135.01 137.10 129.76 134.36 124.19 127.55 129.75 140.99 126.73 122.72 119.25 118.43 116.66 116.39 110.23 112.59 B 39 79.24 73.20 75.19 96.99 134.82 158.28 162.04 167.61 162.56 149.87 149.79 160.77 160.35 146.53 169.96 161.46 152.92 136.48 128.85 134.67 138.21 131.69 121.55 123.97 109.32 111.02 B 40 88.75 78.71 78.88 80.61 98.42 113.55 125.42 140.87 147.13 150.63 156.20 153.34 152.90 160.19 157.47 152.50 158.49 154.06 147.52 147.69 148.03 141.74 140.67 124.92 120.07 120.99 B 41 88.90 80.53 82.44 98.73 123.53 146.86 141.31 163.04 133.70 136.64 141.41 122.30 138.67 147.68 131.75 125.72 120.91 143.46 124.37 118.94 147.04 110.01 123.99 116.24 109.57 101.65 B 42 58.13 53.78 53.58 60.29 75.79 84.43 75.84 86.89 88.15 85.86 88.30 87.49 86.54 88.43 82.10 84.78 82.17 83.06 82.30 86.86 78.56 75.99 82.26 79.92 82.69 B 43 75.57 74.71 76.61 81.40 117.50 126.52 125.73 132.44 121.71 125.72 123.31 130.43 125.43 115.54 115.94 121.95 116.16 112.95 107.94 111.98 109.56 104.97 98.52 96.76 106.05 B 44 60.89 58.94 59.19 65.44 97.52 107.26 101.06 97.42 100.97 97.01 98.43 99.18 95.74 101.54 102.70 98.92 96.50 88.77 99.18 93.16 94.50 87.63 88.12 88.35 75.74 87.21 Arithmetic mean 74.79 71.97 72.49 79.29 101.47 115.84 121.49 126.41 127.71 126.26 126.64 127.59 125.51 130.18 127.55 125.76 124.78 122.10 120.67 17.86 118.27 110.55 108.77 105.08 100.79 13.40 12.77 125.00 12.77 103.31 | - | | 1000 | | | | | | | - | | | | | | | | | - | | | _ | | _ | _ | | | _ |
| B 39 79.4 73.20 75.19 96.99 134.82 158.28 152.04 167.61 162.56 149.67 149.79 160.75 160.35 145.53 145.95 161.46 152.92 136.48 128.85 134.67 138.21 131.69 121.55 123.97 109.32 111.02 B 40 88.75 78.71 78.88 80.61 98.42 113.55 125.42 140.87 147.13 150.63 156.20 153.34 152.50 160.19 157.47 152.50 154.94 154.06 147.52 147.69 148.03 141.74 140.67 124.92 120.07 120.69 B 41 88.90 80.53 82.44 98.73 123.53 146.86 141.31 163.04 133.70 136.64 141.41 122.30 138.67 147.68 131.75 125.77 120.91 143.46 124.37 118.94 147.04 110.01 123.99 116.24 109.57 101.65 B 42 58.13 53.78 53.58 60.29 75.79 84.43 75.84 86.89 89.15 85.86 88.30 87.49 86.54 88.43 82.10 84.78 82.10 84.78 82.15 82.87 83.06 82.30 86.86 78.56 75.99 82.26 79.92 82.69 88.43 75.57 74.71 76.61 81.40 117.50 126.52 125.73 132.44 121.71 125.72 123.31 130.43 126.43 117.58 115.94 121.95 116.16 112.95 107.94 111.98 109.56 104.97 98.52 96.76 106.05 88.44 60.89 58.94 59.19 65.44 97.52 107.26 101.06 97.42 100.97 97.01 98.43 99.18 95.74 101.54 102.70 98.92 96.50 88.77 99.18 93.16 94.50 87.63 88.12 88.35 75.74 87.21 Arithmetic mean 74.79 71.97 72.49 79.29 101.47 115.84 121.69 126.41 127.71 126.26 126.64 127.59 125.51 130.18 127.55 125.76 124.78 122.10 120.67 117.86 118.27 111.05 105.5 108.77 105.08 100.79 97.01 98.43 99.18 90.45 126.54 127.59 125.51 130.18 127.55 125.76 124.78 122.10 120.67 117.86 118.27 111.55 108.77 105.08 100.79 97.01 98.43 99.18 90.45 126.44 127.59 125.51 130.18 127.55 125.76 124.78 122.10 120.67 117.86 118.27 111.05 100.55 108.77 105.08 100.79 97.01 98.43 99.18 90.45 126.44 127.59 125.51 130.18 127.55 125.76 124.78 122.10 120.67 117.86 118.27 110.55 108.77 105.08 100.79 97.01 98.43 99.18 90.45 126.44 127.71 126.26 126.64 127.59 125.51 130.18 127.55 125.76 124.78 122.10 120.67 117.86 118.27 110.55 108.77 105.08 100.79 97.01 98.43 99.18 126.44 127.71 126.26 126.64 127.59 125.51 130.18 127.55 125.76 124.78 122.10 120.67 117.86 118.27 110.55 108.77 105.08 100.79 97.01 98.43 99.18 127.55 125.51 130.18 127.55 125.76 124.78 122.10 120.67 117.86 118.27 110.55 108.77 1 | | | | 4000000 | | 40000 | | | | | | | | | | | | | _ | - | | _ | | | _ | | | |
| B 40 88.75 78.71 78.88 80.61 98.42 113.55 125.42 140.87 147.13 150.63 156.20 153.34 152.50 150.19 157.47 152.50 154.94 154.06 147.52 147.69 148.03 141.74 140.67 124.92 120.07 120.69 B 41 88.90 80.53 82.44 98.73 123.53 146.66 141.31 163.04 133.70 136.64 141.41 122.30 138.67 147.68 131.75 125.72 120.91 143.46 124.37 118.94 147.04 110.01 123.99 116.24 109.57 101.65 B 42 58.13 53.78 53.58 60.29 75.79 84.43 75.84 86.89 89.15 85.86 88.30 87.49 86.54 88.43 82.10 84.78 82.10 84.78 82.15 82.87 83.06 82.30 86.86 78.56 75.99 82.26 79.92 82.69 B 43 75.57 74.71 76.61 81.40 117.50 126.52 125.73 132.44 121.71 125.72 123.31 130.43 126.43 117.58 115.94 112.95 116.16 112.95 107.94 111.98 109.56 104.97 98.52 96.76 106.05 B 44 60.89 58.94 59.19 65.44 97.52 107.26 101.06 97.42 100.97 97.01 98.43 99.18 95.74 101.54 102.70 98.92 96.50 89.77 99.18 93.16 94.50 87.69 87.19 88.12 88.35 75.74 87.21 Arithmetic mean 74.79 71.97 72.49 79.29 101.47 115.84 121.49 126.41 127.71 126.26 126.64 127.59 125.51 130.18 127.55 125.76 124.78 122.10 120.67 117.86 118.27 111.35 110.55 108.77 105.08 100.79 95.04 | | | | | | | | | | | | | | | | | | | | | | | | | | | | - |
| B 41 88.90 80.53 82.44 98.75 123.53 146.86 141.31 163.04 133.70 136.64 141.41 122.30 138.67 147.68 131.75 125.72 120.91 143.46 124.37 118.94 147.04 110.01 123.99 116.24 109.57 101.65 8 42 58.13 53.78 53.58 60.29 75.79 84.63 75.94 86.89 89.15 85.86 88.30 87.49 86.54 88.43 82.10 84.78 82.10 84.7 | - | | | | | | | | | - | | | | | _ | | | | - | | | - | | | _ | | | |
| B 42 58.13 53.78 53.58 60.29 75.79 84.43 75.84 86.89 89.15 85.86 88.30 87.49 86.54 88.43 82.10 84.78 85.15 82.87 83.06 82.30 86.86 78.56 75.99 82.26 79.92 82.69 B 43 75.57 74.71 76.61 81.40 117.50 126.52 125.73 132.44 121.71 125.72 123.31 130.43 126.43 124.03 117.58 115.94 121.95 116.16 112.95 107.94 111.98 109.56 104.97 98.52 96.76 106.05 B 44 60.89 58.94 59.19 65.44 97.52 107.26 101.06 97.42 100.97 97.01 98.43 99.18 99.18 99.18 102.70 98.92 96.50 89.77 99.18 93.16 94.50 87.63 88.12 88.35 75.74 87.21 Arithmetic mean 74.79 71.97 72.49 79.29 101.47 115.84 121.49 126.41 127.71 126.26 126.64 127.59 125.51 130.18 127.55 125.76 124.78 122.10 120.67 117.86 118.27 111.35 110.55 108.77 105.08 100.79 Standard deviation 10.76 9.70 9.89 11.32 18.42 21.28 21.62 21.68 21.19 20.60 20.78 20.45 20.45 20.45 20.45 18.68 18.49 18.13 17.38 18.68 16.17 18.07 14.90 15.83 12.50 12.77 103.38 | _ | _ | | | | | | | | _ | | | _ | | _ | | | | - | | _ | _ | | _ | _ | | | - |
| B 43 75.7 74.71 76.61 81.40 117.50 126.52 125.73 132.44 121.71 125.72 123.31 130.43 125.43 127.58 115.94 121.95 116.16 112.95 107.94 111.98 109.56 104.97 98.52 96.76 106.05 8 44 60.89 58.94 59.19 65.44 97.52 107.26 101.06 97.42 100.97 97.01 98.43 99.18 99.18 95.74 101.54 102.70 98.92 96.50 89.77 99.18 93.16 94.50 87.63 88.12 88.35 75.74 87.21 Arithmetic mean 74.79 71.97 72.49 79.29 101.47 115.84 121.49 126.41 127.71 126.26 126.64 127.59 125.51 130.18 127.55 125.76 124.78 122.10 120.67 17.86 118.27 111.35 110.55 108.77 105.08 100.79 58.44 12.19 12 | - | - | | | | | | | | _ | | | _ | | | | | | | | | _ | _ | _ | _ | | | _ |
| 8 44 60.89 58.94 59.19 65.44 97.52 107.26 100.06 97.42 100.97 97.01 98.43 99.18 95.74 101.54 102.70 98.92 96.50 89.77 99.18 99.16 94.50 87.63 88.12 88.35 75.74 87.21 Arithmetic mean 74.79 71.97 72.49 79.29 101.47 115.84 121.49 126.41 127.71 126.26 126.64 127.59 125.51 130.18 127.55 125.76 124.78 122.10 120.67 117.86 118.27 111.35 110.55 108.77 105.08 100.79 Standard deviation 10.75 9.70 9.70 9.70 9.70 18.42 12.28 21.62 21.68 21.19 20.60 20.78 20.45 20.45 20.45 126.64 127.59 19.66 18.68 18.49 18.13 17.38 18.68 16.17 18.07 14.90 15.43 12.50 12.77 103.3 | - | | | | | | | | | | | | | | _ | | | | | | | - | | | | | | |
| Arithmetic mean 74.79 71.97 72.49 79.29 101.47 115.84 121.49 126.41 127.71 126.26 126.64 127.59 125.51 130.18 127.55 125.76 124.78 122.10 120.67 117.86 118.27 111.35 110.55 108.77 105.08 100.79 13.04 12.04 12.0 | | | | | | | | | | | | | | | | | | | | | _ | | | | | | | - |
| Standard deviation 10.76 9.70 9.69 11.32 18.42 21.28 21.62 21.68 21.19 20.60 20.78 20.45 20.19 19.66 18.68 18.49 18.13 17.38 18.68 16.17 18.07 14.90 15.43 12.50 12.77 10.33 | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| | | | | | | | | | | | | | | | | | | | | | | | | - | | | | |
| CV% 14.39 13.48 13.37 14.28 18.16 18.37 17.80 17.15 16.59 16.31 16.41 16.03 16.08 15.10 14.64 14.71 14.53 14.23 15.48 13.72 15.28 13.38 13.96 11.49 12.15 10.25 | | | | | | | | | | | | | | | | | | | | | | | | | _ | | | |
| | ( | .V% | 14.39 | 13.48 | 13.37 | 14.28 | 18.16 | 18.37 | 17.80 | 17.15 | 16.59 | 16.31 | 16.41 | 16.03 | 16.08 | 15.10 | 14.64 | 14.71 | 1453 | 14.23 | 15.48 | 13.72 | 15.28 | 13.38 | 13.96 | 11.49 | 12.15 | 10.25 |



Table A2.3. Descriptive statistics of the values of the levothyroxine unadjusted concentration in a biological fluid (N = 43).

| | | Euti | Eutirox® approved formulation (A) Eutirox® test formulation (B) Minimum Maximum Standard Arithmetic Minimum Maximum Standard | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time | Arithmetic<br>Mean | Median | Minimum<br>Value | Maximum<br>Value | Standard<br>Deviation | %CV | Arithmetic<br>Mean | Median | Minimum<br>Value | Maximum<br>Value | Standard<br>Deviation | %CV |
| -0.50 | 74.70 | 75.58 | 51.32 | 96.31 | 10.92 | 14.62 | 74.79 | 75.57 | 48.27 | 97.34 | 10.76 | 14.39 |
| -0.25 | 71.35 | 71.52 | 51.97 | 88.14 | 9.82 | 13.76 | 71.97 | 72.77 | 53.78 | 89.15 | 9.70 | 13.48 |
| 0.00 | 71.41 | 73.34 | 38.94 | 92.32 | 11.63 | 16.29 | 72.49 | 72.06 | 53.58 | 90.76 | 9.69 | 13.37 |
| 0.50 | 75.36 | 77.96 | 47.34 | 93.70 | 11.27 | 14.96 | 79.29 | 79.72 | 60.29 | 99.07 | 11.32 | 14.28 |
| 1.00 | 96.62 | 97.06 | 59.66 | 157.65 | 18.78 | 19.44 | 101.47 | 98.42 | 67.54 | 141.56 | 18.42 | 18.16 |
| 1.50 | 112.06 | 114.25 | 75.83 | 165.98 | 18.88 | 16.84 | 115.84 | 113.55 | 69.39 | 161.02 | 21.28 | 18.37 |
| 2.00 | 118.83 | 116.77 | 82.84 | 161.69 | 17.98 | 15.13 | 121.49 | 122.59 | 75.84 | 162.04 | 21.62 | 17.80 |
| 2.50 | 124.88 | 124.02 | 79.51 | 176.09 | 17.35 | 13.90 | 126.41 | 126.68 | 81.42 | 172.13 | 21.68 | 17.15 |
| 3.00 | 127.20 | 128.42 | 81.48 | 170.46 | 18.67 | 14.68 | 127.71 | 127.83 | 80.95 | 179.10 | 21.19 | 16.59 |
| 3.25 | 128.76 | 130.24 | 89.24 | 163.65 | 15.90 | 12.35 | 126.26 | 127.74 | 80.47 | 173.35 | 20.60 | 16.31 |
| 3.50 | 128.85 | 129.32 | 97.75 | 159.19 | 15.64 | 12.14 | 126.64 | 125.74 | 81.89 | 183.00 | 20.78 | 16.41 |
| 3.75 | 128.55 | 129.39 | 95.87 | 163.10 | 14.98 | 11.65 | 127.59 | 128.26 | 87.49 | 184.14 | 20.45 | 16.03 |
| 4.00 | 127.59 | 129.48 | 98.65 | 162.15 | 16.47 | 12.91 | 125.51 | 126.43 | 86.54 | 187.29 | 20.19 | 16.08 |
| 4.25 | 132.28 | 130.90 | 102.57 | 168.47 | 16.21 | 12.25 | 130.18 | 130.88 | 88.43 | 190.12 | 19.66 | 15.10 |
| 4.50 | 128.47 | 128.83 | 101.59 | 165.46 | 15.95 | 12.41 | 127.55 | 124.19 | 82.10 | 179.61 | 18.68 | 14.64 |
| 4.75 | 125.43 | 125.04 | 97.30 | 167.06 | 17.24 | 13.74 | 125.76 | 126.01 | 84.78 | 181.77 | 18.49 | 14.71 |
| 5.00 | 124.78 | 124.72 | 93.84 | 164.72 | 17.17 | 13.76 | 124.78 | 122.51 | 85.15 | 183.27 | 18.13 | 14.53 |
| 5.50 | 123.76 | 124.50 | 93.84 | 161.41 | 17.16 | 13.86 | 122.10 | 121.23 | 82.87 | 180.55 | 17.38 | 14.23 |
| 6.00 | 121.22 | 121.99 | 91.05 | 164.27 | 16.09 | 13.27 | 120.67 | 124.37 | 75.42 | 182.27 | 18.68 | 15.48 |
| 6.50 | 119.14 | 119.15 | 93.42 | 157.78 | 15.03 | 12.62 | 117.86 | 118.85 | 82.30 | 166.36 | 16.17 | 13.72 |
| 8.00 | 119.95 | 120.06 | 92.31 | 157.87 | 14.79 | 12.33 | 118.27 | 119.93 | 76.68 | 159.04 | 18.07 | 15.28 |
| 10.00 | 113.14 | 114.76 | 82.48 | 148.44 | 15.10 | 13.34 | 111.35 | 111.11 | 78.56 | 148.79 | 14.90 | 13.38 |
| 12.00 | 110.35 | 110.33 | 81.44 | 144.12 | 14.08 | 12.76 | 110.55 | 111.01 | 75.99 | 149.12 | 15.43 | 13.96 |
| 24.00 | 108.88 | 109.58 | 83.68 | 128.59 | 11.95 | 10.98 | 108.77 | 111.23 | 82.26 | 127.82 | 12.50 | 11.49 |
| 36.00 | 105.08 | 105.05 | 85.15 | 128.25 | 12.05 | 11.47 | 105.08 | 107.39 | 75.74 | 141.81 | 12.77 | 12.15 |
| 48.00 | 102.11 | 101.26 | 83.29 | 125.68 | 11.45 | 11.22 | 100.79 | 98.86 | 82.69 | 121.52 | 10.33 | 10.25 |

| L | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|

Table A2.4. Individual data and descriptive statistics for the levothyroxine pharmacokinetic parameters ( $C_{max}$  in ng/mL,  $AUC_{0-t}$  in  $ng^*h/mL$ , and  $AUC_{0-\infty}$  in  $ng^*h/mL$ ). Unadjusted data.

| | Per | ind | | | C, | | | | ΔII | Cost | | | AUC<br>Form | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Volunteer | | rm | Sequence | Fo | rm c, | Nax. | | Fo | rm | CO.E | Г | Fo | | ~0.m | Ι |
| VOIGILLEE | A | В | Sequence | A | В | B/A | Ln(B/A) | A | В | B/A | Ln(B/A) | A | В | B/A | Ln(B/A) |
| 1 | 2 | 1 | BA | 154.58 | 161.90 | 1.05 | 0.05 | 5385.00 | 5664.69 | 1.05 | 0.05 | 27555.67 | 22603.71 | 0.82 | -0.20 |
| 2 | 2 | 1 | BA | 141.18 | 145.86 | 1.03 | 0.03 | 5779.14 | 5529.30 | 0.96 | -0.04 | 93377.86 | 32154.93 | 0.34 | -1.07 |
| 3 | 2 | 1 | BA | 124.53 | 126.65 | 1.02 | 0.02 | 4277.06 | 4462.98 | 1.04 | 0.04 | 44552.09 | 36788.29 | 0.83 | -0.19 |
| 4 | 1 | 2 | AB | 145.08 | 147.39 | 1.02 | 0.02 | 5336.10 | 5576.05 | 1.04 | 0.04 | 33127.36 | 30266.17 | 0.91 | -0.09 |
| 5 | 1 | 2 | AB | 130.89 | 131.78 | 1.01 | 0.01 | 5015.92 | 4806.67 | 0.96 | -0.04 | 23732.87 | 57135.11 | 2.41 | 0.88 |
| 6 | 2 | 1 | BA | 119.99 | 113.58 | 0.95 | -0.05 | 4473.20 | 4278.30 | 0.96 | -0.04 | 27328.49 | 28813.20 | 1.05 | 0.05 |
| 7 | 1 | 2 | AB | 123.98 | 127.83 | 1.03 | 0.03 | 4470.88 | 4726.66 | 1.06 | 0.06 | 22435.07 | 38531.61 | 1.72 | 0.54 |
| 8 | 1 | 2 | AB | 135.77 | 134.36 | 0.99 | -0.01 | 5043.45 | 5144.63 | 1.02 | 0.02 | 25621.50 | 26220.45 | 1.02 | 0.02 |
| 9 | 1 | 2 | AB | 167.06 | 190.12 | 1.14 | 0.13 | 5991.53 | 6725.22 | 1.12 | 0.12 | 27293.36 | 20606.86 | 0.76 | -0.28 |
| 10 | 1 | 2 | AB | 160.04 | 168.43 | 1.05 | 0.05 | 5752.82 | 6068.60 | 1.05 | 0.05 | 22639.84 | 34231.86 | 1.51 | 0.41 |
| 11 | 1 | 2 | AB | 148.32 | 146.40 | 0.99 | -0.01 | 5637.75 | 5838.71 | 1.04 | 0.04 | 26441.08 | 29309.72 | 1.11 | 0.10 |
| 12 | 2 | 1 | BA | 141.60 | 138.96 | 0.98 | -0.02 | 5338.26 | 5330.46 | 1.00 | 0.00 | 32249.02 | 17139.15 | 0.53 | -0.63 |
| 13 | 1 | 2 | AB | 124.35 | 118.71 | 0.95 | -0.05 | 4991.51 | 4755.50 | 0.95 | -0.05 | 32366.08 | 54498.84 | 1.68 | 0.52 |
| 14 | 2 | 1 | BA | 135.90 | 126.80 | 0.93 | -0.07 | 5092.51 | 5090.77 | 1.00 | 0.00 | 25474.01 | 23160.87 | 0.91 | -0.10 |
| 15 | 2 | 1 | BA | 141.19 | 133.82 | 0.95 | -0.05 | 5486.66 | 5507.99 | 1.00 | 0.00 | 34430.60 | 56586.85 | 1.64 | 0.50 |
| 16 | 2 | 1 | BA | 148.33 | 139.30 | 0.94 | -0.05 | 5413.91 | 5636.37 | 1.04 | 0.04 | 22972.97 | 18563.57 | 0.81 | -0.21 |
| 17 | 1 | 2 | AB | 149.98 | 148.22 | 0.99 | -0.01 | 5600.98 | 5479.24 | 0.98 | -0.02 | 17477.08 | 19420.11 | 1.11 | 0.11 |
| 18 | 2 | 1 | BA | 123.86 | 126.08 | 1.02 | 0.02 | 4541.62 | 4718.95 | 1.04 | 0.04 | 21671.94 | 35245.75 | 1.63 | 0.11 |
| 19 | 1 | 2 | AB | 132.85 | 125.27 | 0.94 | -0.06 | 4874.73 | 4827.43 | 0.99 | -0.01 | 19071.97 | 27211.76 | 1.43 | 0.49 |
| 20 | 2 | 1 | BA | 150.05 | 145.50 | 0.97 | -0.03 | 5958.66 | 5593.17 | 0.94 | -0.01 | 30288.62 | 40886.79 | 1.35 | 0.30 |
| | 2 | | | | | | | *************************************** | 10007 | 1000 | | 34310.03 | | | -0.63 |
| 21 | _ | 1 | BA | 131.96 | 127.39 | 0.97 | -0.04 | 4904.79 | 4920.17 | 1.00 | 0.00 | | 18272.51 | 0.53 | |
| 22 | 1 | 2 | AB | 120.49 | 110.13 | 0.91 | -0.09 | 4439.99 | 4539.05 | 1.02 | 0.02 | 28954.21 | 40806.98 | 1.41 | 0.34 |
| 23 | 2 | 1 | BA | 133.94 | 150.89 | 1.13 | 0.12 | 5312.71 | 5584.70 | 1.05 | 0.05 | 27710.82 | 54566.68 | 1.97 | 0.68 |
| 24 | 1 | 2 | AB | 153.70 | 130.07 | 0.85 | -0.17 | 5340.45 | 4666.15 | 0.87 | -0.13 | 24452.64 | 33802.74 | 1.38 | 0.32 |
| 25 | 1 | 2 | AB | 128.50 | 131.59 | 1.02 | 0.02 | 4670.87 | 5185.27 | 1.11 | 0.10 | 29279.92 | 17005.57 | 0.58 | -0.54 |
| 26 | 1 | 2 | AB | 138.86 | 138.58 | 1.00 | 0.00 | 5830.70 | 5793.95 | 0.99 | -0.01 | 34861.83 | 34957.39 | 1.00 | 0.00 |
| 27 | 2 | 1 | BA | 127.81 | 132.69 | 1.04 | 0.04 | 5222.86 | 5204.65 | 1.00 | 0.00 | 35904.89 | 20777.14 | 0.58 | -0.55 |
| 28 | 2 | 1 | BA | 170.46 | 168.52 | 0.99 | -0.01 | 4733.75 | 4796.02 | 1.01 | 0.01 | 24098.70 | 16026.55 | 0.67 | -0.41 |
| 29 | 2 | 1 | BA | 143.90 | 150.99 | 1.05 | 0.05 | 5390.91 | 5379.68 | 1.00 | 0.00 | 18180.48 | 14997.88 | 0.82 | -0.19 |
| 30 | 1 | 2 | AB | 125.17 | 128.63 | 1.03 | 0.03 | 4751.73 | 4590.71 | 0.97 | -0.03 | 35758.50 | 42327.77 | 1.18 | 0.17 |
| 31 | 1 | 2 | AB | 123.72 | 120.72 | 0.98 | -0.02 | 4558.22 | 4503.63 | 0.99 | -0.01 | 26417.08 | 20488.47 | 0.78 | -0.25 |
| 32 | 1 | 2 | AB | 133.37 | 135.62 | 1.02 | 0.02 | 4979.99 | 5051.05 | 1.01 | 0.01 | 52815.04 | 21743.55 | 0.41 | -0.89 |
| 33 | 1 | 2 | AB | 157.00 | 161.02 | 1.03 | 0.03 | 6143.29 | 5754.78 | 0.94 | -0.07 | 37077.75 | 28138.76 | 0.76 | -0.28 |
| 34 | 1 | 2 | AB | 150.81 | 156.54 | 1.04 | 0.04 | 5742.75 | 5616.20 | 0.98 | -0.02 | 46512.15 | 26381.86 | 0.57 | -0.57 |
| 35 | 1 | 2 | AB | 136.03 | 129.74 | 0.95 | -0.05 | 5504.45 | 5305.90 | 0.96 | -0.04 | 42525.83 | 75099.89 | 1.77 | 0.57 |
| 36 | 2 | 1 | BA | 163.65 | 151.27 | 0.92 | -0.08 | 5745.78 | 5648.48 | 0.98 | -0.02 | 25958.30 | 34447.89 | 1.33 | 0.28 |
| 37 | 2 | 1 | BA | 137.40 | 140.99 | 1.03 | 0.03 | 5502.46 | 5506.30 | 1.00 | 0.00 | 40925.02 | 63350.40 | 1.55 | 0.44 |
| 39 | 2 | 1 | BA | 176.09 | 169.96 | 0.97 | -0.04 | 6382.19 | 5858.48 | 0.92 | -0.09 | 25291.43 | 27801.24 | 1.10 | 0.09 |
| 40 | 2 | 1 | BA | 168.47 | 160.19 | 0.95 | -0.05 | 6307.53 | 6170.73 | 0.98 | -0.02 | 20848.42 | 25550.79 | 1.23 | 0.20 |
| 41 | 2 | 1 | BA | 145.51 | 163.04 | 1.12 | 0.11 | 5292.27 | 5602.80 | 1.06 | 0.06 | 32314.92 | 24227.96 | 0.75 | -0.29 |
| 42 | 1 | 2 | AB | 103.11 | 89.15 | 0.86 | -0.15 | 4063.30 | 3869.62 | 0.95 | -0.05 | 35999.62 | 68147.40 | 1.89 | 0.64 |
| 43 | 2 | 1 | BA | 125.59 | 132.44 | 1.05 | 0.05 | 5105.17 | 4969.59 | 0.97 | -0.03 | 28249.64 | 26459.22 | 0.94 | -0.07 |
| 44 | 1 | 2 | AB | 116.34 | 107.26 | 0.92 | -0.08 | 4501.21 | 4131.89 | 0.92 | -0.09 | 79270.70 | 22946.99 | 0.29 | -1.24 |
| | N | | | 43.00 | 43.00 | 43.00 | 43.00 | 43.00 | 43.00 | 43.00 | 43.00 | 43.00 | 43.00 | 43.00 | 43.00 |
| | ometr | | | 138.89 | 137.85 | 0.99 | NA | 5200.09 | 5186.00 | 1.00 | NA | 30440.45 | 29984.99 | 0.99 | NA |
| | ithmet | | | 139.80 | 139.17 | 0.99 | -0.01 | 5229.98 | 5218.87 | 1.00 | 0.00 | 32507.57 | 32737.24 | 1.09 | -0.02 |
| Star | ndard o | | on | 16.16 | 19.24 | 0.06 | 0.06 | 562.73 | 587.42 | 0.05 | 0.05 | 14364.09 | 14856.68 | 0.48 | 0.48 |
| | cv | | | 11.56 | 13.83 | 6.15 | -817.63 | 10.76 | 11.26 | 4.99 | -1837.73 | 44.19 | 45.38 | 44.31 | -3205.24 |
| M | inumu | | ė | 103.11 | 89.15 | 0.85 | -0.17 | 4063.30 | 3869.62 | 0.87 | -0.13 | 17477.08 | 14997.88 | 0.29 | -1.24 |
| | Med | | | 137.40 | 135.62 | 0.99 | -0.01 | 5312.71 | 5305.90 | 1.00 | 0.00 | 28249.64 | 28138.76 | 1.02 | 0.02 |
| M | aximur | m valu | e | 176.09 | 190.12 | 1.14 | 0.13 | 6382.19 | 6725.22 | 1.12 | 0.12 | 93377.86 | 75099.89 | 2.41 | 0.88 |



Table A2.5. Levothyroxine Pharmacokinetic Parameters Results, unadjusted value.

| | | | | Fo | rm | | | |
|---|---|---|---|---|---|---|---|---|
| Variable | | Eutirox® appro | ved formulation | on (A) | | Eutirox® tes | t formulation | (B) |
| variable | N | Arithmetic | Standard | %CV | N | Arithmetic | Standard | %CV |
| | | Mean | Deviation | /0CV | IN | Mean | Deviation | /0CV |
| Extrapolated AUC (%) | 43 | 81.90 | 5.81 | 7.10 | 43 | 81.07 | 7.66 | 9.44 |
| $AUC_{0-\infty}$ (ng*h/mL) | 43 | 32507.57 | 14364.09 | 44.19 | 43 | 32737.24 | 14856.68 | 45.38 |
| AUC <sub>0-t</sub> (ng*h/mL) | 43 | 5229.98 | 562.73 | 10.76 | 43 | 5218.87 | 587.42 | 11.26 |
| CI/F (mL/h) | 43 | 20.72 | 6.06 | 29.25 | 43 | 21.63 | 8.24 | 38.10 |
| C <sub>max</sub> (ng/mL) | 43 | 139.80 | 16.16 | 11.56 | 43 | 139.17 | 19.24 | 13.83 |
| t 1/2 (h) | 43 | 186.40 | 96.26 | 51.64 | 43 | 189.10 | 102.07 | 53.98 |
| Kel (1/h) | 43 | 0.00 | 0.00 | 36.92 | 43 | 0.00 | 0.00 | 45.83 |
| MRT (h) | 43 | 270.54 | 138.37 | 51.15 | 43 | 274.33 | 147.48 | 53.76 |
| T <sub>lag</sub> (h) | 43 | 0.00 | 0.00 | NA | 43 | 0.00 | 0.00 | NA |
| T <sub>max</sub> (h) | 43 | 3.52 | 1.19 | 33.96 | 43 | 3.50 | 1.14 | 32.58 |
| Vd/F (L) | 43 | 4.88 | 0.70 — | 14.32 | 43 | 4.87 | 0.66 | 13.62 |

NA: Not applicable

Table A2.6. ANOVA table for the analysis of the unadjusted levothyroxine logarithmicallytransformed pharmacokinetic parameters (Ln).

| Assessed<br>Variable | Source of Variation | Degrees of<br>Freedom | Square Sum | Squared Means | F Value | P Value | Criterion<br>(P > 0.05) |
|---|---|---|---|---|---|---|---|
| Ln(C <sub>max</sub> ) | Sequence | 1 | 0.07 | 0.07 | 2.15 | 0.15 | Cumple |
| Ln(C <sub>max</sub> ) | Sequence*Volunteer | 41 | 1.25 | 0.03 | | | No aplica |
| Ln(C <sub>max</sub> ) | Form | 1 | 1.22 x 10 <sup>-3</sup> | 1.22 x 10 <sup>-3</sup> | 0.64 | 0.43 | Cumple |
| Ln(C <sub>max</sub> ) | Period | 1 | 1.31 x 10 <sup>-3</sup> | 1.31 x 10 <sup>-3</sup> | 0.69 | 0.41 | Cumple |
| Ln(C <sub>max</sub> ) | Error | 41 | 7.86 x 10 <sup>-2</sup> | 1.92 x 10 <sup>-3</sup> | | | No aplica |
| Ln(AUC <sub>0+</sub> ) | Sequence | 1 | 2.69 x 10 <sup>-2</sup> | 2.69 x 10 <sup>-2</sup> | 1.14 | 0.29 | Cumple |
| Ln(AUC <sub>0+</sub> ) | Sequence*Volunteer | 41 | 0.97 | 2.36 x 10 <sup>-2</sup> | | | No aplica |
| Ln(AUC₀+) | Form | 1 | 1.58 x 10 <sup>-4</sup> | 1.58 x 10 <sup>-4</sup> | 0.12 | 0.73 | Cumple |
| Ln(AUC <sub>0+</sub> ) | Period | 1 | 9.64 x 10 <sup>-5</sup> | 9.64 x 10 <sup>-5</sup> | 0.08 | 0.78 | Cumple |
| Ln(AUC <sub>0+</sub> ) | Error | 41 | 5.21 x 10 <sup>-2</sup> | 1.27 x 10 <sup>-3</sup> | | | No aplica |
| Ln(AUC <sub>0-∞</sub> ) | Sequence | 1 | 0.16 | 0.16 | 0.92 | 0.34 | Cumple |
| Ln(AUC <sub>0-∞</sub> ) | Sequence*Volunteer | 41 | 7.00 | 0.17 | | | No aplica |
| Ln(AUC <sub>0∞</sub> ) | Form | 1 | 4.89 x 10 <sup>-3</sup> | 4.89 x 10 <sup>-3</sup> | 0.04 | 0.84 | Cumple |
| Ln(AUC <sub>0.22</sub> ) | Period | 1 | 0.06 | 0.06 | 0.55 | 0.46 | Cumple |
| Ln(AUC <sub>0∞</sub> ) | Error | 41 | 4.84 | 0.12 | | | No aplica |

| La | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|-----|----------------------|---------|-------------|
| PPD | ANALI HOAL ONI | Version | 1.0 |

Table A2.7 shows the results of the bioequivalence statistics for the levothyroxine logarithmically-transformed pharmacokinetic unadjusted data

Table A2.7 Statistics of the Levothyroxine Bioequivalence Determination.

| Parameter | | onfidence | | mann's<br>d-side t | Power | Acceptance | Meets<br>the |
|---|---|---|---|---|---|---|---|
| - didinotor | Inte | erval | P < 80 % | P<br>> 125 % | (%) | Criterion | Criterion |
| LnCmax | 97.70 | 100.85 | 0.00 | 0.00 | 100.00 | (80-125) | YES |
| LnAUC <sub>0-t</sub> | 98.45 | 101.03 | 0.00 | 0.00 | 99.98 | (80-125) | YES |

Table A3.1 Table of individual concentrations corresponding to adjusted levothyroxine, including predose greater than 5% (reference drug [A]). N = 43 subjects.

| Form | Volunteer | | | | | | | | | | | | Time | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 0.00 | 0.50 | 1.00 | 150 | 2.00 | 2.50 | 3.00 | 3.25 | 3.50 | 3.75 | 4.00 | 4.25 | 4.50 | 4.75 | 5.00 | 5.50 | 6.00 | 6.50 | 8.00 | 10.00 | 12.00 | 24.00 | 36.00 | 48.00 |
| A | 1 | 0.00 | 0.00 | 18.08 | 25.76 | 33.62 | 59.36 | 73.07 | 77.18 | 83.03 | 73.97 | 96.39 | 98.33 | 89.28 | 90.42 | 86.81 | 79.36 | 70.08 | 72.76 | 66.78 | 58.76 | 64.49 | 57.99 | 50.27 | 46.44 |
| A | 2 | 0.95 | 3.10 | 19.25 | 33.71 | 42.76 | 45.60 | 46.32 | 54.44 | 52.37 | 51.29 | 49.24 | 55.16 | 53.62 | 49.56 | 59.08 | 45.50 | 44.61 | 44.62 | 45.91 | 44.13 | 38.01 | 34.60 | 38.14 | 39.62 |
| A | 3 | 0.04 | 5.41 | 45.45 | 55.09 | 61.00 | 45.19 | 40.08 | 52.74 | 36.22 | 32.34 | 40.98 | 43.74 | 42.37 | 35.11 | 31.35 | 32.92 | 32.87 | 40.23 | 29.26 | 23.10 | 27.04 | 22.63 | 22.89 | 19.76 |
| A | 4 | 0.24 | 2.22 | 15.74 | 39.37 | 55.52 | 56.51 | 59.29 | 52.39 | 51.70 | 67.12 | 49.86 | 62.41 | 59.12 | 47.28 | 48.65 | 51.19 | 41.04 | 45.56 | 47.40 | 37.83 | 38.98 | 30.15 | 29.06 | 23.10 |
| A | 5 | 0.00 | 1.31 | 22.68 | 32.52 | 36.69 | 37.64 | 53.06 | 45.51 | 52.17 | 47.12 | 51.78 | 51.68 | 52.20 | 48.46 | 46.44 | 48.39 | 41.28 | 34.87 | 33.99 | 32.68 | 26.28 | 25.10 | 19.42 | 28.01 |
| A | 6 | 0.00 | 2.13 | 4.16 | 21.55 | 49.91 | 64.49 | 63.06 | 57.44 | 57.84 | 58.86 | 49.98 | 57.66 | 51.39 | 55.90 | 53.28 | 53.25 | 52.89 | 55.A5 | 53.91 | 44.06 | 42.77 | 36.80 | 32.71 | 28.96 |
| A | 7 | 0.00 | 3.04 | 16.50 | 28.04 | 29.99 | 34.44 | 57.68 | 48.23 | 54.39 | 64.47 | 56.21 | 63.47 | 49.44 | 53.45 | 41.29 | 40.28 | 43.31 | 41.76 | 53.16 | 33.20 | 27.71 | 38.43 | 28.84 | 30.49 |
| A | 8 | 0.00 | 3.03 | 31.05 | 44.07 | 58.34 | 64.72 | 57.08 | 63.33 | 49.74 | 58.34 | 60.40 | 60.22 | 57.79 | 55.20 | 61.69 | 54.74 | 61.39 | 47.24 | 51.10 | 45.10 | 39.51 | 32.40 | 24.89 | 23.33 |
| A | 9 | 0.00 | 7.14 | 11.53 | 15.62 | 12.87 | 19.26 | 26.65 | 47.89 | 54.01 | 64.75 | 59.99 | 77.35 | 76.86 | 84.71 | 80.43 | 71.34 | 71.58 | 62.30 | 60.40 | 49.55 | 39.32 | 46.23 | 37.58 | 38.79 |
| A | 10 | 0.00 | 0.00 | 1.86 | 36.34 | 52.20 | 58.30 | 62.78 | 71.37 | 70.04 | 56.75 | 74.84 | 79.08 | 75.58 | 81.77 | 61.19 | 74.82 | 63.72 | 58.42 | 62.81 | 55.65 | 48.99 | 41.36 | 31.64 | 30.82 |
| A | 11 | 0.00 | 0.00 | 14.75 | 27.54 | 68.86 | 40.49 | 52.38 | 55.51 | 51.51 | 55.85 | 61.42 | 60.76 | 64.98 | 59.66 | 58.66 | 58.59 | 51.79 | 41.77 | 39.55 | 36.52 | 30.60 | 40.18 | 43.35 | 25.62 |
| A | 12 | 0.00 | 6.19 | 26.38 | 50.30 | 54.73 | 63.00 | 69.82 | 61.41 | 63.27 | 65.19 | 60.02 | 65.76 | 56.83 | 51.26 | 52.95 | 55.53 | 54.36 | 47.84 | 57.10 | 45.06 | 42.70 | 40.25 | 32.52 | 29.49 |
| A | 13<br>14 | 0.00 | 7.13 | 29.24 | 59.72 | 46.49 | 62.06 | 60.77 | 60.84 | 58.21 | 50.85<br>59.44 | 40.75 | 60.79 | 53.75<br>56.87 | 54.37<br>69.84 | 50.33 | 55.28<br>55.00 | 52.64<br>58.65 | 41.59 | 48.04 | 47.04 | 35.90<br>48.92 | 42.43 | 43.72 | 34.56 |
| A | 15 | 0.22 | 0.00 | 24.00<br>5.43 | 43.40 | 13.29 | 61.37<br>25.09 | 54.90<br>22.85 | 63.59 | 43.23 | 41.27 | 62.16 | 63.16<br>40.83 | 56.87<br>44.14 | 40.51 | 61.81<br>51.95 | 55.00<br>42.80 | 39.20 | 55.78<br>34.20 | 58.93<br>31.48 | 29.87<br>41.79 | 48.92<br>36.83 | 40.85 | 32.00<br>15.76 | 31.63<br>25.49 |
| A | 16 | 0.00 | 8.00 | 26.69 | 33.12 | 35.23 | 55.66 | 56.88 | 66.06 | 67.07 | 61.11 | 56.07 | 49.65 | 49.91 | 98.86 | 48.93 | 60.42 | 55.01 | 53.01 | 37.59 | 40.86 | 36.36 | 30.10 | 20.19 | 29.89 |
| A | 17 | 0.00 | 4.78 | 11.47 | 14.59 | 24.96 | 42.11 | 66.14 | 60.41 | 54.70 | 50.91 | 59.30 | 62.16 | 46.06 | 52.30 | 58.93 | 50.21 | 49.20 | 54.71 | 54.37 | 43.89 | 41.10 | 36.45 | 23.89 | 14.73 |
| A | 18 | 0.00 | 2.12 | 33.99 | 44.44 | 52.12 | 58.14 | 63.81 | 61.51 | 60.94 | 67.71 | 63.07 | 61.82 | 58.70 | 56.20 | 55.17 | 58.14 | 56.91 | 47.85 | 48.84 | 42.38 | 45.57 | 39.15 | 29.68 | 29.96 |
| A | 19 | 0.09 | 4.33 | 43.58 | 51.94 | 49.37 | 59.52 | 60.20 | 58.16 | 64.98 | 60.57 | 49.71 | 73.11 | 55.00 | 52.70 | 51.18 | 55.10 | 42.80 | 45.87 | 49.52 | 39.35 | 39.24 | 50.09 | 35.00 | 34.00 |
| A | 20 | 0.00 | 6.32 | 34.84 | 68.56 | 71.10 | 66.47 | 74.56 | 67.80 | 74.61 | 68.09 | 68.12 | 67.97 | 64.24 | 63.56 | 67.60 | 67.08 | 59.46 | 56.90 | 60.97 | 49.31 | 44.45 | 48.93 | 49.42 | 37.82 |
| A | 21 | 0.00 | 2.99 | 27.13 | 56.35 | 53.46 | 61.00 | 68.61 | 64.96 | 62.32 | 62.87 | 68.94 | 65.30 | 65.99 | 60.89 | 58.27 | 57.45 | 43.04 | 48.99 | 54.87 | 38.81 | 35.62 | 40.28 | 34.92 | 32.53 |
| A | 22 | 0.00 | 0.00 | 5.47 | 10.20 | 13.43 | 18.87 | 24.83 | 24.02 | 34.94 | 35.63 | 30.05 | 32.89 | 50.81 | 27.92 | 26.94 | 30.33 | 31.08 | 30.71 | 24.96 | 31.68 | 24.79 | 24.17 | 23.12 | 14.56 |
| A | 23 | 0.00 | 2.03 | 36.97 | 47.98 | 46.30 | 49.23 | 47.93 | 48.24 | 44.80 | 50.16 | 45.70 | 48.89 | 45.05 | 37.36 | 44.33 | 40.72 | 37.82 | 34.38 | 36.27 | 28.80 | 21.73 | 25.25 | 26.87 | 19.00 |
| A | 24 | 0.00 | 0.00 | 23.24 | 45.18 | 53.90 | 75.62 | 66.74 | 63.45 | 71.36 | 69.87 | 65.15 | 66.94 | 55.11 | 53.43 | 49.25 | 55.26 | 46.69 | 41.32 | 41.62 | 34.62 | 35.28 | 39.99 | 22.34 | 19.02 |
| A | 25 | 0.00 | 0.00 | 32.21 | 53.96 | 47.94 | 53.88 | 29.00 | 43.37 | 37.39 | 37.45 | 41.45 | 59.68 | 41.38 | 45.81 | 35.74 | 42.69 | 43.87 | 40,04 | 38.76 | 29.82 | 26.81 | 24.73 | 26.95 | 26.58 |
| A | 26 | 3.32 | 4.41 | 10.30 | 27.04 | 37.86 | 49.47 | 40.82 | 46.52 | 36.61 | 42.67 | 34.47 | 39.69 | 35.68 | 30.91 | 36.29 | 43.15 | 35.12 | 42.01 | 51.65 | 37.41 | 33.72 | 36.45 | 34.34 | 25.45 |
| A | 27 | 0.65 | 0.00 | 17.31 | 34.50 | 41.84 | 42.94 | 48.06 | 46.90 | 44.91 | 46.60 | 42.51 | 47.33 | 40.83 | 33.39 | 36.48 | 42.11 | 42.24 | 39.78 | 37.72 | 36.08 | 30.58 | 29.83 | 23.78 | 23.70 |
| A | 28 | 0.00 | 5.77 | 15.58 | 47.72 | 61.94 | 68.74 | 121.16 | 65.30 | 80.02 | 71.97 | 68.57 | 57.51 | 63.91 | 52.81 | 77.31 | 46.12 | 54.33 | 56.03 | 52.65 | 51.64 | 51.99 | 41.44 | 56.27 | 41.17 |
| A | 29 | 0.74 | 12.68 | 11.63 | 31.89 | 56.96 | 65.35 | 39.34 | 55.86 | 54.04 | 41.67 | 55.05 | 53.18 | 50.24 | 46.79 | 41.93 | 42.84 | 36.96 | 36,07 | 49.20 | 36.21 | 31.70 | 41.18 | 28.21 | 20.81 |
| A | 30 | 1.66 | 4.82 | 24.29 | 33.91 | 29.16 | 52.40 | 32.50 | 68.88 | 55.06 | 63.72 | 53.08 | 58.09 | 57.83 | 52.74 | 51.52 | 49.09 | 43.36 | 40.22 | 48.23 | 42.74 | 42.01 | 40.28 | 48.76 | 37.67 |
| A | 31 | 0.00 | 4.57 | 9.30 | 34.95 | 34.96 | 45.12 | 39.65 | 40.99 | 39.33 | 39.99 | 38.43 | 45.02 | 49.54 | 48.10 | 36.09 | 23.02 | 30.45 | 31.71 | 32.90 | 17.75 | 18.83 | 27.31 | 10.97 | 15.01 |
| A | 32 | 3.18 | 6.59 | 50.40 | 53.47 | 61.04 | 43.57 | 39.55 | 38.07 | 39.94 | 44.61 | 36.54 | 42.04 | 36.95 | 3454 | 35.68 | 39.39 | 33.26 | 34.52 | 34.90 | 38.95 | 25.06 | 30.26 | 30.86 | 30.84 |
| A | 33 | 3.27 | 8.57 | 37.56 | 45.26 | 57.55 | 76.35 | 71.51 | 77.89 | 82.25 | 76.90 | 79.66 | 86.93 | 85.56 | 73.60 | 81.06 | 85.56 | 65.23 | 73.26 | 64.06 | 59.41 | 64.31 | 50.72 | 58.18 | 55.61 |
| A | 34 | 0.00 | 0.00 | 9.17 | 12.53 | 22.41 | 25.61 | 40.22 | 48.91 | 60.92 | 47.62 | 48.59 | 57.50 | 43.24 | 44.53 | 38.47 | 42.39 | 36.95 | 27.96 | 40.18 | 31.81 | 30.39 | 36.36 | 22.47 | 26.44 |
| A | 35 | 0.00 | 3.18 | 38.87 | 59.17 | 59.46 | 54.39 | 53.87 | 48.81 | 45.85 | 45.87 | 46.05 | 54.19 | 44.10 | 31.48 | 43.13 | 45.66 | 41.79 | 43.02 | 47.03 | 48.06 | 34.11 | 39.58 | 36.52 | 31.71 |
| A | 36 | 3.49 | 4.87 | 51.03 | 62.19 | 56.79 | 52.03 | 65.33 | 74.82 | 61.33 | 64.84 | 57.09 | 59.12 | 52.43 | 54.17 | 51.54 | 51.65 | 46.36 | 45.53 | 41.02 | 42.03 | 35.39 | 15.52 | 29.58 | 30.34 |
| A | 37 | 0.00 | 0.00 | 36.37 | 47.22 | 60.30 | 55.05 | 54.15 | 57.78 | 59.60 | 55.54 | 52.78 | 54.60 | 52.35 | 47.95 | 49.44 | 53.06 | 53.52 | 47.A5 | 48.10 | 38.77 | 42.02 | 36.21 | 33.56 | 29.36 |
| A | 39 | 2.71 | 7.98 | 81.95 | 90.27 | 85.98 | 100.38 | 86.78 | 82.14 | 79.05 | 82.19 | 83.16 | 89.05 | 86.73 | 78.73 | 73.45 | 85.70 | 79.63 | 77.27 | 68.79 | 68.89 | 64.91 | 51.98 | 47.47 | 49.11 |
| A | 40 | 9.72 | 5.85 | 19.24 | 30.92 | 38.85 | 73.16 | 76.71 | 80.95 | 81.27 | 85.18 | 84.23 | 90.55 | 87.54 | 83.46 | 86.80 | 64.95 | 86.35 | 79.86 | 79.95 | 70.52 | 66.20 | 48.16 | 49.29 | 34.43 |
| A | 41 | 0.00 | 3.33 | 36.99 | 51.23 | 57.14 | 52.66 | 64.01 | 64.35 | 65.86 | 59.42 | 61.18 | 62.57 | 72.78 | 52.99 | 46.20 | 40.05 | 52.40 | 46.A2 | 48.37 | 39.45 | 32.90 | 46.04 | 27.53 | 30.69 |
| A | 42 | 0.00 | 2.16 | 6.44 | 17.24 | 24.25 | 20.91 | 22.88 | 30.64 | 39.15 | 40.03 | 40.06 | 44.51 | 42.99 | 38.71 | 35.24 | 35.24 | 32.46 | 34.83 | 33.72 | 23.89 | 22.85 | 25.08 | 27.12 | 27.15 |
| A | 43 | 0.00 | 9.75 | 0.00 | 51.13 | 47.33 | 44.91 | 48.87 | 41.58 | 43.98 | 45.80 | 46.19 | 49.97 | 43.30 | 45.06 | 44.44 | 39.67 | 40.08 | 35.99 | 44.86 | 30.43 | 31.86 | 29.09 | 34.59 | 23.61 |
| A | 44 | 1.00 | 4.89 | 22.37 | 35.41 | 45.79 | 51.87 | 48.87 | 48.92 | 46.34 | 44.27 | 43.36 | 50.47 | 44.87 | 40.22 | 41.19 | 38.69 | 39.78 | 35.92 | 30.08 | 30.31 | 30.37 | 27.85 | 26.68 | 26.28 |
| | etic Mean | 0.76 | 3.81 | 24.20 | 39.66 | 46.34 | 52.39 | 54.72 | 56.28 | 56.36 | 56.07 | 55.10 | 59.79 | 55.98 | 52.95 | 52.29 | 51.27 | 48.73 | 46.65 | 47.46 | 40.66 | 37.87 | 36.39 | 32.59 | 29.62 |
| | d Deviation | 1.75 | 3.08 | 16.08 | 17.36 | 16.00<br>34.52 | 16.33 | 18.63<br>34.04 | 13.46 | 13.52 | 12.82<br>22.87 | 14.49 | 14.14 | 13.92<br>24.86 | 15.08<br>28.48 | 14.89 | 13.83 | 12.98<br>26.64 | 12.44 | 11.90 | 11.07 | 11.57 | 9.34 | 10.70 | 8.70<br>29.39 |
| , | KCV | 231.17 | 80.71 | 66.46 | 43.78 | 34.52 | 31.17 | 34.04 | 23.91 | 23.99 | 22.87 | 26.30 | 23.65 | 24.86 | 28.48 | 28.47 | 26.98 | 25.54 | 26.66 | 25.06 | 27.24 | 30.56 | 25.68 | 32.83 | 29.39 |



Table A3.2 Table of individual concentrations corresponding to levothyroxine, including predose greater than 5% (reference drug). N = 43 subjects.

| | | | | | | | _ | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Form | Volunteer | | | | | | | | | | | | Time | | | | | | | | | | | | |
| ruill | YVIUILEG | 0.00 | 0.50 | 1.00 | 150 | 2.00 | 2.50 | 3.00 | 3.25 | 3.50 | 3.75 | 4.00 | 4.25 | 4.50 | 4.75 | 5.00 | 5.50 | 6.00 | 6.50 | 8.00 | 10.00 | 12.00 | 24.00 | 36.00 | 48.00 |
| В | 1 | 0.36 | 2.79 | 17.91 | 31.20 | 40.46 | 46.99 | 54.85 | 69.43 | 65.89 | 84.97 | 82.64 | 75.96 | 75.05 | 74.65 | 73.40 | 58.34 | 55.21 | 49.74 | 58.80 | 50.79 | 43.11 | 40.03 | 41.77 | 21.93 |
| В | 2 | 0.00 | 3.77 | 34.31 | 49.71 | 55.52 | 52.76 | 57.53 | 48.95 | 52.17 | 46.50 | 47.92 | 52.87 | 49.14 | 47.08 | 40.16 | 42.16 | 59.26 | 36.21 | 33.32 | 27.19 | 30.20 | 28.83 | 23.76 | 18.41 |
| В | 3 | 0.00 | 4.56 | 42.17 | 56.41 | 39.98 | 44.50 | 35.97 | 34.31 | 41.07 | 39.67 | 24.39 | 34.59 | 48.09 | 36.40 | 36.96 | 24.59 | 25.43 | 20.77 | 6.44 | 12.78 | 13.72 | 20.74 | 27.56 | 24.82 |
| В | 4 | 0.00 | 5.29 | 16.63 | 39.25 | 54.71 | 55.69 | 63.95 | 60.72 | 55.17 | 54.09 | 53.89 | 52.11 | 47.96 | 42.13 | 41.46 | 42.58 | 43.26 | 40.44 | 41.92 | 37.87 | 37.55 | 30.28 | 31.89 | 19.31 |
| В | 5 | 0.00 | 3.60 | 5.15 | 9.40 | 9.21 | 13.56 | 15.13 | 20.55 | 12.57 | 26.79 | 23.36 | 37.49 | 41.91 | 59.02 | 53.80 | 47.48 | 40.41 | 42.82 | 37.95 | 30.38 | 23.75 | 29.37 | 27.62 | 24.90 |
| В | 6 | 0.24 | 0.00 | 4.78 | 15.29 | 14.54 | 16.90 | 16.01 | 25.48 | 28.34 | 33.35 | 39.92 | 48.64 | 45.53 | 40.81 | 33.57 | 38.87 | 34.07 | 33.18 | 29.28 | 28.03 | 30.25 | 25.72 | 17.88 | 23.41 |
| В | 7 | | | | | | | | 55.04 | 55.85 | | | | | | | | | 49.95 | | h | | | | |
| _ | _ | 0.53 | 8.73 | 36.06 | 41.76 | 49.65 | 54.84 | 69.43 | ***** | | 42.18 | 45.25 | 46.82 | 50.46 | 45.27 | 55.71 | 51.90 | 50.42 | 00000 | 43.06 | 45.35 | 38.26 | 40.62 | 36.32 | 39.65 |
| В | 8 | 0.00 | 22.49 | 48.49 | 61.64 | 66.18 | 57.51 | 58.67 | 60.60 | 59.30 | 5333 | 53.95 | 60.19 | 52.90 | 54.45 | 47.68 | 53.99 | 49.81 | 44.60 | 40.06 | 38.55 | 37.62 | 31.20 | 44.63 | 31.79 |
| В | 9 | 2.13 | 0.00 | 25.40 | 43.56 | 69.04 | 86.57 | 93.54 | 87.80 | 97.45 | 98.59 | 101.74 | 104.57 | 94.06 | 96.22 | 97.71 | 95.00 | 96.72 | 80.81 | 73.49 | 63.24 | 63.56 | 42.01 | 56.25 | 35.96 |
| В | 10 | 0.00 | 1.43 | 20.93 | 48.51 | 67.80 | 73.54 | 79.88 | 97.25 | 96.00 | 79.94 | 74.34 | 82.17 | 85.29 | 84.34 | 89.85 | 70.20 | 82.59 | 77.27 | 76.82 | 57.96 | 74.36 | 52.40 | 44.80 | 41.12 |
| В | 11 | 0.39 | 4.73 | 23.43 | 59.64 | 67.87 | 71.66 | 67.73 | 72.27 | 69.20 | 62.75 | 61.72 | 63.41 | 57.79 | 63.43 | 62.11 | 56.08 | 64.38 | 62.71 | 53.65 | 51.28 | 41.67 | 49.91 | 50.30 | 32.51 |
| В | 12 | 0.00 | 1.73 | 24.09 | 40.62 | 54.56 | 63.04 | 54.30 | 58.19 | 57.49 | 57.61 | 60.91 | 69.15 | 55.95 | 56.19 | 53.60 | 48.72 | 52.36 | 44.18 | 53.11 | 38.15 | 35.54 | 48.57 | 40.50 | 27.35 |
| В | 13 | 0.00 | 4.26 | 32.89 | 49.68 | 47.43 | 51.61 | 49.51 | 42.51 | 46.20 | 36.71 | 46.03 | 51.70 | 46.62 | 43.99 | 42.89 | 43.98 | 42.76 | 30.11 | 40.77 | 31.17 | 32.40 | 19.77 | 37.89 | 34.95 |
| В | 14 | 0.20 | 6.14 | 33.16 | 53.17 | 55.00 | 63.97 | 53.37 | 56.39 | 60.64 | 61.77 | 62.86 | 63.12 | 63.19 | 61.68 | 61.09 | 68.12 | 65.83 | 60.17 | 62.76 | 55.44 | 52.45 | 40.06 | 50.94 | 35.83 |
| В | 15 | 0.00 | 1.87 | 19.48 | 33.62 | 24.27 | 41.18 | 46.90 | 50.19 | 44.68 | 45.12 | 44.01 | 53.99 | 4432 | 54.48 | 39.59 | 38.31 | 47.15 | 39.17 | 53.60 | 39.42 | 38.73 | 31.88 | 33.06 | 36.67 |
| В | 16 | 6.49 | 2.41 | 17.61 | 33.54 | 55.08 | 45.07 | 44.78 | 43.47 | 4131 | 39.68 | 43.17 | 48.86 | 45.04 | 41.85 | 39.92 | 45.29 | 36.25 | 41.96 | 38.01 | 34.67 | 29.87 | 43.55 | 27.70 | 20.88 |
| В | 17 | 0.00 | 2.89 | 17.25 | 28.91 | 44.51 | 50.85 | 52.11 | 42.23 | 68.33 | 66.23 | 58.97 | 67.80 | 63.88 | 51.40 | 51.40 | 51.97 | 45.41 | 38.59 | 55.86 | 42.85 | 36.91 | 34.72 | 34.95 | 11.84 |
| В | 18 | 0.00 | 7.27 | 35.61 | 47.18 | 54.82 | 65.71 | 68.11 | 62.74 | 63.33 | 61.82 | 60.32 | 65.35 | 57.65 | 54.51 | 55.82 | 53.49 | 51.41 | 51.62 | 53.01 | 51.62 | 47.24 | 37.26 | 34.72 | 30.84 |
| В | 19 | 0.30 | 2.50 | 29.64 | 42.62 | 56.02 | 41.53 | 52.48 | 46.66 | 42.04 | 38.77 | 36.36 | 50.90 | 4734 | 47.19 | 43.10 | 45.24 | 55.43 | 49.00 | 41.15 | 38.82 | 37.83 | 29.34 | 23.85 | 25.47 |
| В | 20 | 0.01 | 7.07 | 39.40 | 53.19 | 56.06 | 54.98 | 59.97 | 56.63 | 49.46 | 49.00 | 48.20 | 60.44 | 48.90 | 42.34 | 37.45 | 36.18 | 39.47 | 39.90 | 43.58 | 32.28 | 24.00 | 29.55 | 33.42 | 23.14 |
| В | 21 | 3.56 | 15.88 | 35.26 | 58.93 | 59.18 | 66.13 | 66.40 | 59.28 | 65.38 | 62.22 | 62.60 | 67.03 | 61.85 | 49.99 | 53.00 | 53.79 | 54.12 | 59.51 | 64.38 | 46.40 | 43.97 | 39.84 | 41.86 | 24.83 |
| В | 22 | 1.39 | 0.00 | 18.07 | 34.38 | 30.99 | 38.85 | 43.21 | 42.46 | 37.15 | 39.86 | 40.72 | 37.81 | 36.49 | 32.74 | 43.65 | 35.78 | 37.49 | 37.29 | 30.36 | 32.87 | 28.72 | 28.66 | 24.22 | 26.61 |
| В | 23 | 1.89 | 11.64 | 49.76 | 70.84 | 68.59 | 73.24 | 60.25 | 66.61 | 61.33 | 60.29 | 61.24 | 67.83 | 61.56 | 54.26 | 53,77 | 49.82 | 48.79 | 44.34 | 40.53 | 40.50 | 38.97 | 39.37 | 32.88 | 30.72 |
| В | 24 | 0.76 | 0.00 | 0.00 | 0.00 | 934 | 11.89 | 16.72 | 10.93 | 12.35 | 18.55 | 39.45 | 55.64 | 54.80 | 60.54 | 51.26 | 45.55 | 29.73 | 33.85 | 36.69 | 21.42 | 26.65 | 34.25 | 24.89 | 26.37 |
| В | 25 | 0.00 | 20.25 | 50.91 | 60.79 | 55.35 | 47.89 | 56.13 | 42.26 | 55.71 | 62.69 | 42.97 | 51.28 | 40.88 | 54.72 | 45.57 | 57.57 | 41.01 | 53.43 | 44.70 | 50.85 | 34.92 | 47.30 | 31.89 | 26.78 |
| В | 26 | 0.00 | 0.00 | 11.65 | 25.16 | 35.14 | 51.11 | 54.58 | 50.03 | 49.19 | 53.50 | 48.08 | 46.87 | 46.09 | 46.22 | 47.47 | 45.86 | 40.73 | 45.93 | 49.16 | 42.23 | 41.84 | 36.91 | 35.69 | 25.87 |
| В | 27 | 0.00 | 1.22 | 26.36 | 39.15 | 42.23 | 49.84 | 44.22 | 42.60 | 46.63 | 45.42 | 51.14 | 52.34 | 42.09 | 38.86 | 45.57 | 39.84 | 46.78 | 32.39 | 40.71 | 30.76 | 30.65 | 29.61 | 24.19 | 14.63 |
| В | 28 | 0.00 | 10.78 | 40.05 | 31.95 | 44.49 | 35.97 | 105.75 | 93.10 | 57.87 | 91.63 | 58.16 | 46.44 | 69.72 | 71.26 | 80.92 | 49.71 | 12.65 | 45.55 | 25.46 | 34.32 | 40.80 | 41.93 | 32.50 | 24.17 |
| В | | 0.00 | | | | | | | | 47.14 | | 44.35 | | 57.37 | | | | | | | | | | | |
| _ | 29 | | 0.46 | 0.00 | 0.00 | 36.95 | 40.43 | 41.45 | 40.61 | | 44.64 | | 60.17 | 41.41 | 5235 | 49.79 | 49.87 | 45.56 | 39.91 | 44.89 | 26.18 | 37.92 | 34.80 | 0.00 | 6.82 |
| B | 30 | 3.11 | 3.63 | 25.34 | 46.10 | 42.17 | 53.40 | 36.85 | 65.54 | 54.82 | 71.68 | 55.55 | 49.89 | 49.80 | 47.11 | 46.88 | 43.70 | 41.96 | 40.53 | 37.15 | 36.33 | 35.24 | 38.98 | 41.39 | 34.86 |
| H | 31 | 0.00 | 3.80 | 33.71 | 46.73 | 52.87 | 51.74 | 62.01 | 49.53 | 53.25 | 50.33 | 46.42 | 46.59 | 48.00 | 42.24 | 56.14 | 45.41 | 55.85 | 38.69 | 40.30 | 32.69 | 30.85 | 35.30 | 38.03 | 24.01 |
| В | 32 | 0.00 | 9.47 | 4.4 | 56.18 | 47.62 | 56.23 | 57.42 | 50.04 | 4453 | 62.17 | 38.50 | 48.71 | 47.84 | 42.93 | 35.65 | 38.00 | 42.37 | 35.78 | 39.37 | 30.91 | 32.49 | 36.47 | 24.68 | 22.33 |
| В | 33 | 0.00 | 20.22 | 62.72 | 82.18 | 79.02 | 69.15 | 69.81 | 61.80 | 61.79 | 62.31 | 64.57 | 66.39 | 66.69 | 60.32 | 6134 | 53.11 | 5458 | 54.40 | 52.44 | 42.43 | 45.74 | 43.60 | 28.55 | 30.88 |
| В | 34 | 1.28 | 10.99 | 30.74 | 50.42 | 63.83 | 70.24 | 58.56 | 55.87 | 57.01 | 58.08 | 59.78 | 68.78 | 57.30 | 51.35 | 47.19 | 41.26 | 47.67 | 40.39 | 36.00 | 28.07 | 38.33 | 29.43 | 24.24 | 17.34 |
| В | 35 | 0.17 | 0.00 | 0.00 | 16.04 | 20.92 | 49.01 | 52.07 | 36.70 | 41.30 | 49.07 | 28.33 | 38.25 | 44.89 | 44.85 | 39.72 | | 51.67 | | - | 26.76 | 35.85 | | - | 41.01 |
| В | 36 | 1.83 | 17.66 | 60.21 | 64.87 | 70.08 | 66.77 | 45.41 | 52.85 | 63.36 | 47.07 | 57.71 | 63.12 | 54.05 | 56.11 | 5051 | 50.47 | 40.10 | 42.39 | 46.20 | 42.17 | 32.18 | 29.81 | 35.13 | 36.58 |
| В | 37 | 0.00 | 6.08 | 3.52 | 25.64 | 40.87 | 52.82 | 60.91 | 61.67 | 62.32 | 64.41 | 57.07 | 61.67 | 51.50 | 54.86 | 57.06 | 68.30 | 54.04 | 50.03 | 46.56 | 45.74 | 43.97 | 43.70 | 37.54 | 39.90 |
| В | 39 | 0.00 | 21.11 | 58.94 | 82.41 | 86.16 | 91.74 | 86.69 | 73.80 | 73.91 | 84.89 | 84.48 | 70.66 | 94.09 | 85.59 | 77.05 | 60.60 | 52.98 | 58.79 | 62.34 | 55.82 | 45.68 | 48.10 | 33.44 | 35.15 |
| В | 40 | 0.00 | 0.00 | 16.31 | 31.43 | 43.30 | 58.76 | 65.02 | 68.52 | 74.09 | 71.22 | 70.39 | 78.08 | 75.35 | 70.39 | 72.83 | 71.95 | 65.40 | 65.58 | 65.92 | 59.63 | 58.56 | 42.80 | 37.96 | 38.58 |
| В | 41 | 0.00 | 14.77 | 39.58 | 62.91 | 57.36 | 79.08 | 49.75 | 52.69 | 57.46 | 38.34 | 54.72 | 63.73 | 47.79 | 41.76 | 36.95 | 59.50 | 40.42 | 34.98 | 63.09 | 26.06 | 40.04 | 32.28 | 25.61 | 17.70 |
| В | 42 | 0.00 | 5.13 | 20.63 | 29.26 | 20.68 | 31.73 | 33.98 | 30.70 | 33.13 | 32.32 | 31.38 | 33.26 | 26.93 | 29.62 | 29.99 | 27.70 | 27.90 | 27.14 | 31.69 | 23.39 | 20.83 | 27.09 | 24.76 | 27.53 |
| В | 43 | 0.98 | 5.77 | 41.87 | 50.89 | 50.10 | 56.81 | 46.08 | 50.09 | 47.69 | 54.80 | 50.80 | 48.40 | 41.95 | 40.31 | 46.32 | 40.53 | 37.32 | 32.31 | 36.35 | 33.93 | 29.34 | 22.89 | 21.13 | 30.42 |
| В | 44 | 0.00 | 5.77 | 37.85 | 47.59 | 41.39 | 37.75 | 41.29 | 37.34 | 38.76 | 39.51 | 36.07 | 41.87 | 43.03 | 39.25 | 36.83 | 30.10 | 39.51 | 33.49 | 34.83 | 27.96 | 28.45 | 28.68 | 16.07 | 27.54 |
| Arithm | etic Mean | 0.60 | 6.47 | 28.66 | 43.09 | 48.40 | 53.33 | 54.62 | 53.17 | 53.55 | 54.51 | 52.43 | 57.09 | 54.47 | 52.68 | 51.69 | 49.01 | 47.59 | 44.77 | 45.18 | 38.26 | 37.47 | 35.68 | 32.10 | 27.71 |
| Standar | dDeviation | 1.26 | 6.44 | 16.39 | 18.77 | 17.54 | 17.09 | 18.05 | 17.42 | 16.73 | 17.20 | 15.71 | 13.97 | 14.10 | 14.12 | 14.93 | 12.97 | 14.27 | 12.34 | 13.45 | 11.31 | 10.93 | 7.92 | 10.24 | 8.06 |
| 9 | KCV | 211.29 | 99.62 | 57.18 | 43.57 | 36.23 | 32.05 | 33.05 | 32.76 | 31.24 | 31.56 | 29.97 | 24.48 | 25.89 | 26.81 | 28.88 | 26.47 | 29.99 | 27.57 | 29.77 | 29.56 | 29.18 | 22.18 | 31.89 | 29.09 |
| _ | | | | | | | | | | | | | | | | | | | | | | | | | |



| ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|----------------------|---------|-------------|
| ANALITICAL ONLI | Version | 1.0 |
| STATISTICAL DOCUMENT | Page | 65 of 68 |

Table A3.3. Descriptive statistics of the values of the levothyroxine concentration in a biological fluid, including predose greater than 5% (N = 43).

| | | Euti | rox® Approve | d formulation | n (A) | Eutirox® test formulation (B) | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time | Arithmetic | | Minimum | Maximum | Standard | CVIII/ | Arithmetic | Madia | Minimum | Maximum | Standard | C10/ |
| | Mean | Median | value | value | Deviation | CV% | Mean | Median | value | value | Deviation | CV% |
| 0.00 | 0.76 | 0.00 | 0.00 | 9.72 | 1.75 | 231.17 | 0.60 | 0.00 | 0.00 | 6.49 | 1.26 | 211.29 |
| 0.50 | 3.81 | 3.33 | 0.00 | 12.68 | 3.08 | 80.71 | 6.47 | 4.56 | 0.00 | 22.49 | 6.44 | 99.62 |
| 1.00 | 24.20 | 22.68 | 0.00 | 81.95 | 16.08 | 66.46 | 28.66 | 29.64 | 0.00 | 62.72 | 16.39 | 57.18 |
| 1.50 | 39.66 | 39.37 | 0.00 | 90.27 | 17.36 | 43.78 | 43.09 | 46.10 | 0.00 | 82.41 | 18.77 | 43.57 |
| 2.00 | 46.34 | 49.00 | 12.87 | 85.98 | 16.00 | 34.52 | 48.40 | 50.10 | 9.21 | 86.16 | 17.54 | 36.23 |
| 2.50 | 52.39 | 53.88 | 18.87 | 100.38 | 16.33 | 31.17 | 53.33 | 52.82 | 11.89 | 91.74 | 17.09 | 32.05 |
| 3.00 | 54.72 | 54.90 | 22.85 | 121.16 | 18.63 | 34.04 | 54.62 | 54.58 | 15.13 | 105.75 | 18.05 | 33.05 |
| 3.25 | 56.28 | 57.44 | 24.02 | 82.14 | 13.46 | 23.91 | 53.17 | 52.69 | 10.93 | 97.25 | 17.42 | 32.76 |
| 3.50 | 56.36 | 54.70 | 34.94 | 83.03 | 13.52 | 23.99 | 53.55 | 55.17 | 12.35 | 97.45 | 16.73 | 31.24 |
| 3.75 | 56.07 | 56.75 | 32.34 | 85.18 | 12.82 | 22.87 | 54.51 | 53.50 | 18.55 | 98.59 | 17.20 | 31.56 |
| 4.00 | 55.10 | 53.08 | 30.05 | 96.39 | 14.49 | 26.30 | 52.43 | 51.14 | 23.36 | 101.74 | 15.71 | 29.97 |
| 4.25 | 59.79 | 59.12 | 32.89 | 98.33 | 14.14 | 23.65 | 57.09 | 53.99 | 33.26 | 104.57 | 13.97 | 24.48 |
| 4.50 | 55.98 | 52.43 | 35.68 | 89.28 | 13.92 | 24.86 | 54.47 | 49.80 | 26.93 | 94.09 | 14.10 | 25.89 |
| 4.75 | 52.95 | 52.70 | 27.92 | 90.42 | 15.08 | 28.48 | 52.68 | 51.35 | 29.62 | 96.22 | 14.12 | 26.81 |
| 5.00 | 52.29 | 50.33 | 26.94 | 86.81 | 14.89 | 28.47 | 51.69 | 47.68 | 29.99 | 97.71 | 14.93 | 28.88 |
| 5.50 | 51.27 | 50.21 | 23.02 | 85.70 | 13.83 | 26.98 | 49.01 | 47.48 | 24.59 | 95.00 | 12.97 | 26.47 |
| 6.00 | 48.73 | 44.61 | 30.45 | 86.35 | 12.98 | 26.64 | 47.59 | 46.78 | 12.65 | 96.72 | 14.27 | 29.99 |
| 6.50 | 46.65 | 44.62 | 27.96 | 79.86 | 12.44 | 26.66 | 44.77 | 42.39 | 20.77 | 80.81 | 12.34 | 27.57 |
| 8.00 | 47.46 | 48.10 | 24.96 | 79.95 | 11.90 | 25.06 | 45.18 | 41.92 | 6.44 | 76.82 | 13.45 | 29.77 |
| 10.00 | 40.66 | 39.35 | 17.75 | 70.52 | 11.07 | 27.24 | 38.26 | 37.87 | 12.78 | 63.24 | 11.31 | 29.56 |
| 12.00 | 37.87 | 35.90 | 18.83 | 66.20 | 11.57 | 30.56 | 37.47 | 37.55 | 13.72 | 74.36 | 10.93 | 29.18 |
| 24.00 | 36.39 | 36.80 | 15.52 | 57.99 | 9.34 | 25.68 | 35.68 | 35.30 | 19.77 | 52.40 | 7.92 | 22.18 |
| 36.00 | 32.59 | 30.86 | 10.97 | 58.18 | 10.70 | 32.83 | 32.10 | 32.88 | 0.00 | 56.25 | 10.24 | 31.89 |
| 48.00 | 29.62 | 29.49 | 14.56 | 55.61 | 8.70 | 29.39 | 27.71 | 26.78 | 6.82 | 41.12 | 8.06 | 29.09 |



Table A3.4. Individual data and descriptive statistics for the levothyroxine pharmacokinetic parameters (C<sub>max</sub> in ng/mL, AUC<sub>0-t</sub> in ng\*h/mL, and AUC<sub>0-∞</sub> in ng\*h/mL). Including predose greater than 5%

| | Per | riod | | | C <sub>max</sub> | | | | AU | Cot | | | AU | C <sub>0∞</sub> | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Volunteer | Fo | rm | Sequence | Fo | orm | n/a | 1 = (D /A) | Fo | rm | D/A | 1-/D/A) | Fo | rm | D/A | Le/D/A) |
| | Α | В | 1 | Α | В | B/A | Ln(B/A) | Α | В | B/A | Ln(B/A) | Α | В | B/A | Ln(B/A) |
| 1 | 2 | 1 | BA | 98.33 | 84.97 | 0.86 | -0.15 | 2689.21 | 1962.33 | 0.73 | -0.32 | 7629.83 | 3185.87 | 0.42 | -0.87 |
| 2 | 2 | 1 | BA | 59.08 | 59.26 | 1.00 | 0.00 | 1837.68 | 1370.21 | 0.75 | -0.29 | 11399.25 | 2354.71 | 0.21 | -1.58 |
| 3 | 2 | 1 | BA | 61.00 | 56.41 | 0.92 | -0.08 | 1225.73 | 1095.22 | 0.89 | -0.11 | 3777.54 | 3797.19 | 1.01 | 0.01 |
| 4 | 1 | 2 | AB | 67.12 | 63.95 | 0.95 | -0.05 | 1591.53 | 1566.01 | 0.98 | -0.02 | 3378.30 | 2805.99 | 0.83 | -0.19 |
| 5 | 1 | 2 | AB | 53.06 | 59.02 | 1.11 | 0.11 | 1280.47 | 1327.98 | 1.04 | 0.04 | 2783.29 | 5019.26 | 1.80 | 0.59 |
| 6 | 2 | 1 | BA | 64.49 | 48.64 | 0.75 | -0.28 | 1808.01 | 1158.58 | 0.64 | -0.45 | 4711.82 | 3048.40 | 0.65 | -0.44 |
| 7 | 1 | 2 | AB | 64.47 | 69.43 | 1.08 | 0.07 | 1612.86 | 1922.93 | 1.19 | 0.18 | 4049.42 | 7788.41 | 1.92 | 0.65 |
| 8 | 1 | 2 | AB | 64.72 | 66.18 | 1.02 | 0.02 | 1636.89 | 1868.76 | 1.14 | 0.13 | 2868.45 | 4471.12 | 1.56 | 0.44 |
| 9 | 1 | 2 | AB | 84.71 | 104.57 | 1.23 | 0.21 | 2045.76 | 2607.86 | 1.27 | 0.24 | 4703.01 | 4314.79 | 0.92 | -0.09 |
| 10 | 1 | 2 | AB | 81.77 | 97.25 | 1.19 | 0.17 | 1996.53 | 2646.91 | 1.33 | 0.28 | 3703.43 | 6718.92 | 1.81 | 0.60 |
| 11 | 1 | 2 | AB | 68.86 | 72.27 | 1.05 | 0.05 | 1819.09 | 2275.38 | 1.25 | 0.22 | 3550.70 | 4959.64 | 1.40 | 0.33 |
| 12 | 2 | 1 | BA | 69.82 | 69.15 | 0.99 | -0.01 | 1891.63 | 1974.48 | 1.04 | 0.04 | 4532.57 | 3117.95 | 0.69 | -0.37 |
| 13 | 1 | 2 | AB | 62.06 | 51.70 | 0.83 | -0.18 | 2001.92 | 1534.42 | 0.77 | -0.27 | 6086.38 | 7351.71 | 1.21 | 0.19 |
| 14 | 2 | 1 | BA | 69.84 | 68.12 | 0.98 | -0.03 | 2004.14 | 2284.89 | 1.14 | 0.13 | 4664.28 | 5395.53 | 1.16 | 0.15 |
| 15 | 2 | 1 | BA | 51.95 | 54.48 | 1.05 | 0.05 | 1200.24 | 1699.47 | 1.42 | 0.35 | 2732.81 | 7145.54 | 2.61 | 0.96 |
| 16 | 2 | 1 | BA | 67.07 | 55.03 | 0.82 | -0.20 | 1510.80 | 1584.61 | 1.05 | 0.05 | 2995.80 | 2265.70 | 0.76 | -0.28 |
| 17 | 1 | 2 | AB | 66.14 | 68.33 | 1.03 | 0.03 | 1568.88 | 1626.36 | 1.04 | 0.04 | 1958.82 | 2041.21 | 1.04 | 0.04 |
| 18 | 2 | 1 | BA | 67.71 | 68.11 | 1.01 | 0.01 | 1843.99 | 1934.81 | 1.05 | 0.05 | 4232.42 | 5847.67 | 1.38 | 0.32 |
| 19 | 1 | 2 | AB | 73.11 | 56.02 | 0.77 | -0.27 | 2003.61 | 1500.69 | 0.75 | -0.29 | 4107.73 | 3381.13 | 0.82 | -0.19 |
| 20 | 2 | 1 | BA | 74.61 | 60.44 | 0.81 | -0.21 | 2335.65 | 1506.84 | 0.65 | -0.44 | 5651.05 | 3602.09 | 0.64 | -0.45 |
| 21 | 2 | 1 | BA | 68.94 | 67.03 | 0.97 | -0.03 | 1878.60 | 2016.17 | 1.07 | 0.07 | 5532.19 | 3558.37 | 0.64 | -0.44 |
| 22 | 1 | 2 | AB | 50.81 | 43.65 | 0.86 | -0.15 | 1094.52 | 1350.77 | 1.23 | 0.21 | 2115.19 | 4602.71 | 2.18 | 0.78 |
| 23 | 2 | 1 | BA | 50.16 | 73.24 | 1.46 | 0.38 | 1288.89 | 1856.73 | 1.44 | 0.37 | 2389.96 | 6212.32 | 2.60 | 0.96 |
| 24 | 1 | 2 | AB | 75.62 | 60.54 | 0.80 | -0.22 | 1586.03 | 1327.55 | 0.84 | -0.18 | 2452.72 | 3747.07 | 1.53 | 0.42 |
| 25 | 1 | 2 | AB | 59.68 | 62.69 | 1.05 | 0.05 | 1371.46 | 1872.81 | 1.37 | 0.31 | 3601.75 | 3002.78 | 0.83 | -0.18 |
| 26 | 1 | 2 | AB | 51.65 | 54.58 | 1.06 | 0.06 | 1641.62 | 1759.85 | 1.07 | 0.07 | 3342.39 | 3811.39 | 1.14 | 0.13 |
| 27 | 2 | 1 | BA | 48.06 | 52.34 | 1.09 | 0.09 | 1397.92 | 1342.50 | 0.96 | -0.04 | 3116.06 | 1840.81 | 0.59 | -0.53 |
| 28 | 2 | 1 | BA | 121.16 | 105.75 | 0.87 | -0.14 | 2365.84 | 1777.07 | 0.75 | -0.29 | 6969.94 | 2829.90 | 0.41 | -0.90 |
| 29 | 2 | 1 | BA | 65.35 | 60.17 | 0.92 | -0.08 | 1614.56 | 1100.34 | 0.68 | -0.38 | 2345.54 | 1261.22 | 0.54 | -0.62 |
| 30 | 1 | 2 | AB | 68.88 | 71.68 | 1.04 | 0.04 | 2052.91 | 1856.34 | 0.90 | -0.10 | 7712.38 | 7998.73 | 1.04 | 0.04 |
| 31 | 1 | 2 | AB | 49.54 | 62.01 | 1.25 | 0.22 | 984.41 | 1681.30 | 1.71 | 0.54 | 1682.68 | 3464.68 | 2.06 | 0.72 |
| 32 | 1 | 2 | AB | 61.04 | 62.17 | 1.02 | 0.02 | 1508.72 | 1521.89 | 1.01 | 0.01 | 6168.89 | 2613.22 | 0.42 | -0.86 |
| 33 | 1 | 2 | AB | 86.93 | 82.18 | 0.95 | -0.06 | 2777.76 | 1970.60 | 0.71 | -0.34 | 9404.14 | 4094.94 | 0.44 | -0.83 |
| 34 | 1 | 2 | AB | 60.92 | 70.24 | 1.15 | 0.14 | 1423.86 | 1468.97 | 1.03 | 0.03 | 3357.06 | 2278.05 | 0.68 | -0.39 |
| 35 | 1 | 2 | AB | 59.46 | 52.07 | 0.88 | -0.13 | 1829.52 | 1581.34 | 0.86 | -0.15 | 5265.86 | 8982.58 | 1.71 | 0.53 |
| 36 | 2 | 1 | BA | 74.82 | 70.08 | 0.94 | -0.07 | 1468.93 | 1750.43 | 1.19 | 0.18 | 2996.07 | 4872.32 | 1.63 | 0.49 |
| 37 | 2 | 1 | BA | 60.30 | 68.30 | 1.13 | 0.12 | 1801.46 | 2017.01 | 1.12 | 0.11 | 4862.37 | 9642.45 | 1.98 | 0.68 |
| 39 | 2 | 1 | BA | 100.38 | 94.09 | 0.94 | -0.06 | 2748.65 | 2212.77 | 0.81 | -0.22 | 6147.33 | 4801.43 | 0.78 | -0.25 |
| 40 | 2 | 1 | BA | 90.55 | 78.08 | 0.86 | -0.15 | 2560.22 | 2227.62 | 0.87 | -0.14 | 4307.50 | 4618.20 | 1.07 | 0.07 |
| 41 | 2 | 1 | BA | 72.78 | 79.08 | 1.09 | 0.08 | 1795.04 | 1564.48 | 0.87 | -0.14 | 4528.22 | 2357.15 | 0.52 | -0.65 |
| 42 | 1 | 2 | AB | 44.51 | 33.98 | 0.76 | -0.27 | 1250.47 | 1223.34 | 0.98 | -0.02 | 4821.73 | 8541.54 | 1.77 | 0.57 |
| 43 | 2 | 1 | BA | 51.13 | 56.81 | 1.11 | 0.11 | 1529.05 | 1337.85 | 0.87 | -0.13 | 3297.62 | 3246.45 | 0.98 | -0.02 |
| 44 | 1 | 2 | AB | 51.87 | 47.59 | 0.92 | -0.09 | 1426.32 | 1293.80 | 0.91 | -0.10 | 8140.54 | 3276.84 | 0.40 | -0.91 |
| | N | | | 43.00 | 43.00 | 43.00 | 43.00 | 43.00 | 43.00 | 43.00 | 43.00 | 43.00 | 43.00 | 43.00 | 43.00 |
| | ometr | | | 65.78 | 64.47 | 0.98 | NA | 1700.84 | 1670.95 | 0.98 | NA | 4117.37 | 3989.61 | 0.97 | NA |
| | ithmet | | | 67.31 | 66.09 | 0.99 | -0.02 | 1751.20 | 1710.70 | 1.01 | -0.02 | 4513.37 | 4424.84 | 1.13 | -0.03 |
| Star | ndard I | | ion | 15.45 | 15.13 | 0.15 | 0.14 | 435.41 | 378.25 | 0.24 | 0.23 | 2068.32 | 2074.66 | 0.62 | 0.59 |
| | %( | | | 22.95 | 22.90 | 14.72 | -719.49 | 24.86 | 22.11 | 23.54 | -1306.44 | 45.83 | 46.89 | 54.81 | -1869.16 |
| M | linimur | | ie | 44.51 | 33.98 | 0.75 | -0.28 | 984.41 | 1095.22 | 0.64 | -0.45 | 1682.68 | 1261.22 | 0.21 | -1.58 |
| | Med | | | 65.35 | 63.95 | 0.99 | -0.01 | 1641.62 | 1681.30 | 1.01 | 0.01 | 4107.73 | 3797.19 | 1.01 | 0.01 |
| | aximu | | | 121.16 | 105.75 | 1.46 | 0.38 | 2777.76 | 2646.91 | 1.71 | 0.54 | 11399.25 | 9642.45 | 2.61 | 0.96 |
| NA: Not a | applio | cable | • | | | | | | | | | | | | |



Table A3.5. Levothyroxine Pharmacokinetic Parameters Results, including predose greater than 5%.

| | | | | Fo | rm | | | |
|---|---|---|---|---|---|---|---|---|
| Variable | E | Eutirox® approv | ved formulatio | n (A) | | Eutirox® test | formulation ( | B) |
| variable | N | Arithmetic<br>Mean | Standard<br>Deviation | %CV | N | Arithmetic<br>Mean | Standard<br>Deviation | %CV |
| Extrapolated AUC (%) | 43.00 | 56.71 | 12.80 | 22.56 | 43.00 | 54.51 | 17.63 | 32.35 |
| $AUC_{0-\infty}$ (ng*h/mL) | 43.00 | 4513.37 | 2068.32 | 45.83 | 43.00 | 4424.84 | 2074.66 | 46.89 |
| AUC <sub>0-t</sub> (ng*h/mL) | 43.00 | 1751.20 | 435.42 | 24.86 | 43.00 | 1710.70 | 378.25 | 22.11 |
| CI/F (mL/h) | 43.00 | 158.97 | 67.19 | 42.26 | 43.00 | 166.99 | 80.99 | 48.50 |
| C <sub>máx</sub> (ng/mL) | 43.00 | 67.31 | 15.45 | 22.95 | 43.00 | 66.09 | 15.13 | 22.90 |
| t 1/2 (h) | 43.00 | 61.57 | 32.13 | 52.18 | 43.00 | 62.32 | 36.07 | 57.88 |
| Kel (1/h) | 43.00 | 0.01 | 0.01 | 46.06 | 43.00 | 0.01 | 0.01 | 54.74 |
| TMR (h) | 43.00 | 92.33 | 45.56 | 49.35 | 43.00 | 93.19 | 53.14 | 57.02 |
| T <sub>lag</sub> (h) | 43.00 | 0.09 | 0.20 | 211.64 | 43.00 | 0.02 | 0.11 | 458.13 |
| T <sub>máx</sub> (h) | 43.00 | 3.52 | 1.20 | 33.97 | 43.00 | 3.50 | 1.14 | 32.58 |
| Vd/F (mL) | 43.00 | 12013.60 | 3144.99 | 26.18 | 43.00 | 11950.47 | 2697.91 | 22.58 |

Table A3.6. ANOVA table for the analysis of the levothyroxine logarithmically-transformed pharmacokinetic parameters (Ln), including predose greater than 5%.

| Assessed<br>Variable | Source of Variation | Degrees of<br>Freedom | Square Sum | Squared Means | F Value | P Value | Criterion (P > 0.05) |
|---|---|---|---|---|---|---|---|
| Ln(C <sub>max</sub> ) | Sequence | 11 | 0.13 | 0.13 | 1.58 | 0.22 | Pass |
| Ln(C <sub>max</sub> ) | Sequence*Volunteer | 41 | 3.46 | 8.43 x 10 <sup>-2</sup> | | | Not applicable |
| Ln(C <sub>max</sub> ) | Form | 1 | 8.61 x 10 <sup>-3</sup> | 8.61 x 10 <sup>-3</sup> | 0.82 | 0.37 | Pass |
| Ln(C <sub>max</sub> ) | Period | 1 | 2.28 x 10 <sup>-3</sup> | 2.28 x 10 <sup>-3</sup> | 0.22 | 0.64 | Pass |
| Ln(C <sub>max</sub> ) | Error | 41 | 0.43 | 1.05 x 10 <sup>-2</sup> | | | Not applicable |
| Ln(AUC <sub>0-t</sub> ) | Sequence | 1 | 4.79 x 10 <sup>-2</sup> | 4.79 x 10 <sup>-2</sup> | 0.59 | 0.45 | Pass |
| Ln(AUC <sub>0-t</sub> ) | Sequence*Volunteer | 41 | 3.34 | 0.08 | | | Not applicable |
| Ln(AUC <sub>0-t</sub> ) | Form | 1 | 6.76 x 10 <sup>-3</sup> | 6.76 x 10 <sup>-3</sup> | 0.26 | 0.61 | Pass |
| Ln(AUC <sub>0-t</sub> ) | Period | 1 | 7.01 x 10 <sup>-2</sup> | 7.01 x 10 <sup>-2</sup> | 2.72 | 0.11 | Pass |
| Ln(AUC <sub>0-t</sub> ) | Error | 41 | 1.06 | 2.58 x 10 <sup>-2</sup> | | | Not applicable |
| Ln(AUC <sub>0-∞</sub> ) | Sequence | 1 | 3.38 x 10 <sup>-2</sup> | 3.38 x 10 <sup>-2</sup> | 0.15 | 0.70 | Pass |
| Ln(AUC <sub>0-∞</sub> ) | Sequence*Volunteer | 41 | 9.41 | 0.23 | | | Not applicable |
| Ln(AUC <sub>0∞</sub> ) | Form | 1 | 2.14 x 10 <sup>-2</sup> | 2.14 x10 <sup>-2</sup> | 0.13 | 0.72 | Pass |
| Ln(AUC <sub>0∞</sub> ) | Period | 1 | 0.45 | 0.45 | 2.68 | 0.11 | Pass |
| Ln(AUC <sub>0∞</sub> ) | Error | 41 | 6.84 | 0.17 | | | Not applicable |

| T <sub>0</sub> | ANALYTICAL UNIT | Issue | 10-Mar-2020 |
|----------------|----------------------|---------|-------------|
| PPD | ANALYTICAL UNIT | Version | 1.0 |

Table A3.7 shows the results of the bioequivalence statistics for the levothyroxine logarithmically-transformed pharmacokinetic data, including predose greater than 5%.

Table A3.7 Statistics of the Levothyroxine Bioequivalence Determination.

| Parameter | | onfidence | | mann's<br>d-side t | Power | Acceptance | Meets<br>the |
|---|---|---|---|---|---|---|---|
| | Inte | erval | P < 80 % | P<br>> 125 % | (%) | Acceptance<br>Criterion<br>(80-125) | Criterion |
| LnCmax | 94.40 | 101.72 | 0.00 | 0.00 | 100.00 | (80-125) | YES |
| LnAUC <sub>0-t</sub> | 92.55 | 104.00 | 0.00 | 0.00 | 99.99 | (80-125) | YES |

#### 11. References

- Chow S. C. y Liu J. P. (2009). Design and Analysis of Bioavailability and Bioequivalence Studies Third edition. USA: CRC Press.
- Mexican Official Standard NOM-177-SSA1-2013. Which establishes the tests and
  procedures to prove that a drug is interchangeable. The requirements for third parties
  performing interchangeability tests should fulfill. The requirements for conducting
  biocomparability studies. Requirements that third parties, investigational sites, or
  hospital institutions performing interchangeability tests must adhere to.

# 12. History of Changes

| DATE OF CHANGE | CHANGE DESCRIPTION | LEVEL |
|----------------|--------------------|-------|
| | New Document | 1.0 |